CLINICAL TRIAL: NCT02723955
Title: A Phase I Open Label Study of GSK3359609 Administered Alone and in Combination With Anticancer Agents in Subjects With Selected Advanced Solid Tumors
Brief Title: Dose Escalation and Expansion Study of GSK3359609 in Participants With Selected Advanced Solid Tumors (INDUCE-1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 204691; 2016-000148-32 (EudraCT Number)
Record Dates: First submitted 2016-03-24; First posted 2016-03-31 (Estimated); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-11

CONDITIONS: Neoplasms
Keywords: ICOS receptor agonist antibody; Pembrolizumab; KEYNOTE-478; GSK3359609; Cohort expansion; Dose escalation; Dostarlimab; Cobolimab; Bintrafusp alfa
MeSH Terms: conditions — Neoplasms | interventions — pembrolizumab; Docetaxel; Pemetrexed; Paclitaxel; Carboplatin; Gemcitabine; Fluorouracil; Cisplatin; dostarlimab; bintrafusp alfa protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part 1A: Dose escalation feladilimab (GSK3359609) (Experimental): Participants will receive feladilimab (GSK3359609) administered continuously at a dose level dependent on to which dose level the participant is accrued.
  Interventions: Drug: feladilimab (GSK3359609)
- Part 1B: Expansion feladilimab (GSK3359609) (Experimental): Participants will receive feladilimab (GSK3359609) administered continuously at a dose level chosen for further exploration in dose expansion cohorts.
  Interventions: Drug: feladilimab (GSK3359609)
- Part 2A: Dose escalation (feladilimab (GSK3359609)+pembrolizumab) (Experimental): Participants will receive feladilimab (GSK3359609) administered continuously in combination with pembrolizumab.
  Interventions: Drug: feladilimab (GSK3359609); Drug: Pembrolizumab
- Part 2A: Dose escalation (feladilimab (GSK3359609)+GSK3174998) (Experimental): Participants will receive feladilimab (GSK3359609) administered continuously in combination with GSK3174998.
  Interventions: Drug: feladilimab (GSK3359609); Drug: GSK3174998
- Part 2A: Safety run-in (feladilimab (GSK3359609)+chemotherapy) (Experimental): Participants participating in Part 2A chemotherapy combination cohorts will receive feladilimab (GSK3359609) in combination with chemotherapy at doses and schedules based on standard of care practice.
  Interventions: Drug: feladilimab (GSK3359609); Drug: Docetaxel; Drug: Pemetrexed; Drug: Paclitaxel plus Carboplatin; Drug: Gemcitabine plus Carboplatin; Drug: Fluorouracil (5-FU) plus carboplatin or cisplatin
- Part 2B: Expansion-feladilimab (GSK3359609) (Experimental): Participants will receive feladilimab (GSK3359609) administered continuously in combination with pembrolizumab.
  Interventions: Drug: feladilimab (GSK3359609); Drug: Pembrolizumab
- Part 2A: Dose escalation (feladilimab (GSK3359609)+ dostarlimab) (Experimental): Participants will receive feladilimab (GSK3359609) administered continuously in combination with dostarlimab.
  Interventions: Drug: feladilimab (GSK3359609); Drug: Dostarlimab
- Part 2A: Dose escalation (feladilimab (GSK3359609)+dostarlimab+cobolimab) (Experimental): Participants will receive feladilimab (GSK3359609) administered continuously in combination with dostarlimab followed by cobolimab.
  Interventions: Drug: feladilimab (GSK3359609); Drug: Dostarlimab; Drug: Cobolimab
- Part 2A: Dose escalation (feladilimab (GSK3359609)+bintrafusp alfa) (Experimental): Participants will receive feladilimab (GSK3359609) administered continuously in combination with bintrafusp alfa.
  Interventions: Drug: feladilimab (GSK3359609); Drug: Bintrafusp alfa

INTERVENTIONS:
Drug: feladilimab (GSK3359609)
Drug: GSK3174998
  Arms: Part 2A: Dose escalation (feladilimab (GSK3359609)+GSK3174998)
Drug: Pembrolizumab
  Arms: Part 2A: Dose escalation (feladilimab (GSK3359609)+pembrolizumab); Part 2B: Expansion-feladilimab (GSK3359609)
Drug: Docetaxel
  Arms: Part 2A: Safety run-in (feladilimab (GSK3359609)+chemotherapy)
Drug: Pemetrexed
  Arms: Part 2A: Safety run-in (feladilimab (GSK3359609)+chemotherapy)
Drug: Paclitaxel plus Carboplatin
  Arms: Part 2A: Safety run-in (feladilimab (GSK3359609)+chemotherapy)
Drug: Gemcitabine plus Carboplatin
  Arms: Part 2A: Safety run-in (feladilimab (GSK3359609)+chemotherapy)
Drug: Fluorouracil (5-FU) plus carboplatin or cisplatin
  Arms: Part 2A: Safety run-in (feladilimab (GSK3359609)+chemotherapy)
Drug: Dostarlimab
  Arms: Part 2A: Dose escalation (feladilimab (GSK3359609)+ dostarlimab); Part 2A: Dose escalation (feladilimab (GSK3359609)+dostarlimab+cobolimab)
Drug: Cobolimab
  Arms: Part 2A: Dose escalation (feladilimab (GSK3359609)+dostarlimab+cobolimab)
Drug: Bintrafusp alfa
  Arms: Part 2A: Dose escalation (feladilimab (GSK3359609)+bintrafusp alfa)

SUMMARY:
GSK3359609 is an anti-Inducible T cell Co-Stimulator (ICOS) receptor agonist antibody intended for the treatment of cancers of different histology. This is a first-time-in-human (FTIH), open-label, multicenter study designed to investigate the safety, pharmacology, and preliminary antitumor activity in participants with selected, advanced or recurrent solid tumors with the aim to establish recommended dose(s) of GSK3359609 for further exploration as monotherapy and in combination with pembrolizumab or chemotherapy regimens. The study is comprised of two primary parts, each composed of two phases: Part 1: GSK3359609 monotherapy with Part 1A as dose escalation phase and Part 1B as cohort expansion phase; Part 2: GSK3359609 combination therapy with Part 2A pembrolizumab or GSK3174998 or chemotherapy or pembrolizumab plus chemotherapy or dostarlimab plus cobolimab or Bintrafusp alfa combination dose escalation phase and Part 2B expansion phase with pembrolizumab. The primary objective of the study is to determine the safety, tolerability, maximum tolerated dose or the maximum administered dose of GSK3359609 alone or in combination.

ELIGIBILITY:
Inclusion Criteria

* Capable of giving signed, written informed consent.
* Male or female, age 18 to 93 years (at the time consent is obtained).
* Histological or cytological documentation of an invasive malignancy that was diagnosed as locally advanced/metastatic or relapsed/refractory and is of one of the following tumor types: bladder/urothelial cancer of the upper and lower urinary tract; cervical; colorectal (includes appendix); esophagus, squamous cell; head and neck carcinoma; melanoma; malignant pleural mesothelioma (MPM); non-small-cell lung cancer (NSCLC), prostate; Microsatellite Instability-High/deficient mismatch repair (MSI-H/dMMR) tumor (Part 1B and Part 2B) and Human Papilloma Virus (HPV)-positive or Epstein-Barr (EBV)-positive tumor (Part 1B and Part 2B).
* Disease that has progressed after standard therapy for the specific tumor type, or for which standard therapy has proven to be ineffective, intolerable, or is considered inappropriate, or if no further standard therapy exists; exceptions are in these tumor types in which pembrolizumab single agent may be a standard: NSCLC, head and neck squamous cell cancer (HNSCC), bladder/urothelial cancer, MSI-H/dMMR cancers and melanoma and cervical cancer. In Part 2B pembrolizumab combination expansion cohorts, prior treatment with anti-Programmed cell death protein 1(PD-1)/ Ligand-1 (L1) may not be required. 1) Participants must not have received more than 5 prior lines of therapy for advanced disease including both standards of care and investigational therapies. 2) Participants who received prior PD-1/L1 therapy must fulfill the following requirements (Part 1B [except PK/PD cohort]/ Part 2B):a) Have achieved a CR, PR or SD and subsequently had disease progression while still on PD-1/L1 therapy; b) Have received at least 2 doses of an approved PD-1/L1 inhibitor (by any regulatory authority), c) Have demonstrated disease progression as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 within 18 weeks from the last dose of the PD-1/L1 inhibitor. The initial evidence of disease progression is to be confirmed by a second assessment no less than four weeks from the date of the first documented Progressive Disease (PD) (the confirmatory scan could be the Baseline eligibility scan for this study). 3) In Part 2A 5-fluorouracil (FU)/platinum combination with GSK3359609 and pembrolizumab cohort, participants must not have received prior systemic therapy administered in the recurrent or metastatic setting (with the exception of systemic therapy given as part of multimodal treatment for locally advanced disease).
* Archival tumor tissue obtained at any time from the initial diagnosis to study entry; a fresh tumor biopsy using a procedure that is safe for the participant on a lesion not previously irradiated unless lesion progressed will be required if archival tissue is unavailable.
* Agree to undergo a pre-treatment and on treatment biopsy and have disease amenable to biopsy required in pharmacokinetic (PK) / pharmacodynamics (PD), dose randomized HNSCC, Melanoma dose expansion and Biomarker cohorts..
* Measurable disease per RECIST version 1.1. Palpable lesions that are not measurable by radiographic or photographic evaluations may not be utilized as the only measurable lesion. Any measurable lesion biopsied at Screening cannot be followed as a target/index lesion unless agreed upon by GlaxoSmithKline (GSK).
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1.
* Life expectancy of at least 12 weeks.
* Adequate organ function.
* QT interval corrected for heart rate according to Fridericia's formula (QTcF) <450 milliseconds (msec) or QTcF <480 msec for participants with bundle branch block.
* A female participant is eligible to participate if she is not pregnant (as confirmed by a negative serum beta-human chorionic gonadotrophin [beta-hCG] test in females of reproductive potential), and not lactating or reproductive potential agrees to follow one of the options listed in protocol from 30 days prior to the first dose of study medication and until 120 days after the last dose of study treatment.
* Male participants with female partners of child bearing potential must agree to use one of the methods of contraception specified in protocol from time of first dose of study treatment until 120 days after the last dose of study treatment.
* Documented HPV/ EBV-positive tumor as determined by a local laboratory for Part 1B and Part 2B pembrolizumab combination viral-positive expansion cohorts only.
* Documented MSI-H or dMMR-positive tumor as determined by local laboratory for Part 1B and Part 2B pembrolizumab combination MSI-H/dMMR expansion cohorts only.
* ICOS expression result using an analytically validated immunohistochemistry (IHC) assay by central laboratory for Part 1B biomarker cohort only.
* Gene expression (GEX) result using an analytically validated method by central laboratory (Part 1B Biomarker Cohort only).
* PD-L1 combined positive score (CPS) <1 using the Food and Drug Administration (FDA) approved PD-L1 IHC 22C3 pharmdx assay by central laboratory testing for Part 2B HNSCC PD-L1 CPS <1 Cohort. Documented test result from FDA approved PD-L1 IHC 22C3 pharmDx assay in local laboratory, if available, may be accepted in lieu of the central laboratory test result.

Exclusion Criteria

* Prior treatment with the following therapies:

Â• Anticancer therapy within 30 days or 5 half-lives of the drug, whichever is shorter. At least 14 days must have elapsed between the last dose of prior anticancer agent and the first dose of study drug is administered.

Â• Part 2B (GSK3359609/pembrolizumab combination): prior pembrolizumab washout is not required.

Â• Prior radiation therapy: permissible if at least one non-irradiated measurable lesion is available for assessment according to RECIST version 1.1 or if a solitary measurable lesion was irradiated, objective progression is documented. A wash out of at least two weeks before start of study drug for radiation of any intended use to the extremities for bone metastases and 4 weeks for radiation to the chest, brain, or visceral organs is required. Â• Investigational therapy within 30 days or 5 half-lives of the investigational product (whichever is shorter). At least 14 days must have elapsed between the last dose of investigational agent and the first dose of study drug is administered.

* Prior allogeneic or autologous bone marrow transplantation or other solid organ transplantation.
* Toxicity from previous anticancer treatment
* Invasive malignancy or history of invasive malignancy other than disease under study within the last two years except: Any other invasive malignancy for which the participant was definitively treated, has been disease-free for <=2 years and in the opinion of the principal investigator and GSK Medical Monitor will not affect the evaluation of the effects of the study treatment on the currently targeted malignancy, may be included in this clinical trial; and curatively treated non-melanoma skin cancer.
* Central nervous system (CNS) metastases, with the following exception: Â• Participants who have previously-treated CNS metastases, are asymptomatic, and have no requirement for steroids at least 14 days prior to first dose of study drug. Participants with carcinomatous meningitis or leptomeningeal spread are excluded regardless of clinical stability.
* Received transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including granulocyte colony-stimulating factor [G-CSF], granulocyte-macrophage colony-stimulating factor, recombinant erythropoietin) within 14 days prior to the first dose of GSK3359609.
* Major surgery <=4 weeks before the first dose of study treatment. Participants must have also fully recovered from any surgery (major or minor) and/or its complications before initiating study treatment.
* Active autoimmune disease that has required systemic treatment within the last two years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Concurrent medical condition requiring the use of systemic immunosuppressive medications within 7 days before the first dose of study treatment. Physiologic doses of corticosteroids for treatment of endocrinopathies or steroids with minimal systemic absorption, including topical, inhaled, or intranasal corticosteroids may be continued if the participant is on a stable dose.
* Condition requiring treatment with strong inhibitors/inducers of cytochrome p (CYP) 450 3A4 within 7 days prior to first dose of chemotherapy (requirement applies to participants enrolled to Part 2 chemotherapy combination with docetaxel).
* Active infection requiring systemic therapy, known human immunodeficiency virus infection, or positive test for hepatitis B active infection or hepatitis C active infection.
* Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones, liver metastases, or otherwise stable chronic liver disease per investigator assessment).
* Recent history (within the past 6 months) of acute diverticulitis, inflammatory bowel disease, intra-abdominal abscess, or gastrointestinal obstruction that required surgery.
* Receipt of any live vaccine within 4 weeks prior to first dose of study treatment.
* Recent history of allergen desensitization therapy within 4 weeks of starting study treatment.
* History of severe hypersensitivity to monoclonal antibodies or to the chemotherapies under investigation including any ingredient used in the formulation.
* History or evidence of cardiac abnormalities.
* History of (current and past) idiopathic pulmonary fibrosis, pneumonitis (for past pneumonitis exclusion only if steroids were required for treatment), interstitial lung disease, or organizing pneumonia. Note: post-radiation changes in the lung related to prior radiotherapy and/or asymptomatic radiation-induced pneumonitis not requiring treatment may be permitted if agreed by the investigator and Medical Monitor.
* Recent history (within 6 months) of uncontrolled symptomatic ascites or pleural effusions.
* Any serious and/or unstable pre-existing medical, psychiatric disorder, or other condition that could interfere with the participant's safety, obtaining informed consent, or compliance to the study procedures.

Ages: 18 Years to 93 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 829 (Actual)
Dates: Start 2016-06-23 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (25):
- United States (7):
  - GSK Investigational Site, Duarte, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Nashville, Tennessee
- Australia (3):
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- GSK Investigational Site, Toronto, Ontario, Canada
- GSK Investigational Site, Shnghai, China
- France (4):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Villejuif
- GSK Investigational Site, Siena, Tuscany, Italy
- Japan (3):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
- GSK Investigational Site, Amsterdam, Netherlands
- Spain (4):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, MÃ¡ga
  - GSK Investigational Site, Seville

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Turner DC, Wada R, Zhou H, Wang X, de Greef R, Valiathan C, Zhang L, Zhang N, Kuchimanchi M, Chen TT, Ballas M, Visser SAG. Model-based meta-analysis of non-small cell lung cancer with standard of care PD-1 inhibitors and chemotherapy for early development decision making. CPT Pharmacometrics Syst Pharmacol. 2023 Nov;12(11):1751-1763. doi: 10.1002/psp4.12917. Epub 2023 Jan 31. PMID 36642813
- [Derived] Yadavilli S, Waight JD, Brett S, Bi M, Zhang T, Liu YB, Ellis C, Turner DC, Hahn A, Shi H, Seestaller-Wehr L, Jing J, Xie Q, Shaik JS, Ji X, Gagnon R, Fieles W, Hook L, Grant S, Hopley S, DeYoung MP, Blackwell C, Chisamore M, Biddlecombe R, Figueroa DJ, Hopson CB, Srinivasan R, Smothers J, Maio M, Rischin D, Olive D, Paul E, Mayes PA, Hoos A, Ballas M. Activating Inducible T-cell Costimulator Yields Antitumor Activity Alone and in Combination with Anti-PD-1 Checkpoint Blockade. Cancer Res Commun. 2023 Aug 16;3(8):1564-1579. doi: 10.1158/2767-9764.CRC-22-0293. eCollection 2023 Aug. PMID 37593752

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 829 participants were enrolled.
Groups:
- Part 1A: Feladilimab (Fela) 0.001 Milligram/Kilogram (mg/kg): Participants with advanced solid tumors received 0.001 mg/kg feladilimab intravenous (IV) infusion once in a three week (Q3W) of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 1A: Fela 0.003 mg/kg: Participants with advanced solid tumors received 0.003 mg/kg feladilimab IV infusion Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 1A: Fela 0.010 mg/kg: Participants with advanced solid tumors received 0.010 mg/kg feladilimab IV infusion Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 1A: Fela 0.030 mg/kg: Participants with advanced solid tumors received 0.030 mg/kg feladilimab IV infusion Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 1A: Fela 0.100 mg/kg: Participants with advanced solid tumors received 0.100 mg/kg feladilimab IV infusion Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 1A: Fela 0.300 mg/kg; Part 1B: Fela 0.300 mg/kg: Participants with advanced solid tumors received 0.300 mg/kg feladilimab IV infusion Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 1A: Fela 1.000 mg/kg; Part 1B: Fela 1.000 mg/kg: Participants with advanced solid tumors received 1.000 mg/kg feladilimab IV infusion Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 1A: Fela 3.000 mg/kg: Participants with advanced solid tumors received 3.000 mg/kg feladilimab IV infusion Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 1A: Fela 10.000 mg/kg: Participants with advanced solid tumors received 10.000 mg/kg feladilimab IV infusion Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 1B: Fela 24 mg: Participants with advanced solid tumors received 24 mg feladilimab IV infusion Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2A: Fela 0.010 mg/kg + Pembrolizumab (Pembro) 200 mg: Participants with advanced solid tumors received 0.010 mg/kg feladilimab IV infusion in combination with 200 mg of pembro IV infusion Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2A: Fela 0.030 mg/kg + Pembro 200 mg: Participants with advanced solid tumors received 0.030 mg/kg feladilimab IV infusion in combination with 200 mg of pembro IV infusion Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2A: Fela 0.100 mg/kg + Pembro 200 mg: Participants with advanced solid tumors received 0.100 mg/kg feladilimab IV infusion in combination with 200 mg of pembro IV infusion Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2A: Fela 0.300 mg/kg + Pembro 200 mg; Part 2B: Fela 0.300 mg/kg + Pembro 200 mg: Participants with advanced solid tumors received 0.300 mg/kg feladilimab IV infusion in combination with 200 mg of pembro IV infusion Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2A: Fela 1.000 mg/kg + Pembro 200 mg; Part 2B: Fela 1.000 mg/kg + Pembro 200 mg: Participants with advanced solid tumors received 1.000 mg/kg feladilimab IV infusion in combination with 200 mg of pembro IV infusion Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2A: Fela 3.000 mg/kg + Pembro 200 mg; Part 2B: Fela 3.000 mg/kg + Pembro 200 mg: Participants with advanced solid tumors received 3.000 mg/kg feladilimab IV infusion in combination with 200 mg of pembro IV infusion Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2A: Fela 8 mg + GSK3174998 8 mg: Participants with advanced solid tumors received 8 mg feladilimab IV infusion in combination with 8 mg of GSK3174998 IV infusion Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2A: Fela 8 mg + GSK3174998 24 mg: Participants with advanced solid tumors received 8 mg feladilimab IV infusion in combination with 24 mg of GSK3174998 IV infusion Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2A: Fela 24 mg + GSK3174998 24 mg: Participants with advanced solid tumors received 24 mg feladilimab IV infusion in combination with 24 mg of GSK3174998 IV infusion Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2A: Fela 80 mg + GSK3174998 24 mg: Participants with advanced solid tumors received 80 mg feladilimab IV infusion in combination with 24 mg of GSK3174998 IV infusion Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2A: Fela 80 mg + GSK3174998 80 mg: Participants with advanced solid tumors received 80 mg feladilimab IV infusion in combination with 80 mg of GSK3174998 IV infusion Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2A: Fela 24 mg + Chemotherapy: Participants with advanced solid tumors received 24 mg feladilimab IV infusion in combination with chemotherapy Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2A: Fela 80 mg + Chemotherapy: Participants with advanced solid tumors received 80 mg feladilimab IV infusion in combination with chemotherapy Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2A: Fela 24 mg + 200 mg Pembro + Chemotherapy: Participants with advanced solid tumors received 24 mg feladilimab IV infusion in combination with chemotherapy and 200 mg of pembro IV infusion Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2A: Fela 80 mg + 200 mg Pembro + Chemotherapy: Participants with advanced solid tumors received 80 mg feladilimab IV infusion in combination with chemotherapy and 200 mg of pembro IV infusion Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2A: Fela 24 mg + Dostarlimab 500 mg + Cobolimab 300 mg: Participants with advanced solid tumors received 24 mg feladilimab IV infusion in combination with 500 mg dostarlimab and 300 mg cobolimab IV infusion Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2A: Fela 24 mg + Bintrafusp Alfa 2400 mg: Participants with advanced solid tumors received 24 mg feladilimab IV infusion in combination with 2400 mg bintrafusp alfa IV infusion Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2B: Fela 0.100 mg/kg + Pembro 200 mg: Participants with advanced solid tumors received 0.100 mg/kg feladilimab IV infusion in combination with 200 mg of pembro IV infusion every 3 Week (Q3W) of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2B: Fela 24 mg + Pembro 200 mg: Participants with advanced solid tumors received 24 mg feladilimab IV infusion in combination with 200 mg of pembro IV infusion Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2B: Fela 48 mg + Pembro 400 mg: Participants with advanced solid tumors received 48 mg feladilimab IV infusion in combination with 400 mg of pembro IV infusion Q6W of each 42-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2B: Fela 160 mg + Pembro 400 mg: Participants with advanced solid tumors received 160 mg feladilimab IV infusion in combination with 400 mg of pembro IV infusion Q6W of each 42-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2B: Fela 80 mg + Pembro 200 mg: Participants with advanced solid tumors received 80 mg feladilimab IV infusion in combination with 200 mg of pembro IV infusion Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Crossover: Fela 0.100 mg/kg + Pembro 200 mg: Participants with advanced solid tumors who received feladilimab monotherapy administered Q3W (Part 1) were crossover upon disease progression and received 0.100 mg/kg feladilimab IV infusion in combination with 200 mg pembrolizumab Q3W.
- Crossover: Fela 0.300 mg/kg + Pembro 200 mg: Participants with advanced solid tumors who received feladilimab monotherapy administered Q3W (Part 1) were crossover upon disease progression and received 0.300 mg/kg feladilimab IV infusion in combination with 200 mg pembrolizumab IV infusion Q3W.
- Crossover: Fela 1.000 mg/kg + Pembro 200 mg: Participants with advanced solid tumors who received feladilimab monotherapy administered Q3W (Part 1) were crossover upon disease progression and received 1.000 mg/kg feladilimab in combination with 200 mg pembrolizumab Q3W.
- Crossover: Fela 3.000 mg/kg + Pembro 200 mg: Participants with advanced solid tumors who received feladilimab monotherapy administered Q3W (Part 1) were crossover upon disease progression and received 3.000 mg/kg feladilimab IV infusion in combination with 200 mg pembrolizumab IV infusion Q3W.
- Crossover: Fela 24 mg + Pembro 200 mg: Participants with advanced solid tumors who received feladilimab monotherapy administered Q3W (Part 1) were crossover upon disease progression and received 24 mg feladilimab IV infusion in combination with 200 mg pembrolizumab IV infusion Q3W.
- Crossover: Pembro 200 mg: Participants with advanced solid tumors who received feladilimab monotherapy administered Q3W (Part 1) were crossover upon disease progression and received 200 mg pembrolizumab IV infusion Q3W.
Period: Escalation Phase
Arm/Group | Part 1A: Feladilimab (Fela) 0.001 Milligram/Kilogram (mg/kg) | Part 1A: Fela 0.003 mg/kg | Part 1A: Fela 0.010 mg/kg | Part 1A: Fela 0.030 mg/kg | Part 1A: Fela 0.100 mg/kg | Part 1A: Fela 0.300 mg/kg | Part 1A: Fela 1.000 mg/kg | Part 1A: Fela 3.000 mg/kg | Part 1A: Fela 10.000 mg/kg | Part 1B: Fela 0.300 mg/kg | Part 1B: Fela 1.000 mg/kg | Part 1B: Fela 24 mg | Part 2A: Fela 0.010 mg/kg + Pembrolizumab (Pembro) 200 mg | Part 2A: Fela 0.030 mg/kg + Pembro 200 mg | Part 2A: Fela 0.100 mg/kg + Pembro 200 mg | Part 2A: Fela 0.300 mg/kg + Pembro 200 mg | Part 2A: Fela 1.000 mg/kg + Pembro 200 mg | Part 2A: Fela 3.000 mg/kg + Pembro 200 mg | Part 2A: Fela 8 mg + GSK3174998 8 mg | Part 2A: Fela 8 mg + GSK3174998 24 mg | Part 2A: Fela 24 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 80 mg | Part 2A: Fela 24 mg + Chemotherapy | Part 2A: Fela 80 mg + Chemotherapy | Part 2A: Fela 24 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 80 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 24 mg + Dostarlimab 500 mg + Cobolimab 300 mg | Part 2A: Fela 24 mg + Bintrafusp Alfa 2400 mg | Part 2B: Fela 0.100 mg/kg + Pembro 200 mg | Part 2B: Fela 0.300 mg/kg + Pembro 200 mg | Part 2B: Fela 1.000 mg/kg + Pembro 200 mg | Part 2B: Fela 3.000 mg/kg + Pembro 200 mg | Part 2B: Fela 24 mg + Pembro 200 mg | Part 2B: Fela 48 mg + Pembro 400 mg | Part 2B: Fela 160 mg + Pembro 400 mg | Part 2B: Fela 80 mg + Pembro 200 mg | Crossover: Fela 0.100 mg/kg + Pembro 200 mg | Crossover: Fela 0.300 mg/kg + Pembro 200 mg | Crossover: Fela 1.000 mg/kg + Pembro 200 mg | Crossover: Fela 3.000 mg/kg + Pembro 200 mg | Crossover: Fela 24 mg + Pembro 200 mg | Crossover: Pembro 200 mg
Started | 1 | 1 | 2 | 7 | 24 | 25 | 15 | 27 | 7 | 0 | 0 | 0 | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 16 | 4 | 3 | 6 | 36 | 13 | 22 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 2 | 7 | 24 | 24 | 15 | 27 | 7 | 0 | 0 | 0 | 4 | 4 | 5 | 7 | 8 | 11 | 1 | 4 | 16 | 4 | 2 | 6 | 35 | 10 | 21 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 1 | 2 | 7 | 18 | 17 | 11 | 21 | 3 | 0 | 0 | 0 | 2 | 4 | 5 | 6 | 6 | 7 | 1 | 3 | 13 | 3 | 2 | 4 | 31 | 7 | 13 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participants were crossed over OR were re-treated following progression | 0 | 0 | 0 | 0 | 5 | 2 | 2 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Site Closed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Expansion Phase
Arm/Group | Part 1A: Feladilimab (Fela) 0.001 Milligram/Kilogram (mg/kg) | Part 1A: Fela 0.003 mg/kg | Part 1A: Fela 0.010 mg/kg | Part 1A: Fela 0.030 mg/kg | Part 1A: Fela 0.100 mg/kg | Part 1A: Fela 0.300 mg/kg | Part 1A: Fela 1.000 mg/kg | Part 1A: Fela 3.000 mg/kg | Part 1A: Fela 10.000 mg/kg | Part 1B: Fela 0.300 mg/kg | Part 1B: Fela 1.000 mg/kg | Part 1B: Fela 24 mg | Part 2A: Fela 0.010 mg/kg + Pembrolizumab (Pembro) 200 mg | Part 2A: Fela 0.030 mg/kg + Pembro 200 mg | Part 2A: Fela 0.100 mg/kg + Pembro 200 mg | Part 2A: Fela 0.300 mg/kg + Pembro 200 mg | Part 2A: Fela 1.000 mg/kg + Pembro 200 mg | Part 2A: Fela 3.000 mg/kg + Pembro 200 mg | Part 2A: Fela 8 mg + GSK3174998 8 mg | Part 2A: Fela 8 mg + GSK3174998 24 mg | Part 2A: Fela 24 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 80 mg | Part 2A: Fela 24 mg + Chemotherapy | Part 2A: Fela 80 mg + Chemotherapy | Part 2A: Fela 24 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 80 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 24 mg + Dostarlimab 500 mg + Cobolimab 300 mg | Part 2A: Fela 24 mg + Bintrafusp Alfa 2400 mg | Part 2B: Fela 0.100 mg/kg + Pembro 200 mg | Part 2B: Fela 0.300 mg/kg + Pembro 200 mg | Part 2B: Fela 1.000 mg/kg + Pembro 200 mg | Part 2B: Fela 3.000 mg/kg + Pembro 200 mg | Part 2B: Fela 24 mg + Pembro 200 mg | Part 2B: Fela 48 mg + Pembro 400 mg | Part 2B: Fela 160 mg + Pembro 400 mg | Part 2B: Fela 80 mg + Pembro 200 mg | Crossover: Fela 0.100 mg/kg + Pembro 200 mg | Crossover: Fela 0.300 mg/kg + Pembro 200 mg | Crossover: Fela 1.000 mg/kg + Pembro 200 mg | Crossover: Fela 3.000 mg/kg + Pembro 200 mg | Crossover: Fela 24 mg + Pembro 200 mg | Crossover: Pembro 200 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 39 | 115 | 59 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 255 | 44 | 23 | 4 | 6 | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 14 | 2 | 3 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 38 | 112 | 56 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 241 | 42 | 20 | 4 | 3 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 25 | 69 | 48 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 202 | 31 | 17 | 2 | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 19 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participants were crossed over OR were re-treated following progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 36 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Site Closed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 4 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Crossover/ Re-treatment Phase
Arm/Group | Part 1A: Feladilimab (Fela) 0.001 Milligram/Kilogram (mg/kg) | Part 1A: Fela 0.003 mg/kg | Part 1A: Fela 0.010 mg/kg | Part 1A: Fela 0.030 mg/kg | Part 1A: Fela 0.100 mg/kg | Part 1A: Fela 0.300 mg/kg | Part 1A: Fela 1.000 mg/kg | Part 1A: Fela 3.000 mg/kg | Part 1A: Fela 10.000 mg/kg | Part 1B: Fela 0.300 mg/kg | Part 1B: Fela 1.000 mg/kg | Part 1B: Fela 24 mg | Part 2A: Fela 0.010 mg/kg + Pembrolizumab (Pembro) 200 mg | Part 2A: Fela 0.030 mg/kg + Pembro 200 mg | Part 2A: Fela 0.100 mg/kg + Pembro 200 mg | Part 2A: Fela 0.300 mg/kg + Pembro 200 mg | Part 2A: Fela 1.000 mg/kg + Pembro 200 mg | Part 2A: Fela 3.000 mg/kg + Pembro 200 mg | Part 2A: Fela 8 mg + GSK3174998 8 mg | Part 2A: Fela 8 mg + GSK3174998 24 mg | Part 2A: Fela 24 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 80 mg | Part 2A: Fela 24 mg + Chemotherapy | Part 2A: Fela 80 mg + Chemotherapy | Part 2A: Fela 24 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 80 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 24 mg + Dostarlimab 500 mg + Cobolimab 300 mg | Part 2A: Fela 24 mg + Bintrafusp Alfa 2400 mg | Part 2B: Fela 0.100 mg/kg + Pembro 200 mg | Part 2B: Fela 0.300 mg/kg + Pembro 200 mg | Part 2B: Fela 1.000 mg/kg + Pembro 200 mg | Part 2B: Fela 3.000 mg/kg + Pembro 200 mg | Part 2B: Fela 24 mg + Pembro 200 mg | Part 2B: Fela 48 mg + Pembro 400 mg | Part 2B: Fela 160 mg + Pembro 400 mg | Part 2B: Fela 80 mg + Pembro 200 mg | Crossover: Fela 0.100 mg/kg + Pembro 200 mg | Crossover: Fela 0.300 mg/kg + Pembro 200 mg | Crossover: Fela 1.000 mg/kg + Pembro 200 mg | Crossover: Fela 3.000 mg/kg + Pembro 200 mg | Crossover: Fela 24 mg + Pembro 200 mg | Crossover: Pembro 200 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (As prespecified in protocol, participants enrolled in Part 1 (GSK3359609 (feladilimab) monotherapy) upon disease progression were allowed to receive GSK3359609 (feladilimab) in combination with pembrolizumab (defined as crossover)) | 19 (As prespecified in protocol, participants enrolled in Part 1 (GSK3359609 (feladilimab) monotherapy) upon disease progression were allowed to receive GSK3359609 (feladilimab) in combination with pembrolizumab (defined as crossover)) | 42 (As prespecified in protocol, participants enrolled in Part 1 (GSK3359609 (feladilimab) monotherapy) upon disease progression were allowed to receive GSK3359609 (feladilimab) in combination with pembrolizumab (defined as crossover)) | 2 (As prespecified in protocol, participants enrolled in Part 1 (GSK3359609 (feladilimab) monotherapy) upon disease progression were allowed to receive GSK3359609 (feladilimab) in combination with pembrolizumab (defined as crossover)) | 1 (As prespecified in protocol, participants enrolled in Part 1 (GSK3359609 (feladilimab) monotherapy) upon disease progression were allowed to receive GSK3359609 (feladilimab) in combination with pembrolizumab (defined as crossover)) | 1 (As prespecified in protocol, participants enrolled in Part 1 (GSK3359609 (feladilimab) monotherapy) upon disease progression were allowed to receive GSK3359609 (feladilimab) in combination with pembrolizumab (defined as crossover))
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 19 | 39 | 2 | 1 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 14 | 32 | 2 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Not completed — Site Closed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1A: Feladilimab (Fela) 0.001 Milligram/Kilogram (mg/kg) | Part 1A: Fela 0.003 mg/kg | Part 1A: Fela 0.010 mg/kg | Part 1A: Fela 0.030 mg/kg | Part 1A: Fela 0.100 mg/kg | Part 1A: Fela 0.300 mg/kg | Part 1A: Fela 1.000 mg/kg | Part 1A: Fela 3.000 mg/kg | Part 1A: Fela 10.000 mg/kg | Part 1B: Fela 0.300 mg/kg | Part 1B: Fela 1.000 mg/kg | Part 1B: Fela 24 mg | Part 2A: Fela 0.010 mg/kg + Pembrolizumab (Pembro) 200 mg | Part 2A: Fela 0.030 mg/kg + Pembro 200 mg | Part 2A: Fela 0.100 mg/kg + Pembro 200 mg | Part 2A: Fela 0.300 mg/kg + Pembro 200 mg | Part 2A: Fela 1.000 mg/kg + Pembro 200 mg | Part 2A: Fela 3.000 mg/kg + Pembro 200 mg | Part 2A: Fela 8 mg + GSK3174998 8 mg | Part 2A: Fela 8 mg + GSK3174998 24 mg | Part 2A: Fela 24 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 80 mg | Part 2A: Fela 24 mg + Chemotherapy | Part 2A: Fela 80 mg + Chemotherapy | Part 2A: Fela 24 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 80 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 24 mg + Dostarlimab 500 mg + Cobolimab 300 mg | Part 2A: Fela 24 mg + Bintrafusp Alfa 2400 mg | Part 2B: Fela 0.100 mg/kg + Pembro 200 mg | Part 2B: Fela 0.300 mg/kg + Pembro 200 mg | Part 2B: Fela 1.000 mg/kg + Pembro 200 mg | Part 2B: Fela 3.000 mg/kg + Pembro 200 mg | Part 2B: Fela 24 mg + Pembro 200 mg | Part 2B: Fela 48 mg + Pembro 400 mg | Part 2B: Fela 160 mg + Pembro 400 mg | Part 2B: Fela 80 mg + Pembro 200 mg | Total
Number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 15 | 27 | 7 | 39 | 115 | 59 | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 16 | 4 | 3 | 6 | 36 | 13 | 22 | 1 | 4 | 14 | 255 | 44 | 23 | 4 | 6 | 5 | 1 | 829
Age, Customized [Count of Participants; unit: Participants]
  18 - 93 years | 1 | 1 | 2 | 7 | 24 | 25 | 15 | 27 | 7 | 39 | 115 | 59 | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 16 | 4 | 3 | 6 | 36 | 13 | 22 | 1 | 4 | 14 | 255 | 44 | 23 | 4 | 6 | 5 | 1 | 829
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 4 | 11 | 14 | 4 | 11 | 2 | 18 | 47 | 25 | 1 | 2 | 2 | 3 | 4 | 5 | 0 | 1 | 8 | 0 | 3 | 1 | 13 | 1 | 5 | 0 | 0 | 2 | 115 | 15 | 4 | 0 | 0 | 2 | 0 | 325
  Male | 0 | 1 | 1 | 3 | 13 | 11 | 11 | 16 | 5 | 21 | 68 | 34 | 4 | 3 | 3 | 5 | 7 | 6 | 1 | 3 | 8 | 4 | 0 | 5 | 23 | 12 | 17 | 1 | 4 | 12 | 140 | 29 | 19 | 4 | 6 | 3 | 1 | 504
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  HISPANIC OR LATINO | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 4 | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 8 | 1 | 1 | 1 | 0 | 0 | 1 | 33
  NOT HISPANIC OR LATINO | 1 | 1 | 2 | 7 | 22 | 22 | 14 | 23 | 7 | 33 | 98 | 55 | 4 | 4 | 5 | 8 | 10 | 11 | 0 | 3 | 15 | 3 | 2 | 5 | 34 | 11 | 21 | 1 | 4 | 11 | 226 | 39 | 15 | 3 | 5 | 5 | 0 | 730
  Missing | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 3 | 0 | 4 | 13 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 21 | 4 | 7 | 0 | 1 | 0 | 0 | 66

OUTCOME MEASURES:

1. Primary Outcome: Part 1A: Number of Participants With Any Adverse Event(s) (AEs) and Serious Adverse Event(s) (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, or is a congenital anomaly/birth defect, other situations which involve medical or scientific judgment or is associated with liver injury and impaired liver function. SAEs are subset of AEs. A summary of number of participants with any AEs and SAEs is presented. AEs were coded using the Medical Dictionary for Regulatory Affairs (MedDRA dictionary).
Time Frame: Up to approximately 367 weeks
Population: All Treated population included all participants who received at least one dose of feladilimab.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: Feladilimab (Fela) 0.001 Milligram/Kilogram (mg/kg) | Part 1A: Fela 0.003 mg/kg | Part 1A: Fela 0.010 mg/kg | Part 1A: Fela 0.030 mg/kg | Part 1A: Fela 0.100 mg/kg | Part 1A: Fela 0.300 mg/kg | Part 1A: Fela 1.000 mg/kg | Part 1A: Fela 3.000 mg/kg | Part 1A: Fela 10.000 mg/kg
Number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 15 | 27 | 7
Participants
  Any AEs | 1 | 1 | 2 | 7 | 22 | 24 | 13 | 21 | 6
  Any SAEs | 0 | 0 | 1 | 2 | 6 | 8 | 4 | 12 | 1

2. Primary Outcome: Part 1A: Number of Participants With Dose Limiting Toxicity (DLT)
Description: DLT is an AE that is considered by the investigator to be clinically relevant and attributed to the study therapy during the 28-day DLT period and meets at least one of the DLT criteria: Febrile neutropenia; Grade 4 neutropenia of >7 days in duration or requiring Granulocyte Colony-stimulating Factor (G-CSF), anemia, thrombocytopenia, non-hematologic toxicity; Grade 3 thrombocytopenia with bleeding, pneumonitis, toxicity that does not resolve to Grade 1 or baseline within 3 days; Grade 2 ocular toxicity; Toxicity that results in permanent discontinuation of feladilimab during the first four weeks of treatment; any other event which in the judgment of the investigator and GSK Medical Monitor is considered to be a DLT.
Time Frame: Up to 28 days
Population: DLT Evaluable Population included All Treated Population in the dose escalation phase or PK/PD cohorts, who completed the 28-day DLT observation period or experienced a DLT during the determinative period (28 days).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: Feladilimab (Fela) 0.001 Milligram/Kilogram (mg/kg) | Part 1A: Fela 0.003 mg/kg | Part 1A: Fela 0.010 mg/kg | Part 1A: Fela 0.030 mg/kg | Part 1A: Fela 0.100 mg/kg | Part 1A: Fela 0.300 mg/kg | Part 1A: Fela 1.000 mg/kg | Part 1A: Fela 3.000 mg/kg | Part 1A: Fela 10.000 mg/kg
Number analyzed (Participants) | 1 | 1 | 2 | 3 | 5 | 9 | 9 | 7 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

3. Primary Outcome: Part 1A: Number of Participants With Worst-case Grade Change From Baseline in Clinical Chemistry Parameters
Description: Blood samples were collected for analysis of clinical chemistry parameters. Laboratory parameters were graded according to CTCAE v4.03. Grade (G) 0: None; G1: mild; G2: moderate; G3: severe or medically significant; G4: life-threatening consequences. Higher grade indicates greater severity and increase in grade was defined relative to Baseline grade. Baseline (Day 1) was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Only grade change data is presented for Baseline (B) and Worst-Case Post-Baseline (WCPB) as G0, G1, G2, G3, G4, and missing (M) here as "Parameter name, B GX, WCPB GX" where X=grade digit.
Time Frame: Baseline (Day 1) and up to approximately 367 weeks
Population: All Treated Population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: Feladilimab (Fela) 0.001 Milligram/Kilogram (mg/kg) | Part 1A: Fela 0.003 mg/kg | Part 1A: Fela 0.010 mg/kg | Part 1A: Fela 0.030 mg/kg | Part 1A: Fela 0.100 mg/kg | Part 1A: Fela 0.300 mg/kg | Part 1A: Fela 1.000 mg/kg | Part 1A: Fela 3.000 mg/kg | Part 1A: Fela 10.000 mg/kg
Number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 15 | 27 | 7
Participants
  Hypoglycemia , Grade 0, Grade 1 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 1 | 0
  Hypoglycemia , Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Hypoglycemia , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 0, Grade 1 | 0 | 1 | 0 | 1 | 10 | 5 | 7 | 11 | 1
  Hyperglycemia , Grade 0, Grade 2 | 0 | 0 | 0 | 2 | 1 | 3 | 2 | 1 | 0
  Hyperglycemia , Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Hyperglycemia , Grade 1, Grade 2 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1
  Hyperglycemia , Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Hyperglycemia , Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Hyperglycemia , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 0, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypoalbuminemia , Grade 0, Grade 1 | 1 | 0 | 1 | 3 | 6 | 5 | 6 | 9 | 1
  Hypoalbuminemia , Grade 0, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypoalbuminemia , Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 6 | 1 | 1 | 0 | 1
  Hypoalbuminemia , Grade 0, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypoalbuminemia , Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 0, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypoalbuminemia , Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 1, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypoalbuminemia , Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 1, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypoalbuminemia , Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 1 | 0
  Hypoalbuminemia , Grade 1, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypoalbuminemia , Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 1, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypoalbuminemia , Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 2, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypoalbuminemia , Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 2, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypoalbuminemia , Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 2, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypoalbuminemia , Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 2, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypoalbuminemia , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 3, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypoalbuminemia , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 3, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypoalbuminemia , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 3, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypoalbuminemia , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 3, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypoalbuminemia , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 4, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypoalbuminemia , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 4, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypoalbuminemia , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 4, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypoalbuminemia , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 4, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypoalbuminemia , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 0, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AP Increased, Grade 0, Grade 1 | 0 | 0 | 0 | 2 | 4 | 6 | 4 | 3 | 2
  AP Increased, Grade 0, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AP Increased, Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  AP Increased, Grade 0, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AP Increased, Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  AP Increased, Grade 0, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AP Increased, Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 1, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AP Increased, Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 1, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AP Increased, Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
  AP Increased, Grade 1, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AP Increased, Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  AP Increased, Grade 1, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AP Increased, Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 2, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AP Increased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 2, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AP Increased, Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  AP Increased, Grade 2, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AP Increased, Grade 2, Grade 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  AP Increased, Grade 2, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AP Increased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 3, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AP Increased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 3, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AP Increased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 3, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AP Increased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 3, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AP Increased, Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  AP Increased, Grade 4, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AP Increased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 4, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AP Increased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 4, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AP Increased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 4, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AP Increased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 0, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  ALT Increased, Grade 0, Grade 1 | 0 | 0 | 0 | 1 | 3 | 0 | 3 | 5 | 0
  ALT Increased, Grade 0, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  ALT Increased, Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  ALT Increased, Grade 0, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  ALT Increased, Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  ALT Increased, Grade 0, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  ALT Increased, Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  ALT Increased, Grade 1, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  ALT Increased, Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  ALT Increased, Grade 1, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  ALT Increased, Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  ALT Increased, Grade 1, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  ALT Increased, Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 1, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  ALT Increased, Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 2, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  ALT Increased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 2, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  ALT Increased, Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 2, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  ALT Increased, Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 2, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  ALT Increased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 3, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  ALT Increased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 3, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  ALT Increased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 3, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  ALT Increased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 3, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  ALT Increased, Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 4, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  ALT Increased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 4, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  ALT Increased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 4, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  ALT Increased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 4, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  ALT Increased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 0, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AST Increased, Grade 0, Grade 1 | 0 | 0 | 0 | 2 | 5 | 4 | 3 | 9 | 1
  AST Increased, Grade 0, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AST Increased, Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
  AST Increased, Grade 0, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AST Increased, Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  AST Increased, Grade 0, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AST Increased, Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  AST Increased, Grade 1, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AST Increased, Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  AST Increased, Grade 1, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AST Increased, Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 1, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AST Increased, Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  AST Increased, Grade 1, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AST Increased, Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 2, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AST Increased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 2, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AST Increased, Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 2, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AST Increased, Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  AST Increased, Grade 2, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AST Increased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 3, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AST Increased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 3, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AST Increased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 3, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AST Increased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 3, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AST Increased, Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 4, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AST Increased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 4, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AST Increased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 4, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AST Increased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 4, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  AST Increased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 0, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Blood Bilirubin Increased, Grade 0, Grade 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
  Blood Bilirubin Increased, Grade 0, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Blood Bilirubin Increased, Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
  Blood Bilirubin Increased, Grade 0, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Blood Bilirubin Increased, Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Blood Bilirubin Increased, Grade 0, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Blood Bilirubin Increased, Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 1, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Blood Bilirubin Increased, Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Blood Bilirubin Increased, Grade 1, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Blood Bilirubin Increased, Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 1, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Blood Bilirubin Increased, Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 1, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Blood Bilirubin Increased, Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 2, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Blood Bilirubin Increased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 2, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Blood Bilirubin Increased, Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 2, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Blood Bilirubin Increased, Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 2, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Blood Bilirubin Increased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 3, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Blood Bilirubin Increased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 3, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Blood Bilirubin Increased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 3, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Blood Bilirubin Increased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 3, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Blood Bilirubin Increased, Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 4, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Blood Bilirubin Increased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 4, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Blood Bilirubin Increased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 4, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Blood Bilirubin Increased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 4, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Blood Bilirubin Increased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 0, Grade 1 | 0 | 0 | 0 | 1 | 6 | 2 | 2 | 2 | 4
  Creatinine Increased, Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Creatinine Increased, Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 0, Grade 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 0
  Hypokalemia , Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Missing, Grade 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Hypokalemia , Missing, Grade 0 |  |  |  |  | 1 |  |  |  |
  Hypokalemia , Missing, Grade 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Hypokalemia , Missing, Grade 1 |  |  |  |  | 0 |  |  |  |
  Hypokalemia , Missing, Grade 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Hypokalemia , Missing, Grade 2 |  |  |  |  | 0 |  |  |  |
  Hypokalemia , Missing, Grade 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Hypokalemia , Missing, Grade 3 |  |  |  |  | 0 |  |  |  |
  Hypokalemia , Missing, Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Hypokalemia , Missing, Grade 4 |  |  |  |  | 0 |  |  |  |
  Hyperkalemia , Grade 0, Grade 1 | 0 | 1 | 0 | 2 | 5 | 7 | 4 | 6 | 1
  Hyperkalemia , Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Hyperkalemia , Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Hyperkalemia , Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Missing, Grade 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Hyperkalemia , Missing, Grade 0 |  |  |  |  | 1 |  |  |  |
  Hyperkalemia , Missing, Grade 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Hyperkalemia , Missing, Grade 1 |  |  |  |  | 0 |  |  |  |
  Hyperkalemia , Missing, Grade 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Hyperkalemia , Missing, Grade 2 |  |  |  |  | 0 |  |  |  |
  Hyperkalemia , Missing, Grade 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Hyperkalemia , Missing, Grade 3 |  |  |  |  | 0 |  |  |  |
  Hyperkalemia , Missing, Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Hyperkalemia , Missing, Grade 4 |  |  |  |  | 0 |  |  |  |
  Hyponatremia , Grade 0, Grade 1 | 0 | 0 | 1 | 3 | 3 | 7 | 3 | 3 | 0
  Hyponatremia , Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
  Hyponatremia , Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 0, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Hypernatremia , Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Hypernatremia , Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 0, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypocalcemia , Grade 0, Grade 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 3 | 0
  Hypocalcemia , Grade 0, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypocalcemia , Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 0, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypocalcemia , Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 0, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypocalcemia , Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Hypocalcemia , Grade 1, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypocalcemia , Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 1, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypocalcemia , Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 1, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypocalcemia , Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 1, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypocalcemia , Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 2, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypocalcemia , Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Hypocalcemia , Grade 2, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypocalcemia , Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 2, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypocalcemia , Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 2, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypocalcemia , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 3, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypocalcemia , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 3, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypocalcemia , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 3, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypocalcemia , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 3, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypocalcemia , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 4, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypocalcemia , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 4, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypocalcemia , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 4, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypocalcemia , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 4, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypocalcemia , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Missing, Grade 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Hypocalcemia , Missing, Grade 0 |  |  |  |  | 1 |  |  |  |
  Hypocalcemia , Missing, Grade 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Hypocalcemia , Missing, Grade 1 |  |  |  |  | 0 |  |  |  |
  Hypocalcemia , Missing, Grade 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Hypocalcemia , Missing, Grade 2 |  |  |  |  | 0 |  |  |  |
  Hypocalcemia , Missing, Grade 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Hypocalcemia , Missing, Grade 3 |  |  |  |  | 0 |  |  |  |
  Hypocalcemia , Missing, Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Hypocalcemia , Missing, Grade 4 |  |  |  |  | 0 |  |  |  |
  Hypercalcemia , Grade 0, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypercalcemia , Grade 0, Grade 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Hypercalcemia , Grade 0, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypercalcemia , Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 0, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypercalcemia , Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 0, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypercalcemia , Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 1, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypercalcemia , Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Hypercalcemia , Grade 1, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypercalcemia , Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 1, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypercalcemia , Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Hypercalcemia , Grade 1, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypercalcemia , Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 2, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypercalcemia , Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 2, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypercalcemia , Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 2, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypercalcemia , Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 2, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypercalcemia , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 3, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypercalcemia , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 3, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypercalcemia , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 3, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypercalcemia , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 3, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypercalcemia , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 4, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypercalcemia , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 4, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypercalcemia , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 4, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypercalcemia , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 4, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Hypercalcemia , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Missing, Grade 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Hypercalcemia , Missing, Grade 0 |  |  |  |  | 0 |  |  |  |
  Hypercalcemia , Missing, Grade 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Hypercalcemia , Missing, Grade 1 |  |  |  |  | 1 |  |  |  |
  Hypercalcemia , Missing, Grade 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Hypercalcemia , Missing, Grade 2 |  |  |  |  | 0 |  |  |  |
  Hypercalcemia , Missing, Grade 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Hypercalcemia , Missing, Grade 3 |  |  |  |  | 0 |  |  |  |
  Hypercalcemia , Missing, Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Hypercalcemia , Missing, Grade 4 |  |  |  |  | 0 |  |  |  |
  Chronic Kidney Disease , Grade 0, Grade 1: number analyzed (Participants) | 0 | 0 | 0 | 2 | 9 | 6 | 2 | 7 | 2
  Chronic Kidney Disease , Grade 0, Grade 1 |  |  |  | 0 | 1 | 0 | 0 | 0 | 0
  Chronic Kidney Disease , Grade 0, Grade 2: number analyzed (Participants) | 0 | 0 | 0 | 2 | 9 | 6 | 2 | 7 | 2
  Chronic Kidney Disease , Grade 0, Grade 2 |  |  |  | 0 | 0 | 0 | 1 | 0 | 0
  Chronic Kidney Disease , Grade 0, Grade 3: number analyzed (Participants) | 0 | 0 | 0 | 2 | 9 | 6 | 2 | 7 | 2
  Chronic Kidney Disease , Grade 0, Grade 3 |  |  |  | 0 | 0 | 0 | 0 | 0 | 0
  Chronic Kidney Disease , Grade 0, Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 2 | 9 | 6 | 2 | 7 | 2
  Chronic Kidney Disease , Grade 0, Grade 4 |  |  |  | 0 | 0 | 0 | 0 | 0 | 0
  Chronic Kidney Disease , Grade 1, Grade 0: number analyzed (Participants) | 0 | 0 | 0 | 2 | 9 | 6 | 2 | 7 | 2
  Chronic Kidney Disease , Grade 1, Grade 0 |  |  |  | 0 | 0 | 0 | 0 | 0 | 0
  Chronic Kidney Disease , Grade 1, Grade 2: number analyzed (Participants) | 0 | 0 | 0 | 2 | 9 | 6 | 2 | 7 | 2
  Chronic Kidney Disease , Grade 1, Grade 2 |  |  |  | 1 | 3 | 0 | 0 | 0 | 1
  Chronic Kidney Disease , Grade 1, Grade 3: number analyzed (Participants) | 0 | 0 | 0 | 2 | 9 | 6 | 2 | 7 | 2
  Chronic Kidney Disease , Grade 1, Grade 3 |  |  |  | 0 | 0 | 0 | 0 | 0 | 0
  Chronic Kidney Disease , Grade 1, Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 2 | 9 | 6 | 2 | 7 | 2
  Chronic Kidney Disease , Grade 1, Grade 4 |  |  |  | 0 | 0 | 0 | 0 | 0 | 0
  Chronic Kidney Disease , Grade 2, Grade 0: number analyzed (Participants) | 0 | 0 | 0 | 2 | 9 | 6 | 2 | 7 | 2
  Chronic Kidney Disease , Grade 2, Grade 0 |  |  |  | 0 | 0 | 0 | 0 | 0 | 0
  Chronic Kidney Disease , Grade 2, Grade 1: number analyzed (Participants) | 0 | 0 | 0 | 2 | 9 | 6 | 2 | 7 | 2
  Chronic Kidney Disease , Grade 2, Grade 1 |  |  |  | 0 | 0 | 0 | 0 | 0 | 0
  Chronic Kidney Disease , Grade 2, Grade 3: number analyzed (Participants) | 0 | 0 | 0 | 2 | 9 | 6 | 2 | 7 | 2
  Chronic Kidney Disease , Grade 2, Grade 3 |  |  |  | 0 | 0 | 0 | 0 | 0 | 0
  Chronic Kidney Disease , Grade 2, Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 2 | 9 | 6 | 2 | 7 | 2
  Chronic Kidney Disease , Grade 2, Grade 4 |  |  |  | 0 | 0 | 0 | 0 | 0 | 0
  Chronic Kidney Disease , Grade 3, Grade 0: number analyzed (Participants) | 0 | 0 | 0 | 2 | 9 | 6 | 2 | 7 | 2
  Chronic Kidney Disease , Grade 3, Grade 0 |  |  |  | 0 | 0 | 0 | 0 | 0 | 0
  Chronic Kidney Disease , Grade 3, Grade 1: number analyzed (Participants) | 0 | 0 | 0 | 2 | 9 | 6 | 2 | 7 | 2
  Chronic Kidney Disease , Grade 3, Grade 1 |  |  |  | 0 | 0 | 0 | 0 | 0 | 0
  Chronic Kidney Disease , Grade 3, Grade 2: number analyzed (Participants) | 0 | 0 | 0 | 2 | 9 | 6 | 2 | 7 | 2
  Chronic Kidney Disease , Grade 3, Grade 2 |  |  |  | 0 | 0 | 0 | 0 | 0 | 0
  Chronic Kidney Disease , Grade 3, Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 2 | 9 | 6 | 2 | 7 | 2
  Chronic Kidney Disease , Grade 3, Grade 4 |  |  |  | 0 | 0 | 0 | 0 | 0 | 0
  Chronic Kidney Disease , Grade 4, Grade 0: number analyzed (Participants) | 0 | 0 | 0 | 2 | 9 | 6 | 2 | 7 | 2
  Chronic Kidney Disease , Grade 4, Grade 0 |  |  |  | 0 | 0 | 0 | 0 | 0 | 0
  Chronic Kidney Disease , Grade 4, Grade 1: number analyzed (Participants) | 0 | 0 | 0 | 2 | 9 | 6 | 2 | 7 | 2
  Chronic Kidney Disease , Grade 4, Grade 1 |  |  |  | 0 | 0 | 0 | 0 | 0 | 0
  Chronic Kidney Disease , Grade 4, Grade 2: number analyzed (Participants) | 0 | 0 | 0 | 2 | 9 | 6 | 2 | 7 | 2
  Chronic Kidney Disease , Grade 4, Grade 2 |  |  |  | 0 | 0 | 0 | 0 | 0 | 0
  Chronic Kidney Disease , Grade 4, Grade 3: number analyzed (Participants) | 0 | 0 | 0 | 2 | 9 | 6 | 2 | 7 | 2
  Chronic Kidney Disease , Grade 4, Grade 3 |  |  |  | 0 | 0 | 0 | 0 | 0 | 0
  Chronic Kidney Disease , Missing, Grade 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 6 | 0 | 7 | 0
  Chronic Kidney Disease , Missing, Grade 0 |  |  |  |  | 0 | 1 |  | 1 |
  Chronic Kidney Disease , Missing, Grade 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 6 | 0 | 7 | 0
  Chronic Kidney Disease , Missing, Grade 1 |  |  |  |  | 1 | 1 |  | 0 |
  Chronic Kidney Disease , Missing, Grade 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 6 | 0 | 7 | 0
  Chronic Kidney Disease , Missing, Grade 2 |  |  |  |  | 0 | 0 |  | 1 |
  Chronic Kidney Disease , Missing, Grade 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 6 | 0 | 7 | 0
  Chronic Kidney Disease , Missing, Grade 3 |  |  |  |  | 0 | 0 |  | 0 |
  Chronic Kidney Disease , Missing, Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 6 | 0 | 7 | 0
  Chronic Kidney Disease , Missing, Grade 4 |  |  |  |  | 0 | 1 |  | 0 |

4. Primary Outcome: Part 1A: Number of Participants With Worst Case Chemistry Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Normal ranges were 0.1 to 0.3 micromoles (umol)/liter (L) (direct bilirubin); 6 to 8.3 grams/L (protein); 100 to 250 international units (IU)/L (Lactate Dehydrogenase(LDH)); 2.3 - 4.1 picomoles/L (Free Triiodothyronine(T3)); 4.6 to 11.2 picomoles/L (Free Thyroxine(T4)); 0 and 0.04 microgram (ug)/L (Troponin I); 0 - 0.01 ug/L (Troponin T); 0.45 to 4.5 milliunits (Mu)/L (Thyrotropin(TSH)); and 6 to 24 millimoles/L (Urea). Participants were counted in worst case category that their value changes to low, normal or no change [NC] or high), unless there is NC in their category. Participants whose laboratory value category was unchanged (e.g. High to High) or whose value became normal, were recorded in "To Normal or No Change" category. Participants were counted twice if participant had values that changed To Low and To High, so percentages may not add to 100%.
Time Frame: Up to approximately 367 weeks
Population: All Treated Population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: Feladilimab (Fela) 0.001 Milligram/Kilogram (mg/kg) | Part 1A: Fela 0.003 mg/kg | Part 1A: Fela 0.010 mg/kg | Part 1A: Fela 0.030 mg/kg | Part 1A: Fela 0.100 mg/kg | Part 1A: Fela 0.300 mg/kg | Part 1A: Fela 1.000 mg/kg | Part 1A: Fela 3.000 mg/kg | Part 1A: Fela 10.000 mg/kg
Number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 15 | 27 | 7
Participants
  Direct Bilirubin (umol/L), To Low: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Direct Bilirubin (umol/L), To Low |  |  |  |  | 0 |  |  |  |
  Direct Bilirubin (umol/L), To Normal or No Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Direct Bilirubin (umol/L), To Normal or No Change |  |  |  |  | 0 |  |  |  |
  Direct Bilirubin (umol/L), To High: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Direct Bilirubin (umol/L), To High |  |  |  |  | 1 |  |  |  |
  Lactate Dehydrogenase (IU/L), To Low: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0
  Lactate Dehydrogenase (IU/L), To Low |  |  |  |  | 0 | 0 | 0 |  |
  Lactate Dehydrogenase (IU/L), To Normal or No Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0
  Lactate Dehydrogenase (IU/L), To Normal or No Change |  |  |  |  | 0 | 0 | 0 |  |
  Lactate Dehydrogenase (IU/L), To High: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0
  Lactate Dehydrogenase (IU/L), To High |  |  |  |  | 1 | 2 | 1 |  |
  Protein (g/L), To Low: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Protein (g/L), To Low | 0 | 0 | 0 | 2 | 6 | 7 | 1 | 3 | 1
  Protein (g/L), To Normal or No Change: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Protein (g/L), To Normal or No Change | 1 | 1 | 2 | 5 | 18 | 15 | 9 | 21 | 5
  Protein (g/L), To High: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Protein (g/L), To High | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 4 | 1
  Triiodothyronine, Free (pmol/L), To Low: number analyzed (Participants) | 1 | 1 | 1 | 7 | 19 | 23 | 11 | 23 | 7
  Triiodothyronine, Free (pmol/L), To Low | 0 | 0 | 0 | 3 | 5 | 6 | 2 | 2 | 1
  Triiodothyronine, Free (pmol/L), To Normal or No Change: number analyzed (Participants) | 1 | 1 | 1 | 7 | 19 | 23 | 11 | 23 | 7
  Triiodothyronine, Free (pmol/L), To Normal or No Change | 1 | 1 | 0 | 4 | 12 | 16 | 8 | 21 | 5
  Triiodothyronine, Free (pmol/L), To High: number analyzed (Participants) | 1 | 1 | 1 | 7 | 19 | 23 | 11 | 23 | 7
  Triiodothyronine, Free (pmol/L), To High | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 1
  Thyroxine, Free (pmol/L), To Low: number analyzed (Participants) | 1 | 1 | 1 | 7 | 19 | 24 | 11 | 23 | 7
  Thyroxine, Free (pmol/L), To Low | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Thyroxine, Free (pmol/L), To Normal or No Change: number analyzed (Participants) | 1 | 1 | 1 | 7 | 19 | 24 | 11 | 23 | 7
  Thyroxine, Free (pmol/L), To Normal or No Change | 1 | 1 | 1 | 6 | 19 | 21 | 10 | 22 | 5
  Thyroxine, Free (pmol/L), To High: number analyzed (Participants) | 1 | 1 | 1 | 7 | 19 | 24 | 11 | 23 | 7
  Thyroxine, Free (pmol/L), To High | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 1
  Troponin I (ug/L), To Low: number analyzed (Participants) | 1 | 0 | 1 | 4 | 8 | 10 | 2 | 8 | 3
  Troponin I (ug/L), To Low | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Troponin I (ug/L), To Normal or No Change: number analyzed (Participants) | 1 | 0 | 1 | 4 | 8 | 10 | 2 | 8 | 3
  Troponin I (ug/L), To Normal or No Change | 1 |  | 1 | 3 | 6 | 10 | 1 | 8 | 2
  Troponin I (ug/L), To High: number analyzed (Participants) | 1 | 0 | 1 | 4 | 8 | 10 | 2 | 8 | 3
  Troponin I (ug/L), To High | 0 |  | 0 | 1 | 2 | 0 | 1 | 0 | 1
  Troponin T (ug/L), To Low: number analyzed (Participants) | 0 | 0 | 0 | 0 | 11 | 8 | 9 | 13 | 2
  Troponin T (ug/L), To Low |  |  |  |  | 0 | 0 | 0 | 0 | 0
  Troponin T (ug/L), To Normal or No Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 11 | 8 | 9 | 13 | 2
  Troponin T (ug/L), To Normal or No Change |  |  |  |  | 8 | 8 | 8 | 10 | 2
  Troponin T (ug/L), To High: number analyzed (Participants) | 0 | 0 | 0 | 0 | 11 | 8 | 9 | 13 | 2
  Troponin T (ug/L), To High |  |  |  |  | 3 | 0 | 1 | 3 | 0
  Thyrotropin (mU/L), To Low: number analyzed (Participants) | 1 | 1 | 1 | 7 | 19 | 24 | 11 | 23 | 7
  Thyrotropin (mU/L), To Low | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
  Thyrotropin (mU/L), To Normal or No Change: number analyzed (Participants) | 1 | 1 | 1 | 7 | 19 | 24 | 11 | 23 | 7
  Thyrotropin (mU/L), To Normal or No Change | 1 | 1 | 1 | 5 | 18 | 21 | 10 | 20 | 7
  Thyrotropin (mU/L), To High: number analyzed (Participants) | 1 | 1 | 1 | 7 | 19 | 24 | 11 | 23 | 7
  Thyrotropin (mU/L), To High | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 2 | 0
  Urea (mmol/L), To Low: number analyzed (Participants) | 1 | 1 | 2 | 6 | 18 | 19 | 12 | 21 | 5
  Urea (mmol/L), To Low | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 0
  Urea (mmol/L), To Normal or No Change: number analyzed (Participants) | 1 | 1 | 2 | 6 | 18 | 19 | 12 | 21 | 5
  Urea (mmol/L), To Normal or No Change | 1 | 0 | 1 | 3 | 12 | 11 | 7 | 15 | 2
  Urea (mmol/L), To High: number analyzed (Participants) | 1 | 1 | 2 | 6 | 18 | 19 | 12 | 21 | 5
  Urea (mmol/L), To High | 0 | 1 | 1 | 3 | 6 | 6 | 3 | 6 | 3

5. Primary Outcome: Part 1A: Number of Participants With Worst-case Grade Change From Baseline in Hematology Parameters
Description: Blood samples were collected for analysis of hematology parameters. Laboratory parameters were graded according to CTCAE v4.03. Grade (G) 0: None; G1: mild; G2: moderate; G3: severe or medically significant; G4: life-threatening consequences. Higher grade indicates greater severity and increase in grade was defined relative to Baseline grade. Baseline (Day 1) was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Only grade change data is presented for Baseline (B) and Worst-Case Post-Baseline (WCPB) as G0, G1, G2, G3, G4, and missing (M) here as "Parameter name, B GX, WCPB GX" where X=grade digit.
Time Frame: Baseline (Day 1) and up to approximately 367 weeks
Population: All Treated Population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: Feladilimab (Fela) 0.001 Milligram/Kilogram (mg/kg) | Part 1A: Fela 0.003 mg/kg | Part 1A: Fela 0.010 mg/kg | Part 1A: Fela 0.030 mg/kg | Part 1A: Fela 0.100 mg/kg | Part 1A: Fela 0.300 mg/kg | Part 1A: Fela 1.000 mg/kg | Part 1A: Fela 3.000 mg/kg | Part 1A: Fela 10.000 mg/kg
Number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 15 | 27 | 7
Participants
  Anemia , Grade 0, Grade 1 | 1 | 0 | 0 | 3 | 8 | 1 | 2 | 6 | 1
  Anemia , Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
  Anemia , Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Anemia , Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 1, Grade 2 | 0 | 0 | 1 | 1 | 4 | 5 | 2 | 3 | 2
  Anemia , Grade 1, Grade 3 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
  Anemia , Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0
  Anemia , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 0, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hemoglobin Increased, Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 0, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Decreased, Grade 0, Grade 1 | 1 | 0 | 0 | 1 | 5 | 5 | 2 | 6 | 3
  Lymphocyte Count Decreased, Grade 0, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Decreased, Grade 0, Grade 2 | 0 | 0 | 0 | 1 | 3 | 3 | 2 | 2 | 0
  Lymphocyte Count Decreased, Grade 0, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Decreased, Grade 0, Grade 3 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0
  Lymphocyte Count Decreased, Grade 0, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Decreased, Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 1, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Decreased, Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 1, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Decreased, Grade 1, Grade 2 | 0 | 0 | 1 | 0 | 5 | 2 | 1 | 1 | 1
  Lymphocyte Count Decreased, Grade 1, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Decreased, Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0
  Lymphocyte Count Decreased, Grade 1, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Decreased, Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 2, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Decreased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Lymphocyte Count Decreased, Grade 2, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Decreased, Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 2, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Decreased, Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0
  Lymphocyte Count Decreased, Grade 2, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Decreased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 3, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Decreased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 3, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Decreased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 3, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Decreased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 3, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Decreased, Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 4, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Decreased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 4, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Decreased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 4, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Decreased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 4, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Decreased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Missing, Grade 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Missing, Grade 0 |  |  |  |  | 0 |  |  |  |
  Lymphocyte Count Decreased, Missing, Grade 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Missing, Grade 1 |  |  |  |  | 0 |  |  |  |
  Lymphocyte Count Decreased, Missing, Grade 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Missing, Grade 2 |  |  |  |  | 0 |  |  |  |
  Lymphocyte Count Decreased, Missing, Grade 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Missing, Grade 3 |  |  |  |  | 1 |  |  |  |
  Lymphocyte Count Decreased, Missing, Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Missing, Grade 4 |  |  |  |  | 0 |  |  |  |
  Lymphocyte Count Increased, Grade 0, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Increased, Grade 0, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 0, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Increased, Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0
  Lymphocyte Count Increased, Grade 0, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Increased, Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 0, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Increased, Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 1, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Increased, Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 1, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Increased, Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 1, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Increased, Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 1, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Increased, Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 2, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Increased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 2, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Increased, Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 2, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Increased, Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 2, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Increased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 3, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Increased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 3, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Increased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 3, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Increased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 3, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Increased, Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 4, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Increased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 4, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Increased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 4, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Increased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 4, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Lymphocyte Count Increased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Missing, Grade 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Missing, Grade 0 |  |  |  |  | 1 |  |  |  |
  Lymphocyte Count Increased, Missing, Grade 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Missing, Grade 1 |  |  |  |  | 0 |  |  |  |
  Lymphocyte Count Increased, Missing, Grade 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Missing, Grade 2 |  |  |  |  | 0 |  |  |  |
  Lymphocyte Count Increased, Missing, Grade 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Missing, Grade 3 |  |  |  |  | 0 |  |  |  |
  Lymphocyte Count Increased, Missing, Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Missing, Grade 4 |  |  |  |  | 0 |  |  |  |
  Neutrophil Count Decreased, Grade 0, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Neutrophil Count Decreased, Grade 0, Grade 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1
  Neutrophil Count Decreased, Grade 0, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Neutrophil Count Decreased, Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 0, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Neutrophil Count Decreased, Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Neutrophil Count Decreased, Grade 0, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Neutrophil Count Decreased, Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Neutrophil Count Decreased, Grade 1, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Neutrophil Count Decreased, Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 1, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Neutrophil Count Decreased, Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 1, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Neutrophil Count Decreased, Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 1, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Neutrophil Count Decreased, Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 2, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Neutrophil Count Decreased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 2, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Neutrophil Count Decreased, Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 2, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Neutrophil Count Decreased, Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 2, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Neutrophil Count Decreased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 3, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Neutrophil Count Decreased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 3, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Neutrophil Count Decreased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 3, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Neutrophil Count Decreased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 3, Grade 4: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Neutrophil Count Decreased, Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 4, Grade 0: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Neutrophil Count Decreased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 4, Grade 1: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Neutrophil Count Decreased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 4, Grade 2: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Neutrophil Count Decreased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 4, Grade 3: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Neutrophil Count Decreased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Missing, Grade 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Missing, Grade 0 |  |  |  |  | 1 |  |  |  |
  Neutrophil Count Decreased, Missing, Grade 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Missing, Grade 1 |  |  |  |  | 0 |  |  |  |
  Neutrophil Count Decreased, Missing, Grade 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Missing, Grade 2 |  |  |  |  | 0 |  |  |  |
  Neutrophil Count Decreased, Missing, Grade 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Missing, Grade 3 |  |  |  |  | 0 |  |  |  |
  Neutrophil Count Decreased, Missing, Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 24 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Missing, Grade 4 |  |  |  |  | 0 |  |  |  |
  Platelet Count Decreased, Grade 0, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Platelet Count Decreased, Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Platelet Count Decreased, Grade 1, Grade 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Platelet Count Decreased, Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 0, Grade 1 | 0 | 1 | 1 | 1 | 3 | 4 | 1 | 1 | 2
  White Blood Cell Decreased, Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  White Blood Cell Decreased, Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  White Blood Cell Decreased, Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 0, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Part 1A: Number of Participants With Worst Case Hematology Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Normal ranges were 0.01 to 0.3*10^9 cells/L (basophils), 0 to 500 cells /L (eosinophils), 41 to 50 percentage of red blood cells (RBC) in blood (hematocrit), 1,000 - 4,800 lymphocytes per microliter (ÂµL) of blood (lymphocytes), 80-100 femtoliters (fl) (erythrocytes, mean corpuscular volume), 2 to 8 percentage of WBC (monocytes), 40 to 60 cells/mcL (neutrophils) and Women: 4.2 to 5.4 million RBC/ microliter (mcL) of blood and Men: 4.7 to 6.1 million RBC/ mcL (erythrocytes count). Participants were counted in worst case category that their value changes to low, normal or no change [NC] or high), unless there is NC in their category. Participants whose laboratory value category was unchanged (e.g. High to High) or whose value became normal, were recorded in "To Normal or No Change" category. Participants were counted twice if participant had values that changed To Low and To High, so percentages may not add to 100%.
Time Frame: Up to approximately 367 weeks
Population: All Treated Population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: Feladilimab (Fela) 0.001 Milligram/Kilogram (mg/kg) | Part 1A: Fela 0.003 mg/kg | Part 1A: Fela 0.010 mg/kg | Part 1A: Fela 0.030 mg/kg | Part 1A: Fela 0.100 mg/kg | Part 1A: Fela 0.300 mg/kg | Part 1A: Fela 1.000 mg/kg | Part 1A: Fela 3.000 mg/kg | Part 1A: Fela 10.000 mg/kg
Number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 15 | 27 | 7
Participants
  Basophils, To Low: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 24 | 12 | 22 | 7
  Basophils, To Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils, To Normal or No Change: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 24 | 12 | 22 | 7
  Basophils, To Normal or No Change | 1 | 1 | 2 | 6 | 24 | 24 | 11 | 22 | 7
  Basophils, To High: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 24 | 12 | 22 | 7
  Basophils, To High | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
  Eosinophils, To Low: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 13 | 27 | 7
  Eosinophils, To Low | 0 | 1 | 0 | 0 | 3 | 2 | 2 | 2 | 1
  Eosinophils, To Normal or No Change: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 13 | 27 | 7
  Eosinophils, To Normal or No Change | 1 | 0 | 2 | 7 | 20 | 20 | 10 | 21 | 6
  Eosinophils, To High: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 13 | 27 | 7
  Eosinophils, To High | 0 | 0 | 0 | 0 | 3 | 4 | 1 | 5 | 0
  Hematocrit, To Low | 0 | 0 | 1 | 2 | 10 | 7 | 2 | 6 | 2
  Hematocrit, To Normal or No Change | 1 | 1 | 1 | 5 | 14 | 18 | 13 | 21 | 5
  Hematocrit, To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Lymphocytes, To Low: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0
  Lymphocytes, To Low |  |  |  |  | 2 | 1 | 1 |  |
  Lymphocytes, To Normal or No Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0
  Lymphocytes, To Normal or No Change |  |  |  |  | 0 | 0 | 0 |  |
  Lymphocytes, To High: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0
  Lymphocytes, To High |  |  |  |  | 0 | 0 | 0 |  |
  Erythrocytes, Mean Corpuscular Volume, To Low: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Erythrocytes, Mean Corpuscular Volume, To Low |  |  |  |  |  |  | 1 |  |
  Erythrocytes, Mean Corpuscular Volume, To Normal or No Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Erythrocytes, Mean Corpuscular Volume, To Normal or No Change |  |  |  |  |  |  | 0 |  |
  Erythrocytes, Mean Corpuscular Volume, To High: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Erythrocytes, Mean Corpuscular Volume, To High |  |  |  |  |  |  | 0 |  |
  Monocytes, To Low: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Monocytes, To Low | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Monocytes, To Normal or No Change: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Monocytes, To Normal or No Change | 0 | 1 | 1 | 5 | 18 | 21 | 11 | 21 | 6
  Monocytes, To High: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Monocytes, To High | 1 | 0 | 1 | 2 | 5 | 3 | 3 | 6 | 1
  Neutrophils, To Low: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
  Neutrophils, To Low |  |  |  |  | 0 | 0 | 0 |  |
  Neutrophils, To Normal or No Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
  Neutrophils, To Normal or No Change |  |  |  |  | 0 | 0 | 0 |  |
  Neutrophils, To High: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
  Neutrophils, To High |  |  |  |  | 1 | 1 | 1 |  |
  Erythrocytes, To Low: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Erythrocytes, To Low | 0 | 0 | 1 | 0 | 7 | 7 | 0 | 3 | 3
  Erythrocytes, To Normal or No Change: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Erythrocytes, To Normal or No Change | 1 | 1 | 1 | 7 | 17 | 18 | 14 | 24 | 3
  Erythrocytes, To High: number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
  Erythrocytes, To High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

7. Primary Outcome: Part 1A: Number of Participants With Worst Case Urinalysis Results Post-Baseline Relative to Baseline
Description: Urine samples were collected to assess urine glucose, ketones and occult blood using dipstick method. The dipstick test gave results in a semi-quantitative manner, and results for urinalysis parameters were recorded as negative, trace, 1+, 2+, 3+ indicating proportional concentrations in the urine sample. Baseline (Day 1) was defined as the most recent, non-missing value prior to or on the first study treatment dose date. Result for urinalysis parameters were recorded as no change/decreased and any increase.
Time Frame: Up to approximately 367 weeks
Population: All treated population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: Feladilimab (Fela) 0.001 Milligram/Kilogram (mg/kg) | Part 1A: Fela 0.003 mg/kg | Part 1A: Fela 0.010 mg/kg | Part 1A: Fela 0.030 mg/kg | Part 1A: Fela 0.100 mg/kg | Part 1A: Fela 0.300 mg/kg | Part 1A: Fela 1.000 mg/kg | Part 1A: Fela 3.000 mg/kg | Part 1A: Fela 10.000 mg/kg
Number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 14 | 27 | 7
Participants
  Glucose, No Change/Decreased | 1 | 1 | 2 | 7 | 23 | 22 | 12 | 25 | 7
  Glucose, any increase | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 2 | 0
  Ketones, No Change/Decreased: number analyzed (Participants) | 1 | 1 | 2 | 7 | 23 | 25 | 14 | 27 | 7
  Ketones, No Change/Decreased | 0 | 0 | 1 | 6 | 19 | 21 | 10 | 15 | 5
  Ketones, any increase: number analyzed (Participants) | 1 | 1 | 2 | 7 | 23 | 25 | 14 | 27 | 7
  Ketones, any increase | 1 | 1 | 1 | 1 | 4 | 4 | 4 | 12 | 2
  Occult Blood, No Change/Decreased: number analyzed (Participants) | 1 | 1 | 2 | 7 | 23 | 25 | 14 | 27 | 7
  Occult Blood, No Change/Decreased | 1 | 1 | 1 | 5 | 17 | 18 | 8 | 15 | 7
  Occult Blood, any increase: number analyzed (Participants) | 1 | 1 | 2 | 7 | 23 | 25 | 14 | 27 | 7
  Occult Blood, any increase | 0 | 0 | 1 | 2 | 6 | 7 | 6 | 12 | 0

8. Primary Outcome: Part 1A: Number of Participants With Dose Modifications of Feladilimab
Description: Number of participants with dose modifications (including dose delays, dose escalations and infusion interruptions) were reported for Feladilimab.
Time Frame: Up to approximately 367 weeks
Population: All treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: Feladilimab (Fela) 0.001 Milligram/Kilogram (mg/kg) | Part 1A: Fela 0.003 mg/kg | Part 1A: Fela 0.010 mg/kg | Part 1A: Fela 0.030 mg/kg | Part 1A: Fela 0.100 mg/kg | Part 1A: Fela 0.300 mg/kg | Part 1A: Fela 1.000 mg/kg | Part 1A: Fela 3.000 mg/kg | Part 1A: Fela 10.000 mg/kg
Number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 15 | 27 | 7
Participants
  Dose Delays | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 3 | 1
  Dose Escalations | 0 | 0 | 0 | 2 | 3 | 1 | 1 | 0 | 0
  infusion interruptions | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Part 2A: Number of Participants With Any Adverse Event(s) (AEs) and Serious Adverse Event(s) (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. SAE is defined as any untoward medical occurrence that, at any dose results in death, Is life-threatening, Requires inpatient hospitalization or prolongation of existing hospitalization, Results in persistent disability/incapacity or Is a congenital anomaly/birth defect, Other situations which involve medical or scientific judgment or is associated with liver injury and impaired liver function. SAEs are subset of AEs. A summary of number of participants with any AEs and SAEs is presented. AEs were coded using the MedDRA dictionary.
Time Frame: Up to approximately 367 weeks
Population: All Treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: Fela 0.010 mg/kg + Pembrolizumab (Pembro) 200 mg | Part 2A: Fela 0.030 mg/kg + Pembro 200 mg | Part 2A: Fela 0.100 mg/kg + Pembro 200 mg | Part 2A: Fela 0.300 mg/kg + Pembro 200 mg | Part 2A: Fela 1.000 mg/kg + Pembro 200 mg | Part 2A: Fela 3.000 mg/kg + Pembro 200 mg | Part 2A: Fela 8 mg + GSK3174998 8 mg | Part 2A: Fela 8 mg + GSK3174998 24 mg | Part 2A: Fela 24 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 80 mg | Part 2A: Fela 24 mg + Chemotherapy | Part 2A: Fela 80 mg + Chemotherapy | Part 2A: Fela 24 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 80 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 24 mg + Dostarlimab 500 mg + Cobolimab 300 mg | Part 2A: Fela 24 mg + Bintrafusp Alfa 2400 mg
Number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 16 | 4 | 3 | 6 | 36 | 13 | 22 | 1 | 4
Participants
  Any AEs | 5 | 5 | 5 | 5 | 8 | 10 | 0 | 4 | 15 | 4 | 3 | 6 | 36 | 13 | 22 | 1 | 4
  Any SAEs | 3 | 2 | 3 | 2 | 3 | 4 | 0 | 2 | 5 | 2 | 1 | 4 | 13 | 3 | 17 | 0 | 1

10. Primary Outcome: Part 2A: Number of Participants With Dose Limiting Toxicity (DLT)
Description: DLT is an AE that is considered by the investigator to be clinically relevant and attributed to the study therapy during the 28-day DLT period and meets at least one of the DLT criteria: Febrile neutropenia; Grade 4 neutropenia of >7 days in duration or requiring Granulocyte Colony-stimulating Factor (G-CSF), anemia, thrombocytopenia, non-hematologic toxicity; Grade 3 thrombocytopenia with bleeding, pneumonitis, toxicity that does not resolve to Grade 1 or baseline within 3 days; Grade 2 ocular toxicity; Toxicity that results in permanent discontinuation of feladilimab monotherapy or in combination during the first four weeks of treatment; any other event which in the judgment of the investigator and GSK Medical Monitor is considered to be a DLT.
Time Frame: Up to 28 days
Population: DLT Evaluable Population. As pre-specified in the protocol, only specified treatment arms were planned and hence there are 0 participants analyzed for rest of the arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: Fela 0.010 mg/kg + Pembrolizumab (Pembro) 200 mg | Part 2A: Fela 0.030 mg/kg + Pembro 200 mg | Part 2A: Fela 0.100 mg/kg + Pembro 200 mg | Part 2A: Fela 0.300 mg/kg + Pembro 200 mg | Part 2A: Fela 1.000 mg/kg + Pembro 200 mg | Part 2A: Fela 3.000 mg/kg + Pembro 200 mg | Part 2A: Fela 8 mg + GSK3174998 8 mg | Part 2A: Fela 8 mg + GSK3174998 24 mg | Part 2A: Fela 24 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 80 mg | Part 2A: Fela 24 mg + Chemotherapy | Part 2A: Fela 80 mg + Chemotherapy | Part 2A: Fela 24 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 80 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 24 mg + Dostarlimab 500 mg + Cobolimab 300 mg | Part 2A: Fela 24 mg + Bintrafusp Alfa 2400 mg
Number analyzed (Participants) | 5 | 4 | 5 | 8 | 11 | 11 | 1 | 3 | 14 | 4 | 3 | 6 | 34 | 13 | 22 | 0 | 0
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3 |  |

11. Primary Outcome: Part 2A: Number of Participants With Worst-case Grade Change From Baseline in Clinical Chemistry Parameters
Description: as for outcome 3
Time Frame: Baseline (Day 1) and up to approximately 367 weeks
Population: All Treated Population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: Fela 0.010 mg/kg + Pembrolizumab (Pembro) 200 mg | Part 2A: Fela 0.030 mg/kg + Pembro 200 mg | Part 2A: Fela 0.100 mg/kg + Pembro 200 mg | Part 2A: Fela 0.300 mg/kg + Pembro 200 mg | Part 2A: Fela 1.000 mg/kg + Pembro 200 mg | Part 2A: Fela 3.000 mg/kg + Pembro 200 mg | Part 2A: Fela 8 mg + GSK3174998 8 mg | Part 2A: Fela 8 mg + GSK3174998 24 mg | Part 2A: Fela 24 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 80 mg | Part 2A: Fela 24 mg + Chemotherapy | Part 2A: Fela 80 mg + Chemotherapy | Part 2A: Fela 24 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 80 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 24 mg + Dostarlimab 500 mg + Cobolimab 300 mg | Part 2A: Fela 24 mg + Bintrafusp Alfa 2400 mg
Number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 16 | 4 | 3 | 6 | 36 | 13 | 22 | 1 | 4
Participants
  Hypoglycemia , Grade 0, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypoglycemia , Grade 0, Grade 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 5 | 1 | 1 | 0 | 0
  Hypoglycemia , Grade 0, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypoglycemia , Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
  Hypoglycemia , Grade 0, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypoglycemia , Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 0, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypoglycemia , Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 1, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypoglycemia , Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 1, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypoglycemia , Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 1, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypoglycemia , Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 1, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypoglycemia , Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 2, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypoglycemia , Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 2, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypoglycemia , Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 2, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypoglycemia , Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 2, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypoglycemia , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 3, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypoglycemia , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 3, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypoglycemia , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 3, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypoglycemia , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 3, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypoglycemia , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 4, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypoglycemia , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 4, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypoglycemia , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 4, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypoglycemia , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 4, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypoglycemia , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 0, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperglycemia , Grade 0, Grade 1 | 0 | 3 | 2 | 5 | 3 | 4 | 0 | 0 | 4 | 0 | 0 | 1 | 12 | 5 | 9 | 0 | 3
  Hyperglycemia , Grade 0, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperglycemia , Grade 0, Grade 2 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 1 | 0 | 1 | 4 | 2 | 1 | 0 | 0
  Hyperglycemia , Grade 0, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperglycemia , Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Hyperglycemia , Grade 0, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperglycemia , Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 1, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperglycemia , Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 1, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperglycemia , Grade 1, Grade 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0
  Hyperglycemia , Grade 1, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperglycemia , Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Hyperglycemia , Grade 1, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperglycemia , Grade 1, Grade 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 2, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperglycemia , Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 2, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperglycemia , Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Hyperglycemia , Grade 2, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperglycemia , Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Hyperglycemia , Grade 2, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperglycemia , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Hyperglycemia , Grade 3, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperglycemia , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 3, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperglycemia , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 3, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperglycemia , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 3, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperglycemia , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 4, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperglycemia , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 4, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperglycemia , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 4, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperglycemia , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 4, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperglycemia , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 0, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypoalbuminemia , Grade 0, Grade 1 | 2 | 1 | 1 | 1 | 3 | 3 | 0 | 0 | 2 | 0 | 0 | 1 | 5 | 5 | 6 | 0 | 0
  Hypoalbuminemia , Grade 0, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypoalbuminemia , Grade 0, Grade 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 5 | 1 | 3 | 0 | 0
  Hypoalbuminemia , Grade 0, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypoalbuminemia , Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 0, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypoalbuminemia , Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 1, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypoalbuminemia , Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 1, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypoalbuminemia , Grade 1, Grade 2 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 0 | 0 | 0
  Hypoalbuminemia , Grade 1, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypoalbuminemia , Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 1, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypoalbuminemia , Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 2, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypoalbuminemia , Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 2, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypoalbuminemia , Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 2, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypoalbuminemia , Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 2, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypoalbuminemia , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 3, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypoalbuminemia , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 3, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypoalbuminemia , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 3, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypoalbuminemia , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 3, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypoalbuminemia , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 4, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypoalbuminemia , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 4, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypoalbuminemia , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 4, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypoalbuminemia , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 4, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypoalbuminemia , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Missing, Grade 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 35 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Missing, Grade 0 |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  |  |  |
  Hypoalbuminemia , Missing, Grade 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 35 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Missing, Grade 1 |  |  |  |  |  |  |  |  |  |  |  |  | 1 |  |  |  |
  Hypoalbuminemia , Missing, Grade 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 35 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Missing, Grade 2 |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  |  |  |
  Hypoalbuminemia , Missing, Grade 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 35 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Missing, Grade 3 |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  |  |  |
  Hypoalbuminemia , Missing, Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 35 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Missing, Grade 4 |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  |  |  |
  AP Increased, Grade 0, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AP Increased, Grade 0, Grade 1 | 1 | 0 | 2 | 3 | 3 | 2 | 1 | 0 | 6 | 0 | 1 | 1 | 7 | 3 | 6 | 0 | 1
  AP Increased, Grade 0, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AP Increased, Grade 0, Grade 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 0, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AP Increased, Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  AP Increased, Grade 0, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AP Increased, Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 1, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AP Increased, Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 1, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AP Increased, Grade 1, Grade 2 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  AP Increased, Grade 1, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AP Increased, Grade 1, Grade 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 1, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AP Increased, Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 2, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AP Increased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 2, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AP Increased, Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 2, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AP Increased, Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 2, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AP Increased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 3, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AP Increased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 3, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AP Increased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 3, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AP Increased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  AP Increased, Grade 3, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AP Increased, Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 4, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AP Increased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 4, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AP Increased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 4, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AP Increased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 4, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AP Increased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 0, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  ALT Increased, Grade 0, Grade 1 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 10 | 5 | 7 | 0 | 0
  ALT Increased, Grade 0, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  ALT Increased, Grade 0, Grade 2 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  ALT Increased, Grade 0, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  ALT Increased, Grade 0, Grade 3 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 0, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  ALT Increased, Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  ALT Increased, Grade 1, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  ALT Increased, Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  ALT Increased, Grade 1, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  ALT Increased, Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 1, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  ALT Increased, Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 1, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  ALT Increased, Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 2, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  ALT Increased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 2, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  ALT Increased, Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  ALT Increased, Grade 2, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  ALT Increased, Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 2, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  ALT Increased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 3, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  ALT Increased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 3, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  ALT Increased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 3, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  ALT Increased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 3, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  ALT Increased, Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 4, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  ALT Increased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 4, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  ALT Increased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 4, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  ALT Increased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 4, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  ALT Increased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 0, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AST Increased, Grade 0, Grade 1 | 0 | 1 | 3 | 5 | 2 | 6 | 0 | 0 | 1 | 1 | 0 | 0 | 9 | 2 | 5 | 0 | 2
  AST Increased, Grade 0, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AST Increased, Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  AST Increased, Grade 0, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AST Increased, Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 0, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AST Increased, Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  AST Increased, Grade 1, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AST Increased, Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  AST Increased, Grade 1, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AST Increased, Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
  AST Increased, Grade 1, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AST Increased, Grade 1, Grade 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 1, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AST Increased, Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 2, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AST Increased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 2, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AST Increased, Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 2, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AST Increased, Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 2, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AST Increased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 3, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AST Increased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 3, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AST Increased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 3, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AST Increased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 3, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AST Increased, Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 4, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AST Increased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 4, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AST Increased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 4, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AST Increased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 4, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  AST Increased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 0, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 12 | 21 | 1 | 4
  Blood Bilirubin Increased, Grade 0, Grade 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 2 | 0 | 0
  Blood Bilirubin Increased, Grade 0, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 12 | 21 | 1 | 4
  Blood Bilirubin Increased, Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 0, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 12 | 21 | 1 | 4
  Blood Bilirubin Increased, Grade 0, Grade 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Blood Bilirubin Increased, Grade 0, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 12 | 21 | 1 | 4
  Blood Bilirubin Increased, Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 1, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 12 | 21 | 1 | 4
  Blood Bilirubin Increased, Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 1, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 12 | 21 | 1 | 4
  Blood Bilirubin Increased, Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 1, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 12 | 21 | 1 | 4
  Blood Bilirubin Increased, Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 1, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 12 | 21 | 1 | 4
  Blood Bilirubin Increased, Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 2, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 12 | 21 | 1 | 4
  Blood Bilirubin Increased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 2, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 12 | 21 | 1 | 4
  Blood Bilirubin Increased, Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 2, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 12 | 21 | 1 | 4
  Blood Bilirubin Increased, Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 2, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 12 | 21 | 1 | 4
  Blood Bilirubin Increased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 3, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 12 | 21 | 1 | 4
  Blood Bilirubin Increased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 3, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 12 | 21 | 1 | 4
  Blood Bilirubin Increased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 3, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 12 | 21 | 1 | 4
  Blood Bilirubin Increased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 3, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 12 | 21 | 1 | 4
  Blood Bilirubin Increased, Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 4, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 12 | 21 | 1 | 4
  Blood Bilirubin Increased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 4, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 12 | 21 | 1 | 4
  Blood Bilirubin Increased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 4, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 12 | 21 | 1 | 4
  Blood Bilirubin Increased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 4, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 12 | 21 | 1 | 4
  Blood Bilirubin Increased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 0, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Creatinine Increased, Grade 0, Grade 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 2 | 2 | 0 | 0
  Creatinine Increased, Grade 0, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Creatinine Increased, Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0
  Creatinine Increased, Grade 0, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Creatinine Increased, Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 0, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Creatinine Increased, Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 1, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Creatinine Increased, Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 1, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Creatinine Increased, Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 1, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Creatinine Increased, Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 1, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Creatinine Increased, Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 2, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Creatinine Increased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 2, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Creatinine Increased, Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 2, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Creatinine Increased, Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 2, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Creatinine Increased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 3, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Creatinine Increased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 3, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Creatinine Increased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 3, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Creatinine Increased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 3, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Creatinine Increased, Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 4, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Creatinine Increased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 4, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Creatinine Increased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 4, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Creatinine Increased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 4, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Creatinine Increased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Missing, Grade 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 35 | 0 | 21 | 0 | 0
  Creatinine Increased, Missing, Grade 0 |  |  |  |  |  |  |  |  |  |  |  |  | 1 |  | 0 |  |
  Creatinine Increased, Missing, Grade 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 35 | 0 | 21 | 0 | 0
  Creatinine Increased, Missing, Grade 1 |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  | 0 |  |
  Creatinine Increased, Missing, Grade 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 35 | 0 | 21 | 0 | 0
  Creatinine Increased, Missing, Grade 2 |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  | 0 |  |
  Creatinine Increased, Missing, Grade 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 35 | 0 | 21 | 0 | 0
  Creatinine Increased, Missing, Grade 3 |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  | 0 |  |
  Creatinine Increased, Missing, Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 35 | 0 | 21 | 0 | 0
  Creatinine Increased, Missing, Grade 4 |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  | 1 |  |
  Hypokalemia , Grade 0, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypokalemia , Grade 0, Grade 1 | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 4 | 5 | 3 | 0 | 0
  Hypokalemia , Grade 0, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypokalemia , Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 0, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypokalemia , Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0
  Hypokalemia , Grade 0, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypokalemia , Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 1, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypokalemia , Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Hypokalemia , Grade 1, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypokalemia , Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 1, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypokalemia , Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Hypokalemia , Grade 1, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypokalemia , Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 2, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypokalemia , Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 2, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypokalemia , Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 2, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypokalemia , Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 2, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypokalemia , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 3, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypokalemia , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 3, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypokalemia , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 3, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypokalemia , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 3, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypokalemia , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 4, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypokalemia , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 4, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypokalemia , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 4, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypokalemia , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 4, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypokalemia , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 0, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperkalemia , Grade 0, Grade 1 | 0 | 1 | 1 | 2 | 2 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 6 | 4 | 3 | 0 | 0
  Hyperkalemia , Grade 0, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperkalemia , Grade 0, Grade 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 0, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperkalemia , Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 0, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperkalemia , Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 1, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperkalemia , Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Hyperkalemia , Grade 1, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperkalemia , Grade 1, Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 1, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperkalemia , Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 1, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperkalemia , Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 2, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperkalemia , Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 2, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperkalemia , Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 2, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperkalemia , Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 2, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperkalemia , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 3, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperkalemia , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 3, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperkalemia , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 3, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperkalemia , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 3, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperkalemia , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 4, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperkalemia , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 4, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperkalemia , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 4, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperkalemia , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 4, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyperkalemia , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 0, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyponatremia , Grade 0, Grade 1 | 1 | 0 | 2 | 2 | 5 | 6 | 0 | 2 | 1 | 2 | 0 | 2 | 8 | 9 | 12 | 0 | 1
  Hyponatremia , Grade 0, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyponatremia , Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 0, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyponatremia , Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 1 | 0 | 0
  Hyponatremia , Grade 0, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyponatremia , Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 1, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyponatremia , Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 1, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyponatremia , Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 1, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyponatremia , Grade 1, Grade 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Hyponatremia , Grade 1, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyponatremia , Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 2, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyponatremia , Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 2, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyponatremia , Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 2, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyponatremia , Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 2, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyponatremia , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 3, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyponatremia , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 3, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyponatremia , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 3, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyponatremia , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 3, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyponatremia , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 4, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyponatremia , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 4, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyponatremia , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 4, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyponatremia , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 4, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hyponatremia , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 0, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypernatremia , Grade 0, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 0 | 0 | 0
  Hypernatremia , Grade 0, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypernatremia , Grade 0, Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 0, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypernatremia , Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 0, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypernatremia , Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
  Hypernatremia , Grade 1, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypernatremia , Grade 1, Grade 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 1, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypernatremia , Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 1, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypernatremia , Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 1, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypernatremia , Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 2, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypernatremia , Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 2, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypernatremia , Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 2, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypernatremia , Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 2, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypernatremia , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 3, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypernatremia , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 3, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypernatremia , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 3, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypernatremia , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 3, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypernatremia , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 4, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypernatremia , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 4, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypernatremia , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 4, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypernatremia , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 4, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hypernatremia , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 0, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypocalcemia , Grade 0, Grade 1 | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 7 | 5 | 1 | 0 | 0
  Hypocalcemia , Grade 0, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypocalcemia , Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
  Hypocalcemia , Grade 0, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypocalcemia , Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 0, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypocalcemia , Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Hypocalcemia , Grade 1, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypocalcemia , Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 1, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypocalcemia , Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 1, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypocalcemia , Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 1, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypocalcemia , Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 2, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypocalcemia , Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 2, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypocalcemia , Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 2, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypocalcemia , Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 2, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypocalcemia , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 3, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypocalcemia , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 3, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypocalcemia , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 3, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypocalcemia , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 3, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypocalcemia , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 4, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypocalcemia , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 4, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypocalcemia , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 4, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypocalcemia , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 4, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypocalcemia , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Missing, Grade 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 35 | 0 | 0 | 0 | 0
  Hypocalcemia , Missing, Grade 0 |  |  |  |  |  |  |  |  |  |  |  |  | 1 |  |  |  |
  Hypocalcemia , Missing, Grade 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 35 | 0 | 0 | 0 | 0
  Hypocalcemia , Missing, Grade 1 |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  |  |  |
  Hypocalcemia , Missing, Grade 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 35 | 0 | 0 | 0 | 0
  Hypocalcemia , Missing, Grade 2 |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  |  |  |
  Hypocalcemia , Missing, Grade 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 35 | 0 | 0 | 0 | 0
  Hypocalcemia , Missing, Grade 3 |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  |  |  |
  Hypocalcemia , Missing, Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 35 | 0 | 0 | 0 | 0
  Hypocalcemia , Missing, Grade 4 |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  |  |  |
  Hypercalcemia , Grade 0, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypercalcemia , Grade 0, Grade 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 4 | 2 | 1 | 0 | 0
  Hypercalcemia , Grade 0, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypercalcemia , Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 0, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypercalcemia , Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Hypercalcemia , Grade 0, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypercalcemia , Grade 0, Grade 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 1, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypercalcemia , Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
  Hypercalcemia , Grade 1, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypercalcemia , Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 1, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypercalcemia , Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 1, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypercalcemia , Grade 1, Grade 4 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 2, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypercalcemia , Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 2, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypercalcemia , Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 2, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypercalcemia , Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 4 | 0 | 1
  Hypercalcemia , Grade 2, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypercalcemia , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 3, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypercalcemia , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 3, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypercalcemia , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 3, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypercalcemia , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 3, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypercalcemia , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 4, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypercalcemia , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 4, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypercalcemia , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 4, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypercalcemia , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 4, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 18 | 1 | 4
  Hypercalcemia , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Missing, Grade 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 35 | 0 | 0 | 0 | 0
  Hypercalcemia , Missing, Grade 0 |  |  |  |  |  |  |  |  |  |  |  |  | 1 |  |  |  |
  Hypercalcemia , Missing, Grade 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 35 | 0 | 0 | 0 | 0
  Hypercalcemia , Missing, Grade 1 |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  |  |  |
  Hypercalcemia , Missing, Grade 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 35 | 0 | 0 | 0 | 0
  Hypercalcemia , Missing, Grade 2 |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  |  |  |
  Hypercalcemia , Missing, Grade 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 35 | 0 | 0 | 0 | 0
  Hypercalcemia , Missing, Grade 3 |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  |  |  |
  Hypercalcemia , Missing, Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 35 | 0 | 0 | 0 | 0
  Hypercalcemia , Missing, Grade 4 |  |  |  |  |  |  |  |  |  |  |  |  | 0 |  |  |  |
  Chronic Kidney Disease , Grade 0, Grade 1: number analyzed (Participants) | 0 | 1 | 1 | 2 | 2 | 5 | 0 | 0 | 3 | 0 | 0 | 3 | 15 | 5 | 3 | 0 | 0
  Chronic Kidney Disease , Grade 0, Grade 1 |  | 0 | 0 | 0 | 1 | 1 |  |  | 0 |  |  | 0 | 0 | 0 | 0 |  |
  Chronic Kidney Disease , Grade 0, Grade 2: number analyzed (Participants) | 0 | 1 | 1 | 2 | 2 | 5 | 0 | 0 | 3 | 0 | 0 | 3 | 15 | 5 | 3 | 0 | 0
  Chronic Kidney Disease , Grade 0, Grade 2 |  | 0 | 0 | 0 | 0 | 0 |  |  | 0 |  |  | 0 | 0 | 1 | 0 |  |
  Chronic Kidney Disease , Grade 0, Grade 3: number analyzed (Participants) | 0 | 1 | 1 | 2 | 2 | 5 | 0 | 0 | 3 | 0 | 0 | 3 | 15 | 5 | 3 | 0 | 0
  Chronic Kidney Disease , Grade 0, Grade 3 |  | 0 | 0 | 0 | 0 | 0 |  |  | 0 |  |  | 0 | 0 | 0 | 0 |  |
  Chronic Kidney Disease , Grade 0, Grade 4: number analyzed (Participants) | 0 | 1 | 1 | 2 | 2 | 5 | 0 | 0 | 3 | 0 | 0 | 3 | 15 | 5 | 3 | 0 | 0
  Chronic Kidney Disease , Grade 0, Grade 4 |  | 0 | 0 | 0 | 0 | 0 |  |  | 0 |  |  | 0 | 0 | 0 | 0 |  |
  Chronic Kidney Disease , Grade 1, Grade 0: number analyzed (Participants) | 0 | 1 | 1 | 2 | 2 | 5 | 0 | 0 | 3 | 0 | 0 | 3 | 15 | 5 | 3 | 0 | 0
  Chronic Kidney Disease , Grade 1, Grade 0 |  | 0 | 0 | 0 | 0 | 0 |  |  | 0 |  |  | 0 | 0 | 0 | 0 |  |
  Chronic Kidney Disease , Grade 1, Grade 2: number analyzed (Participants) | 0 | 1 | 1 | 2 | 2 | 5 | 0 | 0 | 3 | 0 | 0 | 3 | 15 | 5 | 3 | 0 | 0
  Chronic Kidney Disease , Grade 1, Grade 2 |  | 0 | 0 | 1 | 0 | 0 |  |  | 1 |  |  | 0 | 0 | 0 | 0 |  |
  Chronic Kidney Disease , Grade 1, Grade 3: number analyzed (Participants) | 0 | 1 | 1 | 2 | 2 | 5 | 0 | 0 | 3 | 0 | 0 | 3 | 15 | 5 | 3 | 0 | 0
  Chronic Kidney Disease , Grade 1, Grade 3 |  | 0 | 0 | 0 | 0 | 0 |  |  | 0 |  |  | 0 | 0 | 0 | 0 |  |
  Chronic Kidney Disease , Grade 1, Grade 4: number analyzed (Participants) | 0 | 1 | 1 | 2 | 2 | 5 | 0 | 0 | 3 | 0 | 0 | 3 | 15 | 5 | 3 | 0 | 0
  Chronic Kidney Disease , Grade 1, Grade 4 |  | 0 | 0 | 0 | 0 | 0 |  |  | 0 |  |  | 0 | 0 | 0 | 0 |  |
  Chronic Kidney Disease , Grade 2, Grade 0: number analyzed (Participants) | 0 | 1 | 1 | 2 | 2 | 5 | 0 | 0 | 3 | 0 | 0 | 3 | 15 | 5 | 3 | 0 | 0
  Chronic Kidney Disease , Grade 2, Grade 0 |  | 0 | 0 | 0 | 0 | 0 |  |  | 0 |  |  | 0 | 0 | 0 | 0 |  |
  Chronic Kidney Disease , Grade 2, Grade 1: number analyzed (Participants) | 0 | 1 | 1 | 2 | 2 | 5 | 0 | 0 | 3 | 0 | 0 | 3 | 15 | 5 | 3 | 0 | 0
  Chronic Kidney Disease , Grade 2, Grade 1 |  | 0 | 0 | 0 | 0 | 0 |  |  | 0 |  |  | 0 | 0 | 0 | 0 |  |
  Chronic Kidney Disease , Grade 2, Grade 3: number analyzed (Participants) | 0 | 1 | 1 | 2 | 2 | 5 | 0 | 0 | 3 | 0 | 0 | 3 | 15 | 5 | 3 | 0 | 0
  Chronic Kidney Disease , Grade 2, Grade 3 |  | 0 | 0 | 0 | 0 | 0 |  |  | 0 |  |  | 0 | 0 | 0 | 0 |  |
  Chronic Kidney Disease , Grade 2, Grade 4: number analyzed (Participants) | 0 | 1 | 1 | 2 | 2 | 5 | 0 | 0 | 3 | 0 | 0 | 3 | 15 | 5 | 3 | 0 | 0
  Chronic Kidney Disease , Grade 2, Grade 4 |  | 0 | 0 | 0 | 0 | 0 |  |  | 0 |  |  | 0 | 0 | 0 | 0 |  |
  Chronic Kidney Disease , Grade 3, Grade 0: number analyzed (Participants) | 0 | 1 | 1 | 2 | 2 | 5 | 0 | 0 | 3 | 0 | 0 | 3 | 15 | 5 | 3 | 0 | 0
  Chronic Kidney Disease , Grade 3, Grade 0 |  | 0 | 0 | 0 | 0 | 0 |  |  | 0 |  |  | 0 | 0 | 0 | 0 |  |
  Chronic Kidney Disease , Grade 3, Grade 1: number analyzed (Participants) | 0 | 1 | 1 | 2 | 2 | 5 | 0 | 0 | 3 | 0 | 0 | 3 | 15 | 5 | 3 | 0 | 0
  Chronic Kidney Disease , Grade 3, Grade 1 |  | 0 | 0 | 0 | 0 | 0 |  |  | 0 |  |  | 0 | 0 | 0 | 0 |  |
  Chronic Kidney Disease , Grade 3, Grade 2: number analyzed (Participants) | 0 | 1 | 1 | 2 | 2 | 5 | 0 | 0 | 3 | 0 | 0 | 3 | 15 | 5 | 3 | 0 | 0
  Chronic Kidney Disease , Grade 3, Grade 2 |  | 0 | 0 | 0 | 0 | 0 |  |  | 0 |  |  | 0 | 0 | 0 | 0 |  |
  Chronic Kidney Disease , Grade 3, Grade 4: number analyzed (Participants) | 0 | 1 | 1 | 2 | 2 | 5 | 0 | 0 | 3 | 0 | 0 | 3 | 15 | 5 | 3 | 0 | 0
  Chronic Kidney Disease , Grade 3, Grade 4 |  | 0 | 0 | 0 | 0 | 0 |  |  | 0 |  |  | 0 | 0 | 0 | 0 |  |
  Chronic Kidney Disease , Grade 4, Grade 0: number analyzed (Participants) | 0 | 1 | 1 | 2 | 2 | 5 | 0 | 0 | 3 | 0 | 0 | 3 | 15 | 5 | 3 | 0 | 0
  Chronic Kidney Disease , Grade 4, Grade 0 |  | 0 | 0 | 0 | 0 | 0 |  |  | 0 |  |  | 0 | 0 | 0 | 0 |  |
  Chronic Kidney Disease , Grade 4, Grade 1: number analyzed (Participants) | 0 | 1 | 1 | 2 | 2 | 5 | 0 | 0 | 3 | 0 | 0 | 3 | 15 | 5 | 3 | 0 | 0
  Chronic Kidney Disease , Grade 4, Grade 1 |  | 0 | 0 | 0 | 0 | 0 |  |  | 0 |  |  | 0 | 0 | 0 | 0 |  |
  Chronic Kidney Disease , Grade 4, Grade 2: number analyzed (Participants) | 0 | 1 | 1 | 2 | 2 | 5 | 0 | 0 | 3 | 0 | 0 | 3 | 15 | 5 | 3 | 0 | 0
  Chronic Kidney Disease , Grade 4, Grade 2 |  | 0 | 0 | 0 | 0 | 0 |  |  | 0 |  |  | 0 | 0 | 0 | 0 |  |
  Chronic Kidney Disease , Grade 4, Grade 3: number analyzed (Participants) | 0 | 1 | 1 | 2 | 2 | 5 | 0 | 0 | 3 | 0 | 0 | 3 | 15 | 5 | 3 | 0 | 0
  Chronic Kidney Disease , Grade 4, Grade 3 |  | 0 | 0 | 0 | 0 | 0 |  |  | 0 |  |  | 0 | 0 | 0 | 0 |  |
  Chronic Kidney Disease , Missing, Grade 0: number analyzed (Participants) | 0 | 0 | 0 | 2 | 2 | 5 | 0 | 0 | 3 | 0 | 0 | 3 | 15 | 5 | 3 | 0 | 0
  Chronic Kidney Disease , Missing, Grade 0 |  |  |  | 0 | 0 | 0 |  |  | 0 |  |  | 1 | 1 | 0 | 0 |  |
  Chronic Kidney Disease , Missing, Grade 1: number analyzed (Participants) | 0 | 0 | 0 | 2 | 2 | 5 | 0 | 0 | 3 | 0 | 0 | 3 | 15 | 5 | 3 | 0 | 0
  Chronic Kidney Disease , Missing, Grade 1 |  |  |  | 1 | 0 | 1 |  |  | 1 |  |  | 0 | 3 | 1 | 2 |  |
  Chronic Kidney Disease , Missing, Grade 2: number analyzed (Participants) | 0 | 0 | 0 | 2 | 2 | 5 | 0 | 0 | 3 | 0 | 0 | 3 | 15 | 5 | 3 | 0 | 0
  Chronic Kidney Disease , Missing, Grade 2 |  |  |  | 0 | 1 | 0 |  |  | 0 |  |  | 1 | 5 | 0 | 0 |  |
  Chronic Kidney Disease , Missing, Grade 3: number analyzed (Participants) | 0 | 0 | 0 | 2 | 2 | 5 | 0 | 0 | 3 | 0 | 0 | 3 | 15 | 5 | 3 | 0 | 0
  Chronic Kidney Disease , Missing, Grade 3 |  |  |  | 0 | 0 | 0 |  |  | 0 |  |  | 1 | 0 | 0 | 0 |  |
  Chronic Kidney Disease , Missing, Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 2 | 2 | 5 | 0 | 0 | 3 | 0 | 0 | 3 | 15 | 5 | 3 | 0 | 0
  Chronic Kidney Disease , Missing, Grade 4 |  |  |  | 0 | 0 | 1 |  |  | 0 |  |  | 0 | 0 | 1 | 0 |  |

12. Primary Outcome: Part 2A: Number of Participants With Worst Case Chemistry Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Normal ranges were 6 to 8.3 grams/L (protein); 100 to 250 international units (IU)/L (Lactate Dehydrogenase(LDH)); 2.3 - 4.1 picomoles/L (Free Triiodothyronine(T3)); 4.6 to 11.2 picomoles/L (Free Thyroxine(T4)); 0 and 0.04 microgram (ug)/L (Troponin I); 0 - 0.01 ug/L (Troponin T); 0.45 to 4.5 milliunits (Mu)/L (Thyrotropin(TSH)); and 6 to 24 millimoles/L (Urea). Participants were counted in worst case category that their value changes to low, normal or no change [NC] or high), unless there is NC in their category. Participants whose laboratory value category was unchanged (e.g. High to High) or whose value became normal, were recorded in "To Normal or No Change" category. Participants were counted twice if participant had values that changed To Low and To High, so percentages may not add to 100%.
Time Frame: Up to approximately 367 weeks
Population: All Treated Population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: Fela 0.010 mg/kg + Pembrolizumab (Pembro) 200 mg | Part 2A: Fela 0.030 mg/kg + Pembro 200 mg | Part 2A: Fela 0.100 mg/kg + Pembro 200 mg | Part 2A: Fela 0.300 mg/kg + Pembro 200 mg | Part 2A: Fela 1.000 mg/kg + Pembro 200 mg | Part 2A: Fela 3.000 mg/kg + Pembro 200 mg | Part 2A: Fela 8 mg + GSK3174998 8 mg | Part 2A: Fela 8 mg + GSK3174998 24 mg | Part 2A: Fela 24 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 80 mg | Part 2A: Fela 24 mg + Chemotherapy | Part 2A: Fela 80 mg + Chemotherapy | Part 2A: Fela 24 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 80 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 24 mg + Dostarlimab 500 mg + Cobolimab 300 mg | Part 2A: Fela 24 mg + Bintrafusp Alfa 2400 mg
Number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 16 | 4 | 3 | 6 | 36 | 13 | 22 | 1 | 4
Participants
  Lactate Dehydrogenase (IU/L), To Low: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 1 | 1 | 5 | 0 | 3
  Lactate Dehydrogenase (IU/L), To Low |  |  |  |  |  |  |  |  | 0 | 0 | 0 |  | 0 | 0 | 0 |  | 0
  Lactate Dehydrogenase (IU/L), To Normal or No Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 1 | 1 | 5 | 0 | 3
  Lactate Dehydrogenase (IU/L), To Normal or No Change |  |  |  |  |  |  |  |  | 2 | 2 | 1 |  | 1 | 1 | 3 |  | 1
  Lactate Dehydrogenase (IU/L), To High: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 1 | 1 | 5 | 0 | 3
  Lactate Dehydrogenase (IU/L), To High |  |  |  |  |  |  |  |  | 0 | 0 | 0 |  | 0 | 0 | 2 |  | 2
  Protein (g/L), To Low: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Protein (g/L), To Low | 2 | 2 | 2 | 3 | 1 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 16 | 6 | 12 | 0 | 2
  Protein (g/L), To Normal or No Change: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Protein (g/L), To Normal or No Change | 3 | 3 | 3 | 3 | 8 | 10 | 0 | 4 | 12 | 2 | 3 | 3 | 18 | 6 | 9 | 1 | 1
  Protein (g/L), To High: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Protein (g/L), To High | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 0 | 0 | 2
  Triiodothyronine, Free (pmol/L), To Low: number analyzed (Participants) | 3 | 5 | 4 | 8 | 9 | 10 | 1 | 2 | 13 | 2 | 3 | 4 | 31 | 13 | 20 | 1 | 4
  Triiodothyronine, Free (pmol/L), To Low | 0 | 0 | 0 | 1 | 4 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 5 | 4 | 2 | 0 | 0
  Triiodothyronine, Free (pmol/L), To Normal or No Change: number analyzed (Participants) | 3 | 5 | 4 | 8 | 9 | 10 | 1 | 2 | 13 | 2 | 3 | 4 | 31 | 13 | 20 | 1 | 4
  Triiodothyronine, Free (pmol/L), To Normal or No Change | 2 | 5 | 3 | 6 | 4 | 6 | 1 | 2 | 10 | 2 | 3 | 3 | 26 | 7 | 18 | 1 | 3
  Triiodothyronine, Free (pmol/L), To High: number analyzed (Participants) | 3 | 5 | 4 | 8 | 9 | 10 | 1 | 2 | 13 | 2 | 3 | 4 | 31 | 13 | 20 | 1 | 4
  Triiodothyronine, Free (pmol/L), To High | 1 | 0 | 1 | 2 | 2 | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 1
  Thyroxine, Free (pmol/L), To Low: number analyzed (Participants) | 4 | 5 | 4 | 8 | 9 | 10 | 1 | 2 | 14 | 2 | 3 | 4 | 31 | 13 | 20 | 1 | 4
  Thyroxine, Free (pmol/L), To Low | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
  Thyroxine, Free (pmol/L), To Normal or No Change: number analyzed (Participants) | 4 | 5 | 4 | 8 | 9 | 10 | 1 | 2 | 14 | 2 | 3 | 4 | 31 | 13 | 20 | 1 | 4
  Thyroxine, Free (pmol/L), To Normal or No Change | 3 | 5 | 3 | 6 | 8 | 6 | 1 | 2 | 13 | 2 | 2 | 3 | 31 | 12 | 14 | 1 | 4
  Thyroxine, Free (pmol/L), To High: number analyzed (Participants) | 4 | 5 | 4 | 8 | 9 | 10 | 1 | 2 | 14 | 2 | 3 | 4 | 31 | 13 | 20 | 1 | 4
  Thyroxine, Free (pmol/L), To High | 1 | 0 | 1 | 1 | 0 | 4 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0
  Troponin I (ug/L), To Low: number analyzed (Participants) | 2 | 1 | 2 | 4 | 5 | 4 | 0 | 1 | 3 | 2 | 2 | 4 | 12 | 9 | 17 | 1 | 3
  Troponin I (ug/L), To Low | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
  Troponin I (ug/L), To Normal or No Change: number analyzed (Participants) | 2 | 1 | 2 | 4 | 5 | 4 | 0 | 1 | 3 | 2 | 2 | 4 | 12 | 9 | 17 | 1 | 3
  Troponin I (ug/L), To Normal or No Change | 1 | 1 | 2 | 3 | 4 | 3 |  | 1 | 3 | 2 | 1 | 4 | 11 | 9 | 9 | 1 | 2
  Troponin I (ug/L), To High: number analyzed (Participants) | 2 | 1 | 2 | 4 | 5 | 4 | 0 | 1 | 3 | 2 | 2 | 4 | 12 | 9 | 17 | 1 | 3
  Troponin I (ug/L), To High | 1 | 0 | 0 | 1 | 1 | 1 |  | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 6 | 0 | 1
  Troponin T (ug/L), To Low: number analyzed (Participants) | 2 | 1 | 1 | 3 | 2 | 3 | 0 | 0 | 10 | 0 | 1 | 0 | 13 | 3 | 2 | 0 | 3
  Troponin T (ug/L), To Low | 0 | 0 | 0 | 0 | 0 | 0 |  |  | 0 |  | 0 |  | 0 | 0 | 0 |  | 0
  Troponin T (ug/L), To Normal or No Change: number analyzed (Participants) | 2 | 1 | 1 | 3 | 2 | 3 | 0 | 0 | 10 | 0 | 1 | 0 | 13 | 3 | 2 | 0 | 3
  Troponin T (ug/L), To Normal or No Change | 2 | 1 | 1 | 2 | 2 | 3 |  |  | 8 |  | 1 |  | 12 | 2 | 2 |  | 3
  Troponin T (ug/L), To High: number analyzed (Participants) | 2 | 1 | 1 | 3 | 2 | 3 | 0 | 0 | 10 | 0 | 1 | 0 | 13 | 3 | 2 | 0 | 3
  Troponin T (ug/L), To High | 0 | 0 | 0 | 1 | 0 | 0 |  |  | 2 |  | 0 |  | 1 | 1 | 0 |  | 0
  Thyrotropin (mU/L), To Low: number analyzed (Participants) | 4 | 5 | 5 | 8 | 9 | 10 | 1 | 2 | 14 | 2 | 3 | 4 | 31 | 13 | 20 | 1 | 4
  Thyrotropin (mU/L), To Low | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
  Thyrotropin (mU/L), To Normal or No Change: number analyzed (Participants) | 4 | 5 | 5 | 8 | 9 | 10 | 1 | 2 | 14 | 2 | 3 | 4 | 31 | 13 | 20 | 1 | 4
  Thyrotropin (mU/L), To Normal or No Change | 2 | 5 | 2 | 5 | 6 | 9 | 1 | 1 | 8 | 1 | 2 | 2 | 23 | 11 | 17 | 1 | 3
  Thyrotropin (mU/L), To High: number analyzed (Participants) | 4 | 5 | 5 | 8 | 9 | 10 | 1 | 2 | 14 | 2 | 3 | 4 | 31 | 13 | 20 | 1 | 4
  Thyrotropin (mU/L), To High | 1 | 0 | 1 | 3 | 3 | 0 | 0 | 1 | 4 | 1 | 1 | 2 | 6 | 1 | 3 | 0 | 1
  Urea (mmol/L), To Low: number analyzed (Participants) | 5 | 4 | 5 | 7 | 10 | 11 | 1 | 4 | 12 | 4 | 3 | 5 | 24 | 11 | 17 | 1 | 4
  Urea (mmol/L), To Low | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 2 | 0 | 0 | 0
  Urea (mmol/L), To Normal or No Change: number analyzed (Participants) | 5 | 4 | 5 | 7 | 10 | 11 | 1 | 4 | 12 | 4 | 3 | 5 | 24 | 11 | 17 | 1 | 4
  Urea (mmol/L), To Normal or No Change | 3 | 3 | 2 | 4 | 4 | 6 | 1 | 2 | 9 | 2 | 1 | 1 | 17 | 3 | 12 | 1 | 2
  Urea (mmol/L), To High: number analyzed (Participants) | 5 | 4 | 5 | 7 | 10 | 11 | 1 | 4 | 12 | 4 | 3 | 5 | 24 | 11 | 17 | 1 | 4
  Urea (mmol/L), To High | 1 | 1 | 3 | 3 | 4 | 3 | 0 | 1 | 3 | 2 | 1 | 3 | 6 | 8 | 5 | 0 | 2

13. Primary Outcome: Part 2A: Number of Participants With Worst-case Grade Change From Baseline in Hematology Parameters
Description: as for outcome 5
Time Frame: Baseline (Day 1) and up to approximately 367 weeks
Population: All Treated Population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: Fela 0.010 mg/kg + Pembrolizumab (Pembro) 200 mg | Part 2A: Fela 0.030 mg/kg + Pembro 200 mg | Part 2A: Fela 0.100 mg/kg + Pembro 200 mg | Part 2A: Fela 0.300 mg/kg + Pembro 200 mg | Part 2A: Fela 1.000 mg/kg + Pembro 200 mg | Part 2A: Fela 3.000 mg/kg + Pembro 200 mg | Part 2A: Fela 8 mg + GSK3174998 8 mg | Part 2A: Fela 8 mg + GSK3174998 24 mg | Part 2A: Fela 24 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 80 mg | Part 2A: Fela 24 mg + Chemotherapy | Part 2A: Fela 80 mg + Chemotherapy | Part 2A: Fela 24 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 80 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 24 mg + Dostarlimab 500 mg + Cobolimab 300 mg | Part 2A: Fela 24 mg + Bintrafusp Alfa 2400 mg
Number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 16 | 4 | 3 | 6 | 36 | 13 | 22 | 1 | 4
Participants
  Anemia , Grade 0, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Anemia , Grade 0, Grade 1 | 0 | 1 | 0 | 2 | 4 | 2 | 0 | 1 | 3 | 0 | 2 | 2 | 5 | 2 | 2 | 0 | 1
  Anemia , Grade 0, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Anemia , Grade 0, Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 4 | 4 | 4 | 0 | 0
  Anemia , Grade 0, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Anemia , Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
  Anemia , Grade 0, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Anemia , Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 1, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Anemia , Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 1, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Anemia , Grade 1, Grade 2 | 0 | 3 | 2 | 1 | 2 | 2 | 0 | 0 | 2 | 1 | 1 | 1 | 9 | 2 | 7 | 0 | 1
  Anemia , Grade 1, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Anemia , Grade 1, Grade 3 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 0 | 3 | 0 | 0
  Anemia , Grade 1, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Anemia , Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 2, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Anemia , Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 2, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Anemia , Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 2, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Anemia , Grade 2, Grade 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 4 | 1 | 0 | 0 | 0
  Anemia , Grade 2, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Anemia , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 3, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Anemia , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 3, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Anemia , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 3, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Anemia , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 3, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Anemia , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 4, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Anemia , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 4, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Anemia , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 4, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Anemia , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 4, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Anemia , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 0, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hemoglobin Increased, Grade 0, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 0, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hemoglobin Increased, Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 0, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hemoglobin Increased, Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 0, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hemoglobin Increased, Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 1, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hemoglobin Increased, Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 1, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hemoglobin Increased, Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 1, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hemoglobin Increased, Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 1, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hemoglobin Increased, Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 2, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hemoglobin Increased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 2, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hemoglobin Increased, Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 2, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hemoglobin Increased, Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 2, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hemoglobin Increased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 3, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hemoglobin Increased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 3, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hemoglobin Increased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 3, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hemoglobin Increased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 3, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hemoglobin Increased, Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 4, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hemoglobin Increased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 4, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hemoglobin Increased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 4, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hemoglobin Increased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 4, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hemoglobin Increased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 0, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Decreased, Grade 0, Grade 1 | 0 | 2 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 8 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 0, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Decreased, Grade 0, Grade 2 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 7 | 3 | 3 | 0 | 0
  Lymphocyte Count Decreased, Grade 0, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Decreased, Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 3 | 0 | 0
  Lymphocyte Count Decreased, Grade 0, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Decreased, Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 1, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Decreased, Grade 1, Grade 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 1, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Decreased, Grade 1, Grade 2 | 1 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 4 | 0 | 1 | 1 | 3 | 2 | 3 | 0 | 0
  Lymphocyte Count Decreased, Grade 1, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Decreased, Grade 1, Grade 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 2 | 4 | 0 | 0
  Lymphocyte Count Decreased, Grade 1, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Decreased, Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 2, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Decreased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 2, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Decreased, Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 2, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Decreased, Grade 2, Grade 3 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 4 | 0 | 0
  Lymphocyte Count Decreased, Grade 2, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Decreased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 3, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Decreased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 3, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Decreased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 3, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Decreased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Lymphocyte Count Decreased, Grade 3, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Decreased, Grade 3, Grade 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 4, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Decreased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 4, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Decreased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 4, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Decreased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 4, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Decreased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 0, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Increased, Grade 0, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 0, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Increased, Grade 0, Grade 2 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 0, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Increased, Grade 0, Grade 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Lymphocyte Count Increased, Grade 0, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Increased, Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 1, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Increased, Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 1, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Increased, Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 1, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Increased, Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 1, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Increased, Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 2, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Increased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 2, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Increased, Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 2, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Increased, Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 2, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Increased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 3, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Increased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 3, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Increased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 3, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Increased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 3, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Increased, Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 4, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Increased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 4, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Increased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 4, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Increased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 4, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Lymphocyte Count Increased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 0, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Neutrophil Count Decreased, Grade 0, Grade 1 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 0, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Neutrophil Count Decreased, Grade 0, Grade 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 8 | 2 | 3 | 0 | 0
  Neutrophil Count Decreased, Grade 0, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Neutrophil Count Decreased, Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 8 | 5 | 10 | 0 | 0
  Neutrophil Count Decreased, Grade 0, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Neutrophil Count Decreased, Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 2 | 4 | 0 | 0
  Neutrophil Count Decreased, Grade 1, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Neutrophil Count Decreased, Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 1, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Neutrophil Count Decreased, Grade 1, Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 1, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Neutrophil Count Decreased, Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 1, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Neutrophil Count Decreased, Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 2, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Neutrophil Count Decreased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 2, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Neutrophil Count Decreased, Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 2, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Neutrophil Count Decreased, Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 2, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Neutrophil Count Decreased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 3, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Neutrophil Count Decreased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 3, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Neutrophil Count Decreased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 3, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Neutrophil Count Decreased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 3, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Neutrophil Count Decreased, Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 4, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Neutrophil Count Decreased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 4, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Neutrophil Count Decreased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 4, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Neutrophil Count Decreased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 4, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Neutrophil Count Decreased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 0, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Platelet Count Decreased, Grade 0, Grade 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 13 | 6 | 4 | 1 | 0
  Platelet Count Decreased, Grade 0, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Platelet Count Decreased, Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 0 | 0
  Platelet Count Decreased, Grade 0, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Platelet Count Decreased, Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 1 | 0 | 0
  Platelet Count Decreased, Grade 0, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Platelet Count Decreased, Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 2 | 0 | 0
  Platelet Count Decreased, Grade 1, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Platelet Count Decreased, Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 1, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Platelet Count Decreased, Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 1, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Platelet Count Decreased, Grade 1, Grade 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 1, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Platelet Count Decreased, Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Platelet Count Decreased, Grade 2, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Platelet Count Decreased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 2, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Platelet Count Decreased, Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 2, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Platelet Count Decreased, Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 2, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Platelet Count Decreased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 3, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Platelet Count Decreased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 3, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Platelet Count Decreased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 3, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Platelet Count Decreased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 3, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Platelet Count Decreased, Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 4, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Platelet Count Decreased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 4, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Platelet Count Decreased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Platelet Count Decreased, Grade 4, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Platelet Count Decreased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 4, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Platelet Count Decreased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 0, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  White Blood Cell Decreased, Grade 0, Grade 1 | 1 | 0 | 2 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 5 | 0 | 0
  White Blood Cell Decreased, Grade 0, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  White Blood Cell Decreased, Grade 0, Grade 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 11 | 6 | 5 | 0 | 0
  White Blood Cell Decreased, Grade 0, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  White Blood Cell Decreased, Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 13 | 3 | 7 | 0 | 0
  White Blood Cell Decreased, Grade 0, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  White Blood Cell Decreased, Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
  White Blood Cell Decreased, Grade 1, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  White Blood Cell Decreased, Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White Blood Cell Decreased, Grade 1, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  White Blood Cell Decreased, Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 1, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  White Blood Cell Decreased, Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0
  White Blood Cell Decreased, Grade 1, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  White Blood Cell Decreased, Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 2, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  White Blood Cell Decreased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 2, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  White Blood Cell Decreased, Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 2, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  White Blood Cell Decreased, Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 2, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  White Blood Cell Decreased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 3, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  White Blood Cell Decreased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 3, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  White Blood Cell Decreased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 3, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  White Blood Cell Decreased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 3, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  White Blood Cell Decreased, Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 4, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  White Blood Cell Decreased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 4, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  White Blood Cell Decreased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 4, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  White Blood Cell Decreased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 4, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  White Blood Cell Decreased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 0, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Leukocytosis , Grade 0, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 0, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Leukocytosis , Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 0, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Leukocytosis , Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 0, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Leukocytosis , Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 1, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Leukocytosis , Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 1, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Leukocytosis , Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 1, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Leukocytosis , Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 1, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Leukocytosis , Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 2, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Leukocytosis , Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 2, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Leukocytosis , Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 2, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Leukocytosis , Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 2, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Leukocytosis , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 3, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Leukocytosis , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 3, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Leukocytosis , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 3, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Leukocytosis , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 3, Grade 4: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Leukocytosis , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 4, Grade 0: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Leukocytosis , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 4, Grade 1: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Leukocytosis , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 4, Grade 2: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Leukocytosis , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 4, Grade 3: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Leukocytosis , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Primary Outcome: Part 2A: Number of Participants With Worst Case Hematology Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Normal ranges were 0.01 to 0.3*10^9 cells/L (basophils), 0 to 500 cells /L (eosinophils), 41 to 50 percentage of RBC in blood (hematocrit), 2 to 8 percentage of WBC (monocytes), 40 to 60 cells/mcL (neutrophils) and Women: 4.2 to 5.4 million RBC/mcL of blood and Men: 4.7 to 6.1 million RBC/ mcL (erythrocytes count). Participants were counted in worst case category that their value changes to low, normal or no change [NC] or high), unless there is NC in their category. Participants whose laboratory value category was unchanged (e.g. High to High) or whose value became normal, were recorded in "To Normal or No Change" category. Participants were counted twice if participant had values that changed To Low and To High, so percentages may not add to 100%.
Time Frame: Up to approximately 367 weeks
Population: All Treated Population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: Fela 0.010 mg/kg + Pembrolizumab (Pembro) 200 mg | Part 2A: Fela 0.030 mg/kg + Pembro 200 mg | Part 2A: Fela 0.100 mg/kg + Pembro 200 mg | Part 2A: Fela 0.300 mg/kg + Pembro 200 mg | Part 2A: Fela 1.000 mg/kg + Pembro 200 mg | Part 2A: Fela 3.000 mg/kg + Pembro 200 mg | Part 2A: Fela 8 mg + GSK3174998 8 mg | Part 2A: Fela 8 mg + GSK3174998 24 mg | Part 2A: Fela 24 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 80 mg | Part 2A: Fela 24 mg + Chemotherapy | Part 2A: Fela 80 mg + Chemotherapy | Part 2A: Fela 24 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 80 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 24 mg + Dostarlimab 500 mg + Cobolimab 300 mg | Part 2A: Fela 24 mg + Bintrafusp Alfa 2400 mg
Number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 16 | 4 | 3 | 6 | 36 | 13 | 22 | 1 | 4
Participants
  Basophils, To Low: number analyzed (Participants) | 5 | 4 | 5 | 8 | 11 | 11 | 1 | 4 | 12 | 4 | 3 | 5 | 27 | 13 | 21 | 1 | 4
  Basophils, To Low | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 0 | 0
  Basophils, To Normal or No Change: number analyzed (Participants) | 5 | 4 | 5 | 8 | 11 | 11 | 1 | 4 | 12 | 4 | 3 | 5 | 27 | 13 | 21 | 1 | 4
  Basophils, To Normal or No Change | 5 | 3 | 5 | 6 | 11 | 11 | 1 | 4 | 11 | 4 | 3 | 5 | 23 | 9 | 17 | 1 | 2
  Basophils, To High: number analyzed (Participants) | 5 | 4 | 5 | 8 | 11 | 11 | 1 | 4 | 12 | 4 | 3 | 5 | 27 | 13 | 21 | 1 | 4
  Basophils, To High | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 3 | 1 | 0 | 2
  Eosinophils, To Low: number analyzed (Participants) | 5 | 4 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 32 | 13 | 21 | 1 | 4
  Eosinophils, To Low | 1 | 2 | 1 | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 6 | 2 | 6 | 0 | 0
  Eosinophils, To Normal or No Change: number analyzed (Participants) | 5 | 4 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 32 | 13 | 21 | 1 | 4
  Eosinophils, To Normal or No Change | 4 | 2 | 3 | 5 | 8 | 8 | 1 | 3 | 9 | 4 | 3 | 3 | 23 | 7 | 12 | 1 | 2
  Eosinophils, To High: number analyzed (Participants) | 5 | 4 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 32 | 13 | 21 | 1 | 4
  Eosinophils, To High | 0 | 0 | 1 | 3 | 1 | 3 | 0 | 1 | 4 | 0 | 0 | 1 | 3 | 6 | 6 | 0 | 2
  Hematocrit, To Low: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hematocrit, To Low | 1 | 1 | 0 | 3 | 4 | 2 | 0 | 0 | 3 | 0 | 2 | 3 | 15 | 7 | 9 | 0 | 0
  Hematocrit, To Normal or No Change: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hematocrit, To Normal or No Change | 4 | 4 | 5 | 5 | 6 | 9 | 1 | 4 | 11 | 4 | 1 | 1 | 21 | 6 | 12 | 1 | 4
  Hematocrit, To High: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Hematocrit, To High | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
  Monocytes, To Low: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Monocytes, To Low | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 7 | 10 | 0 | 0
  Monocytes, To Normal or No Change: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Monocytes, To Normal or No Change | 3 | 3 | 4 | 4 | 9 | 9 | 1 | 3 | 12 | 3 | 3 | 2 | 16 | 4 | 6 | 1 | 4
  Monocytes, To High: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 35 | 13 | 21 | 1 | 4
  Monocytes, To High | 2 | 2 | 1 | 4 | 2 | 2 | 0 | 1 | 3 | 1 | 0 | 3 | 12 | 6 | 13 | 0 | 0
  Neutrophils, To Low: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils, To Low |  |  | 0 |  |  |  |  |  |  |  |  |  |  |  |  |  |
  Neutrophils, To Normal or No Change: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils, To Normal or No Change |  |  | 0 |  |  |  |  |  |  |  |  |  |  |  |  |  |
  Neutrophils, To High: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils, To High |  |  | 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |
  Erythrocytes, To Low: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Erythrocytes, To Low | 1 | 1 | 0 | 3 | 6 | 3 | 0 | 0 | 2 | 2 | 2 | 3 | 17 | 9 | 13 | 0 | 2
  Erythrocytes, To Normal or No Change: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Erythrocytes, To Normal or No Change | 4 | 4 | 5 | 5 | 4 | 8 | 1 | 4 | 13 | 2 | 1 | 2 | 19 | 4 | 8 | 1 | 2
  Erythrocytes, To High: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 5 | 36 | 13 | 21 | 1 | 4
  Erythrocytes, To High | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1

15. Primary Outcome: Part 2A: Number of Participants With Worst Case Urinalysis Results Post-Baseline Relative to Baseline
Description: as for outcome 7
Time Frame: Up to approximately 367 weeks
Population: All treated population. Only those participants with data available at specified categories have been analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: Fela 0.010 mg/kg + Pembrolizumab (Pembro) 200 mg | Part 2A: Fela 0.030 mg/kg + Pembro 200 mg | Part 2A: Fela 0.100 mg/kg + Pembro 200 mg | Part 2A: Fela 0.300 mg/kg + Pembro 200 mg | Part 2A: Fela 1.000 mg/kg + Pembro 200 mg | Part 2A: Fela 3.000 mg/kg + Pembro 200 mg | Part 2A: Fela 8 mg + GSK3174998 8 mg | Part 2A: Fela 8 mg + GSK3174998 24 mg | Part 2A: Fela 24 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 80 mg | Part 2A: Fela 24 mg + Chemotherapy | Part 2A: Fela 80 mg + Chemotherapy | Part 2A: Fela 24 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 80 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 24 mg + Dostarlimab 500 mg + Cobolimab 300 mg | Part 2A: Fela 24 mg + Bintrafusp Alfa 2400 mg
Number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 6 | 34 | 13 | 22 | 1 | 4
Participants
  Glucose, No Change/Decreased | 5 | 4 | 4 | 8 | 10 | 10 | 1 | 3 | 14 | 4 | 3 | 5 | 33 | 8 | 16 | 1 | 4
  Glucose, Any increase | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 5 | 6 | 0 | 0
  Ketones, No Change/Decreased | 1 | 5 | 3 | 6 | 9 | 9 | 1 | 4 | 14 | 3 | 2 | 2 | 28 | 7 | 15 | 0 | 3
  Ketones, Any increase | 4 | 0 | 2 | 2 | 2 | 2 | 0 | 0 | 1 | 1 | 1 | 4 | 6 | 6 | 7 | 1 | 1
  Occult Blood, No Change/Decreased: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 6 | 32 | 13 | 22 | 1 | 4
  Occult Blood, No Change/Decreased | 3 | 4 | 1 | 4 | 7 | 5 | 1 | 4 | 13 | 3 | 2 | 3 | 23 | 7 | 12 | 1 | 4
  Occult Blood, Any increase: number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 15 | 4 | 3 | 6 | 32 | 13 | 22 | 1 | 4
  Occult Blood, Any increase | 2 | 1 | 4 | 4 | 4 | 6 | 0 | 0 | 2 | 1 | 1 | 3 | 9 | 6 | 10 | 0 | 0

16. Primary Outcome: Part 2A: Number of Participants With Dose Modifications of Feladilimab
Description: Number of participants with dose modifications (including dose delays, dose escalations, and infusion interruptions) were reported for Feladilimab
Time Frame: Up to approximately 367 weeks
Population: All Treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: Fela 0.010 mg/kg + Pembrolizumab (Pembro) 200 mg | Part 2A: Fela 0.030 mg/kg + Pembro 200 mg | Part 2A: Fela 0.100 mg/kg + Pembro 200 mg | Part 2A: Fela 0.300 mg/kg + Pembro 200 mg | Part 2A: Fela 1.000 mg/kg + Pembro 200 mg | Part 2A: Fela 3.000 mg/kg + Pembro 200 mg | Part 2A: Fela 8 mg + GSK3174998 8 mg | Part 2A: Fela 8 mg + GSK3174998 24 mg | Part 2A: Fela 24 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 80 mg | Part 2A: Fela 24 mg + Chemotherapy | Part 2A: Fela 80 mg + Chemotherapy | Part 2A: Fela 24 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 80 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 24 mg + Dostarlimab 500 mg + Cobolimab 300 mg | Part 2A: Fela 24 mg + Bintrafusp Alfa 2400 mg
Number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 16 | 4 | 3 | 6 | 36 | 13 | 22 | 1 | 4
Participants
  Dose delays | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 4 | 7 | 11 | 0 | 0
  Dose escalations | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Infusion interruptions | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Part 1B: Number of Participants With Any Adverse Event(s) (AEs) and Serious Adverse Event(s) (SAEs)
Description: as for outcome 9
Time Frame: Up to approximately 367 weeks
Population: All Treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1B: Fela 0.300 mg/kg | Part 1B: Fela 1.000 mg/kg | Part 1B: Fela 24 mg
Number analyzed (Participants) | 39 | 115 | 59
Participants
  Any AEs | 34 | 111 | 55
  Any SAEs | 9 | 44 | 19

18. Secondary Outcome: Part 1B: Number of Participants With Worst-case Grade Change From Baseline in Clinical Chemistry Parameters
Description: as for outcome 3
Time Frame: Baseline (Day 1) and up to approximately 367 weeks
Population: All Treated Population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1B: Fela 0.300 mg/kg | Part 1B: Fela 1.000 mg/kg | Part 1B: Fela 24 mg
Number analyzed (Participants) | 39 | 115 | 59
Participants
  Hypoglycemia , Grade 0, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Hypoglycemia , Grade 0, Grade 1 | 4 | 7 | 6
  Hypoglycemia , Grade 0, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Hypoglycemia , Grade 0, Grade 2 | 0 | 2 | 1
  Hypoglycemia , Grade 0, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Hypoglycemia , Grade 0, Grade 3 | 0 | 0 | 0
  Hypoglycemia , Grade 0, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Hypoglycemia , Grade 0, Grade 4 | 0 | 0 | 0
  Hypoglycemia , Grade 1, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Hypoglycemia , Grade 1, Grade 0 | 1 | 2 | 0
  Hypoglycemia , Grade 1, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Hypoglycemia , Grade 1, Grade 2 | 0 | 0 | 0
  Hypoglycemia , Grade 1, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Hypoglycemia , Grade 1, Grade 3 | 0 | 0 | 0
  Hypoglycemia , Grade 1, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Hypoglycemia , Grade 1, Grade 4 | 0 | 0 | 0
  Hypoglycemia , Grade 2, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Hypoglycemia , Grade 2, Grade 0 | 0 | 0 | 0
  Hypoglycemia , Grade 2, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Hypoglycemia , Grade 2, Grade 1 | 0 | 0 | 0
  Hypoglycemia , Grade 2, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Hypoglycemia , Grade 2, Grade 3 | 0 | 0 | 0
  Hypoglycemia , Grade 2, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Hypoglycemia , Grade 2, Grade 4 | 0 | 0 | 0
  Hypoglycemia , Grade 3, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Hypoglycemia , Grade 3, Grade 0 | 0 | 0 | 0
  Hypoglycemia , Grade 3, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Hypoglycemia , Grade 3, Grade 1 | 0 | 0 | 0
  Hypoglycemia , Grade 3, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Hypoglycemia , Grade 3, Grade 2 | 0 | 0 | 0
  Hypoglycemia , Grade 3, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Hypoglycemia , Grade 3, Grade 4 | 0 | 0 | 0
  Hypoglycemia , Grade 4, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Hypoglycemia , Grade 4, Grade 0 | 0 | 0 | 0
  Hypoglycemia , Grade 4, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Hypoglycemia , Grade 4, Grade 1 | 0 | 0 | 0
  Hypoglycemia , Grade 4, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Hypoglycemia , Grade 4, Grade 2 | 0 | 0 | 0
  Hypoglycemia , Grade 4, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Hypoglycemia , Grade 4, Grade 3 | 0 | 0 | 0
  Hypoglycemia , Missing, Grade 0: number analyzed (Participants) | 0 | 113 | 58
  Hypoglycemia , Missing, Grade 0 |  | 2 | 2
  Hypoglycemia , Missing, Grade 1: number analyzed (Participants) | 0 | 113 | 58
  Hypoglycemia , Missing, Grade 1 |  | 0 | 1
  Hypoglycemia , Missing, Grade 2: number analyzed (Participants) | 0 | 113 | 58
  Hypoglycemia , Missing, Grade 2 |  | 0 | 0
  Hypoglycemia , Missing, Grade 3: number analyzed (Participants) | 0 | 113 | 58
  Hypoglycemia , Missing, Grade 3 |  | 0 | 0
  Hypoglycemia , Missing, Grade 4: number analyzed (Participants) | 0 | 113 | 58
  Hypoglycemia , Missing, Grade 4 |  | 0 | 0
  Hyperglycemia , Grade 0, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Hyperglycemia , Grade 0, Grade 1 | 11 | 38 | 19
  Hyperglycemia , Grade 0, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Hyperglycemia , Grade 0, Grade 2 | 1 | 8 | 3
  Hyperglycemia , Grade 0, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Hyperglycemia , Grade 0, Grade 3 | 0 | 0 | 0
  Hyperglycemia , Grade 0, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Hyperglycemia , Grade 0, Grade 4 | 0 | 0 | 0
  Hyperglycemia , Grade 1, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Hyperglycemia , Grade 1, Grade 0 | 2 | 0 | 1
  Hyperglycemia , Grade 1, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Hyperglycemia , Grade 1, Grade 2 | 0 | 1 | 4
  Hyperglycemia , Grade 1, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Hyperglycemia , Grade 1, Grade 3 | 0 | 2 | 0
  Hyperglycemia , Grade 1, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Hyperglycemia , Grade 1, Grade 4 | 0 | 1 | 0
  Hyperglycemia , Grade 2, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Hyperglycemia , Grade 2, Grade 0 | 0 | 0 | 0
  Hyperglycemia , Grade 2, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Hyperglycemia , Grade 2, Grade 1 | 0 | 1 | 0
  Hyperglycemia , Grade 2, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Hyperglycemia , Grade 2, Grade 3 | 0 | 0 | 0
  Hyperglycemia , Grade 2, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Hyperglycemia , Grade 2, Grade 4 | 0 | 0 | 0
  Hyperglycemia , Grade 3, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Hyperglycemia , Grade 3, Grade 0 | 0 | 0 | 0
  Hyperglycemia , Grade 3, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Hyperglycemia , Grade 3, Grade 1 | 0 | 0 | 0
  Hyperglycemia , Grade 3, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Hyperglycemia , Grade 3, Grade 2 | 0 | 0 | 1
  Hyperglycemia , Grade 3, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Hyperglycemia , Grade 3, Grade 4 | 0 | 0 | 0
  Hyperglycemia , Grade 4, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Hyperglycemia , Grade 4, Grade 0 | 0 | 0 | 0
  Hyperglycemia , Grade 4, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Hyperglycemia , Grade 4, Grade 1 | 0 | 0 | 0
  Hyperglycemia , Grade 4, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Hyperglycemia , Grade 4, Grade 2 | 0 | 0 | 0
  Hyperglycemia , Grade 4, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Hyperglycemia , Grade 4, Grade 3 | 0 | 0 | 0
  Hyperglycemia , Missing, Grade 0: number analyzed (Participants) | 0 | 113 | 58
  Hyperglycemia , Missing, Grade 0 |  | 1 | 3
  Hyperglycemia , Missing, Grade 1: number analyzed (Participants) | 0 | 113 | 58
  Hyperglycemia , Missing, Grade 1 |  | 1 | 0
  Hyperglycemia , Missing, Grade 2: number analyzed (Participants) | 0 | 113 | 58
  Hyperglycemia , Missing, Grade 2 |  | 0 | 0
  Hyperglycemia , Missing, Grade 3: number analyzed (Participants) | 0 | 113 | 58
  Hyperglycemia , Missing, Grade 3 |  | 0 | 0
  Hyperglycemia , Missing, Grade 4: number analyzed (Participants) | 0 | 113 | 58
  Hyperglycemia , Missing, Grade 4 |  | 0 | 0
  Hypoalbuminemia , Grade 0, Grade 1: number analyzed (Participants) | 37 | 112 | 58
  Hypoalbuminemia , Grade 0, Grade 1 | 4 | 12 | 10
  Hypoalbuminemia , Grade 0, Grade 2: number analyzed (Participants) | 37 | 112 | 58
  Hypoalbuminemia , Grade 0, Grade 2 | 1 | 12 | 2
  Hypoalbuminemia , Grade 0, Grade 3: number analyzed (Participants) | 37 | 112 | 58
  Hypoalbuminemia , Grade 0, Grade 3 | 0 | 0 | 1
  Hypoalbuminemia , Grade 0, Grade 4: number analyzed (Participants) | 37 | 112 | 58
  Hypoalbuminemia , Grade 0, Grade 4 | 0 | 0 | 0
  Hypoalbuminemia , Grade 1, Grade 0: number analyzed (Participants) | 37 | 112 | 58
  Hypoalbuminemia , Grade 1, Grade 0 | 1 | 1 | 1
  Hypoalbuminemia , Grade 1, Grade 2: number analyzed (Participants) | 37 | 112 | 58
  Hypoalbuminemia , Grade 1, Grade 2 | 2 | 5 | 2
  Hypoalbuminemia , Grade 1, Grade 3: number analyzed (Participants) | 37 | 112 | 58
  Hypoalbuminemia , Grade 1, Grade 3 | 0 | 1 | 0
  Hypoalbuminemia , Grade 1, Grade 4: number analyzed (Participants) | 37 | 112 | 58
  Hypoalbuminemia , Grade 1, Grade 4 | 0 | 0 | 0
  Hypoalbuminemia , Grade 2, Grade 0: number analyzed (Participants) | 37 | 112 | 58
  Hypoalbuminemia , Grade 2, Grade 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 2, Grade 1: number analyzed (Participants) | 37 | 112 | 58
  Hypoalbuminemia , Grade 2, Grade 1 | 0 | 0 | 1
  Hypoalbuminemia , Grade 2, Grade 3: number analyzed (Participants) | 37 | 112 | 58
  Hypoalbuminemia , Grade 2, Grade 3 | 0 | 2 | 1
  Hypoalbuminemia , Grade 2, Grade 4: number analyzed (Participants) | 37 | 112 | 58
  Hypoalbuminemia , Grade 2, Grade 4 | 0 | 0 | 0
  Hypoalbuminemia , Grade 3, Grade 0: number analyzed (Participants) | 37 | 112 | 58
  Hypoalbuminemia , Grade 3, Grade 0 | 0 | 0 | 1
  Hypoalbuminemia , Grade 3, Grade 1: number analyzed (Participants) | 37 | 112 | 58
  Hypoalbuminemia , Grade 3, Grade 1 | 0 | 0 | 0
  Hypoalbuminemia , Grade 3, Grade 2: number analyzed (Participants) | 37 | 112 | 58
  Hypoalbuminemia , Grade 3, Grade 2 | 0 | 0 | 0
  Hypoalbuminemia , Grade 3, Grade 4: number analyzed (Participants) | 37 | 112 | 58
  Hypoalbuminemia , Grade 3, Grade 4 | 0 | 0 | 0
  Hypoalbuminemia , Grade 4, Grade 0: number analyzed (Participants) | 37 | 112 | 58
  Hypoalbuminemia , Grade 4, Grade 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 4, Grade 1: number analyzed (Participants) | 37 | 112 | 58
  Hypoalbuminemia , Grade 4, Grade 1 | 0 | 0 | 0
  Hypoalbuminemia , Grade 4, Grade 2: number analyzed (Participants) | 37 | 112 | 58
  Hypoalbuminemia , Grade 4, Grade 2 | 0 | 0 | 0
  Hypoalbuminemia , Grade 4, Grade 3: number analyzed (Participants) | 37 | 112 | 58
  Hypoalbuminemia , Grade 4, Grade 3 | 0 | 0 | 0
  Hypoalbuminemia , Missing, Grade 0: number analyzed (Participants) | 0 | 112 | 0
  Hypoalbuminemia , Missing, Grade 0 |  | 1 |
  Hypoalbuminemia , Missing, Grade 1: number analyzed (Participants) | 0 | 112 | 0
  Hypoalbuminemia , Missing, Grade 1 |  | 0 |
  Hypoalbuminemia , Missing, Grade 2: number analyzed (Participants) | 0 | 112 | 0
  Hypoalbuminemia , Missing, Grade 2 |  | 0 |
  Hypoalbuminemia , Missing, Grade 3: number analyzed (Participants) | 0 | 112 | 0
  Hypoalbuminemia , Missing, Grade 3 |  | 0 |
  Hypoalbuminemia , Missing, Grade 4: number analyzed (Participants) | 0 | 112 | 0
  Hypoalbuminemia , Missing, Grade 4 |  | 0 |
  AP Increased, Grade 0, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  AP Increased, Grade 0, Grade 1 | 7 | 20 | 8
  AP Increased, Grade 0, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  AP Increased, Grade 0, Grade 2 | 2 | 3 | 0
  AP Increased, Grade 0, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  AP Increased, Grade 0, Grade 3 | 0 | 0 | 0
  AP Increased, Grade 0, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  AP Increased, Grade 0, Grade 4 | 0 | 0 | 0
  AP Increased, Grade 1, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  AP Increased, Grade 1, Grade 0 | 0 | 1 | 2
  AP Increased, Grade 1, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  AP Increased, Grade 1, Grade 2 | 3 | 9 | 1
  AP Increased, Grade 1, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  AP Increased, Grade 1, Grade 3 | 0 | 1 | 1
  AP Increased, Grade 1, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  AP Increased, Grade 1, Grade 4 | 0 | 0 | 0
  AP Increased, Grade 2, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  AP Increased, Grade 2, Grade 0 | 0 | 0 | 0
  AP Increased, Grade 2, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  AP Increased, Grade 2, Grade 1 | 0 | 0 | 0
  AP Increased, Grade 2, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  AP Increased, Grade 2, Grade 3 | 1 | 0 | 0
  AP Increased, Grade 2, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  AP Increased, Grade 2, Grade 4 | 0 | 0 | 0
  AP Increased, Grade 3, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  AP Increased, Grade 3, Grade 0 | 0 | 0 | 0
  AP Increased, Grade 3, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  AP Increased, Grade 3, Grade 1 | 0 | 0 | 0
  AP Increased, Grade 3, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  AP Increased, Grade 3, Grade 2 | 0 | 0 | 0
  AP Increased, Grade 3, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  AP Increased, Grade 3, Grade 4 | 0 | 0 | 0
  AP Increased, Grade 4, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  AP Increased, Grade 4, Grade 0 | 0 | 0 | 0
  AP Increased, Grade 4, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  AP Increased, Grade 4, Grade 1 | 0 | 0 | 0
  AP Increased, Grade 4, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  AP Increased, Grade 4, Grade 2 | 0 | 0 | 0
  AP Increased, Grade 4, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  AP Increased, Grade 4, Grade 3 | 0 | 0 | 0
  AP Increased, Missing, Grade 0: number analyzed (Participants) | 37 | 0 | 0
  AP Increased, Missing, Grade 0 | 1 |  |
  AP Increased, Missing, Grade 1: number analyzed (Participants) | 37 | 0 | 0
  AP Increased, Missing, Grade 1 | 0 |  |
  AP Increased, Missing, Grade 2: number analyzed (Participants) | 37 | 0 | 0
  AP Increased, Missing, Grade 2 | 0 |  |
  AP Increased, Missing, Grade 3: number analyzed (Participants) | 37 | 0 | 0
  AP Increased, Missing, Grade 3 | 0 |  |
  AP Increased, Missing, Grade 4: number analyzed (Participants) | 37 | 0 | 0
  AP Increased, Missing, Grade 4 | 0 |  |
  ALT Increased, Grade 0, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  ALT Increased, Grade 0, Grade 1 | 4 | 18 | 8
  ALT Increased, Grade 0, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  ALT Increased, Grade 0, Grade 2 | 0 | 2 | 1
  ALT Increased, Grade 0, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  ALT Increased, Grade 0, Grade 3 | 0 | 1 | 1
  ALT Increased, Grade 0, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  ALT Increased, Grade 0, Grade 4 | 0 | 0 | 0
  ALT Increased, Grade 1, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  ALT Increased, Grade 1, Grade 0 | 0 | 2 | 0
  ALT Increased, Grade 1, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  ALT Increased, Grade 1, Grade 2 | 2 | 0 | 1
  ALT Increased, Grade 1, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  ALT Increased, Grade 1, Grade 3 | 0 | 2 | 0
  ALT Increased, Grade 1, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  ALT Increased, Grade 1, Grade 4 | 0 | 0 | 0
  ALT Increased, Grade 2, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  ALT Increased, Grade 2, Grade 0 | 0 | 0 | 0
  ALT Increased, Grade 2, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  ALT Increased, Grade 2, Grade 1 | 0 | 0 | 0
  ALT Increased, Grade 2, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  ALT Increased, Grade 2, Grade 3 | 0 | 0 | 0
  ALT Increased, Grade 2, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  ALT Increased, Grade 2, Grade 4 | 0 | 0 | 0
  ALT Increased, Grade 3, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  ALT Increased, Grade 3, Grade 0 | 0 | 0 | 0
  ALT Increased, Grade 3, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  ALT Increased, Grade 3, Grade 1 | 0 | 0 | 0
  ALT Increased, Grade 3, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  ALT Increased, Grade 3, Grade 2 | 0 | 0 | 0
  ALT Increased, Grade 3, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  ALT Increased, Grade 3, Grade 4 | 0 | 0 | 0
  ALT Increased, Grade 4, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  ALT Increased, Grade 4, Grade 0 | 0 | 0 | 0
  ALT Increased, Grade 4, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  ALT Increased, Grade 4, Grade 1 | 0 | 0 | 0
  ALT Increased, Grade 4, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  ALT Increased, Grade 4, Grade 2 | 0 | 0 | 0
  ALT Increased, Grade 4, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  ALT Increased, Grade 4, Grade 3 | 0 | 0 | 0
  ALT Increased, Missing, Grade 0: number analyzed (Participants) | 0 | 0 | 58
  ALT Increased, Missing, Grade 0 |  |  | 1
  ALT Increased, Missing, Grade 1: number analyzed (Participants) | 0 | 0 | 58
  ALT Increased, Missing, Grade 1 |  |  | 0
  ALT Increased, Missing, Grade 2: number analyzed (Participants) | 0 | 0 | 58
  ALT Increased, Missing, Grade 2 |  |  | 0
  ALT Increased, Missing, Grade 3: number analyzed (Participants) | 0 | 0 | 58
  ALT Increased, Missing, Grade 3 |  |  | 0
  ALT Increased, Missing, Grade 4: number analyzed (Participants) | 0 | 0 | 58
  ALT Increased, Missing, Grade 4 |  |  | 0
  AST Increased, Grade 0, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  AST Increased, Grade 0, Grade 1 | 9 | 25 | 15
  AST Increased, Grade 0, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  AST Increased, Grade 0, Grade 2 | 0 | 0 | 1
  AST Increased, Grade 0, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  AST Increased, Grade 0, Grade 3 | 0 | 3 | 2
  AST Increased, Grade 0, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  AST Increased, Grade 0, Grade 4 | 0 | 0 | 0
  AST Increased, Grade 1, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  AST Increased, Grade 1, Grade 0 | 0 | 1 | 0
  AST Increased, Grade 1, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  AST Increased, Grade 1, Grade 2 | 1 | 1 | 0
  AST Increased, Grade 1, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  AST Increased, Grade 1, Grade 3 | 0 | 1 | 0
  AST Increased, Grade 1, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  AST Increased, Grade 1, Grade 4 | 0 | 0 | 0
  AST Increased, Grade 2, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  AST Increased, Grade 2, Grade 0 | 0 | 0 | 0
  AST Increased, Grade 2, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  AST Increased, Grade 2, Grade 1 | 0 | 1 | 0
  AST Increased, Grade 2, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  AST Increased, Grade 2, Grade 3 | 0 | 0 | 0
  AST Increased, Grade 2, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  AST Increased, Grade 2, Grade 4 | 0 | 0 | 0
  AST Increased, Grade 3, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  AST Increased, Grade 3, Grade 0 | 0 | 0 | 0
  AST Increased, Grade 3, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  AST Increased, Grade 3, Grade 1 | 0 | 0 | 0
  AST Increased, Grade 3, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  AST Increased, Grade 3, Grade 2 | 0 | 0 | 0
  AST Increased, Grade 3, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  AST Increased, Grade 3, Grade 4 | 0 | 0 | 0
  AST Increased, Grade 4, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  AST Increased, Grade 4, Grade 0 | 0 | 0 | 0
  AST Increased, Grade 4, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  AST Increased, Grade 4, Grade 1 | 0 | 0 | 0
  AST Increased, Grade 4, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  AST Increased, Grade 4, Grade 2 | 0 | 0 | 0
  AST Increased, Grade 4, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  AST Increased, Grade 4, Grade 3 | 0 | 0 | 0
  AST Increased, Missing, Grade 0: number analyzed (Participants) | 0 | 113 | 0
  AST Increased, Missing, Grade 0 |  | 1 |
  AST Increased, Missing, Grade 1: number analyzed (Participants) | 0 | 113 | 0
  AST Increased, Missing, Grade 1 |  | 0 |
  AST Increased, Missing, Grade 2: number analyzed (Participants) | 0 | 113 | 0
  AST Increased, Missing, Grade 2 |  | 0 |
  AST Increased, Missing, Grade 3: number analyzed (Participants) | 0 | 113 | 0
  AST Increased, Missing, Grade 3 |  | 0 |
  AST Increased, Missing, Grade 4: number analyzed (Participants) | 0 | 113 | 0
  AST Increased, Missing, Grade 4 |  | 0 |
  Blood Bilirubin Increased, Grade 0, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Blood Bilirubin Increased, Grade 0, Grade 1 | 2 | 2 | 1
  Blood Bilirubin Increased, Grade 0, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Blood Bilirubin Increased, Grade 0, Grade 2 | 0 | 1 | 0
  Blood Bilirubin Increased, Grade 0, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Blood Bilirubin Increased, Grade 0, Grade 3 | 1 | 1 | 3
  Blood Bilirubin Increased, Grade 0, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Blood Bilirubin Increased, Grade 0, Grade 4 | 0 | 1 | 1
  Blood Bilirubin Increased, Grade 1, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Blood Bilirubin Increased, Grade 1, Grade 0 | 0 | 1 | 0
  Blood Bilirubin Increased, Grade 1, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Blood Bilirubin Increased, Grade 1, Grade 2 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 1, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Blood Bilirubin Increased, Grade 1, Grade 3 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 1, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Blood Bilirubin Increased, Grade 1, Grade 4 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 2, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Blood Bilirubin Increased, Grade 2, Grade 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 2, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Blood Bilirubin Increased, Grade 2, Grade 1 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 2, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Blood Bilirubin Increased, Grade 2, Grade 3 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 2, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Blood Bilirubin Increased, Grade 2, Grade 4 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 3, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Blood Bilirubin Increased, Grade 3, Grade 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 3, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Blood Bilirubin Increased, Grade 3, Grade 1 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 3, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Blood Bilirubin Increased, Grade 3, Grade 2 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 3, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Blood Bilirubin Increased, Grade 3, Grade 4 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 4, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Blood Bilirubin Increased, Grade 4, Grade 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 4, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Blood Bilirubin Increased, Grade 4, Grade 1 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 4, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Blood Bilirubin Increased, Grade 4, Grade 2 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 4, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Blood Bilirubin Increased, Grade 4, Grade 3 | 0 | 0 | 0
  Blood Bilirubin Increased, Missing, Grade 0: number analyzed (Participants) | 0 | 113 | 0
  Blood Bilirubin Increased, Missing, Grade 0 |  | 2 |
  Blood Bilirubin Increased, Missing, Grade 1: number analyzed (Participants) | 0 | 113 | 0
  Blood Bilirubin Increased, Missing, Grade 1 |  | 0 |
  Blood Bilirubin Increased, Missing, Grade 2: number analyzed (Participants) | 0 | 113 | 0
  Blood Bilirubin Increased, Missing, Grade 2 |  | 0 |
  Blood Bilirubin Increased, Missing, Grade 3: number analyzed (Participants) | 0 | 113 | 0
  Blood Bilirubin Increased, Missing, Grade 3 |  | 1 |
  Blood Bilirubin Increased, Missing, Grade 4: number analyzed (Participants) | 0 | 113 | 0
  Blood Bilirubin Increased, Missing, Grade 4 |  | 0 |
  Creatinine Increased, Grade 0, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Creatinine Increased, Grade 0, Grade 1 | 2 | 11 | 9
  Creatinine Increased, Grade 0, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Creatinine Increased, Grade 0, Grade 2 | 0 | 0 | 1
  Creatinine Increased, Grade 0, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Creatinine Increased, Grade 0, Grade 3 | 0 | 2 | 0
  Creatinine Increased, Grade 0, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Creatinine Increased, Grade 0, Grade 4 | 0 | 1 | 0
  Creatinine Increased, Grade 1, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Creatinine Increased, Grade 1, Grade 0 | 0 | 2 | 1
  Creatinine Increased, Grade 1, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Creatinine Increased, Grade 1, Grade 2 | 1 | 4 | 0
  Creatinine Increased, Grade 1, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Creatinine Increased, Grade 1, Grade 3 | 0 | 0 | 0
  Creatinine Increased, Grade 1, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Creatinine Increased, Grade 1, Grade 4 | 0 | 0 | 0
  Creatinine Increased, Grade 2, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Creatinine Increased, Grade 2, Grade 0 | 0 | 0 | 0
  Creatinine Increased, Grade 2, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Creatinine Increased, Grade 2, Grade 1 | 0 | 0 | 0
  Creatinine Increased, Grade 2, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Creatinine Increased, Grade 2, Grade 3 | 0 | 0 | 0
  Creatinine Increased, Grade 2, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Creatinine Increased, Grade 2, Grade 4 | 0 | 0 | 0
  Creatinine Increased, Grade 3, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Creatinine Increased, Grade 3, Grade 0 | 0 | 0 | 0
  Creatinine Increased, Grade 3, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Creatinine Increased, Grade 3, Grade 1 | 0 | 0 | 0
  Creatinine Increased, Grade 3, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Creatinine Increased, Grade 3, Grade 2 | 0 | 0 | 0
  Creatinine Increased, Grade 3, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Creatinine Increased, Grade 3, Grade 4 | 0 | 0 | 0
  Creatinine Increased, Grade 4, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Creatinine Increased, Grade 4, Grade 0 | 0 | 0 | 0
  Creatinine Increased, Grade 4, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Creatinine Increased, Grade 4, Grade 1 | 0 | 0 | 0
  Creatinine Increased, Grade 4, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Creatinine Increased, Grade 4, Grade 2 | 0 | 0 | 0
  Creatinine Increased, Grade 4, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Creatinine Increased, Grade 4, Grade 3 | 0 | 0 | 0
  Creatinine Increased, Missing, Grade 0: number analyzed (Participants) | 37 | 0 | 58
  Creatinine Increased, Missing, Grade 0 | 3 |  | 1
  Creatinine Increased, Missing, Grade 1: number analyzed (Participants) | 37 | 0 | 58
  Creatinine Increased, Missing, Grade 1 | 0 |  | 0
  Creatinine Increased, Missing, Grade 2: number analyzed (Participants) | 37 | 0 | 58
  Creatinine Increased, Missing, Grade 2 | 0 |  | 0
  Creatinine Increased, Missing, Grade 3: number analyzed (Participants) | 37 | 0 | 58
  Creatinine Increased, Missing, Grade 3 | 0 |  | 0
  Creatinine Increased, Missing, Grade 4: number analyzed (Participants) | 37 | 0 | 58
  Creatinine Increased, Missing, Grade 4 | 0 |  | 0
  Hypokalemia , Grade 0, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Hypokalemia , Grade 0, Grade 1 | 2 | 7 | 4
  Hypokalemia , Grade 0, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Hypokalemia , Grade 0, Grade 2 | 0 | 0 | 0
  Hypokalemia , Grade 0, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Hypokalemia , Grade 0, Grade 3 | 1 | 0 | 1
  Hypokalemia , Grade 0, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Hypokalemia , Grade 0, Grade 4 | 0 | 1 | 0
  Hypokalemia , Grade 1, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Hypokalemia , Grade 1, Grade 0 | 0 | 0 | 0
  Hypokalemia , Grade 1, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Hypokalemia , Grade 1, Grade 2 | 0 | 0 | 0
  Hypokalemia , Grade 1, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Hypokalemia , Grade 1, Grade 3 | 0 | 0 | 1
  Hypokalemia , Grade 1, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Hypokalemia , Grade 1, Grade 4 | 0 | 0 | 0
  Hypokalemia , Grade 2, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Hypokalemia , Grade 2, Grade 0 | 0 | 0 | 0
  Hypokalemia , Grade 2, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Hypokalemia , Grade 2, Grade 1 | 0 | 0 | 0
  Hypokalemia , Grade 2, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Hypokalemia , Grade 2, Grade 3 | 0 | 0 | 0
  Hypokalemia , Grade 2, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Hypokalemia , Grade 2, Grade 4 | 0 | 0 | 0
  Hypokalemia , Grade 3, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Hypokalemia , Grade 3, Grade 0 | 0 | 0 | 0
  Hypokalemia , Grade 3, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Hypokalemia , Grade 3, Grade 1 | 0 | 0 | 0
  Hypokalemia , Grade 3, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Hypokalemia , Grade 3, Grade 2 | 0 | 0 | 0
  Hypokalemia , Grade 3, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Hypokalemia , Grade 3, Grade 4 | 0 | 0 | 0
  Hypokalemia , Grade 4, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Hypokalemia , Grade 4, Grade 0 | 0 | 0 | 0
  Hypokalemia , Grade 4, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Hypokalemia , Grade 4, Grade 1 | 0 | 0 | 0
  Hypokalemia , Grade 4, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Hypokalemia , Grade 4, Grade 2 | 0 | 0 | 0
  Hypokalemia , Grade 4, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Hypokalemia , Grade 4, Grade 3 | 0 | 0 | 0
  Hyperkalemia , Grade 0, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Hyperkalemia , Grade 0, Grade 1 | 1 | 19 | 6
  Hyperkalemia , Grade 0, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Hyperkalemia , Grade 0, Grade 2 | 2 | 5 | 2
  Hyperkalemia , Grade 0, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Hyperkalemia , Grade 0, Grade 3 | 0 | 1 | 0
  Hyperkalemia , Grade 0, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Hyperkalemia , Grade 0, Grade 4 | 1 | 0 | 2
  Hyperkalemia , Grade 1, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Hyperkalemia , Grade 1, Grade 0 | 0 | 0 | 1
  Hyperkalemia , Grade 1, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Hyperkalemia , Grade 1, Grade 2 | 0 | 0 | 0
  Hyperkalemia , Grade 1, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Hyperkalemia , Grade 1, Grade 3 | 0 | 0 | 0
  Hyperkalemia , Grade 1, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Hyperkalemia , Grade 1, Grade 4 | 0 | 0 | 0
  Hyperkalemia , Grade 2, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Hyperkalemia , Grade 2, Grade 0 | 0 | 0 | 0
  Hyperkalemia , Grade 2, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Hyperkalemia , Grade 2, Grade 1 | 0 | 0 | 0
  Hyperkalemia , Grade 2, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Hyperkalemia , Grade 2, Grade 3 | 0 | 0 | 0
  Hyperkalemia , Grade 2, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Hyperkalemia , Grade 2, Grade 4 | 0 | 0 | 0
  Hyperkalemia , Grade 3, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Hyperkalemia , Grade 3, Grade 0 | 0 | 0 | 0
  Hyperkalemia , Grade 3, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Hyperkalemia , Grade 3, Grade 1 | 0 | 0 | 0
  Hyperkalemia , Grade 3, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Hyperkalemia , Grade 3, Grade 2 | 0 | 0 | 0
  Hyperkalemia , Grade 3, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Hyperkalemia , Grade 3, Grade 4 | 0 | 0 | 0
  Hyperkalemia , Grade 4, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Hyperkalemia , Grade 4, Grade 0 | 0 | 0 | 0
  Hyperkalemia , Grade 4, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Hyperkalemia , Grade 4, Grade 1 | 0 | 0 | 0
  Hyperkalemia , Grade 4, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Hyperkalemia , Grade 4, Grade 2 | 0 | 0 | 0
  Hyperkalemia , Grade 4, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Hyperkalemia , Grade 4, Grade 3 | 0 | 0 | 0
  Hyponatremia , Grade 0, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Hyponatremia , Grade 0, Grade 1 | 7 | 24 | 12
  Hyponatremia , Grade 0, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Hyponatremia , Grade 0, Grade 2 | 0 | 0 | 0
  Hyponatremia , Grade 0, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Hyponatremia , Grade 0, Grade 3 | 1 | 4 | 3
  Hyponatremia , Grade 0, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Hyponatremia , Grade 0, Grade 4 | 1 | 1 | 2
  Hyponatremia , Grade 1, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Hyponatremia , Grade 1, Grade 0 | 1 | 1 | 0
  Hyponatremia , Grade 1, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Hyponatremia , Grade 1, Grade 2 | 0 | 0 | 0
  Hyponatremia , Grade 1, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Hyponatremia , Grade 1, Grade 3 | 0 | 2 | 0
  Hyponatremia , Grade 1, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Hyponatremia , Grade 1, Grade 4 | 0 | 0 | 1
  Hyponatremia , Grade 2, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Hyponatremia , Grade 2, Grade 0 | 0 | 0 | 0
  Hyponatremia , Grade 2, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Hyponatremia , Grade 2, Grade 1 | 0 | 0 | 0
  Hyponatremia , Grade 2, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Hyponatremia , Grade 2, Grade 3 | 0 | 0 | 0
  Hyponatremia , Grade 2, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Hyponatremia , Grade 2, Grade 4 | 0 | 0 | 0
  Hyponatremia , Grade 3, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Hyponatremia , Grade 3, Grade 0 | 0 | 0 | 1
  Hyponatremia , Grade 3, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Hyponatremia , Grade 3, Grade 1 | 0 | 0 | 0
  Hyponatremia , Grade 3, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Hyponatremia , Grade 3, Grade 2 | 0 | 0 | 0
  Hyponatremia , Grade 3, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Hyponatremia , Grade 3, Grade 4 | 0 | 0 | 0
  Hyponatremia , Grade 4, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Hyponatremia , Grade 4, Grade 0 | 0 | 0 | 0
  Hyponatremia , Grade 4, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Hyponatremia , Grade 4, Grade 1 | 0 | 0 | 0
  Hyponatremia , Grade 4, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Hyponatremia , Grade 4, Grade 2 | 0 | 0 | 0
  Hyponatremia , Grade 4, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Hyponatremia , Grade 4, Grade 3 | 0 | 0 | 0
  Hypernatremia , Grade 0, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Hypernatremia , Grade 0, Grade 1 | 3 | 5 | 1
  Hypernatremia , Grade 0, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Hypernatremia , Grade 0, Grade 2 | 0 | 0 | 0
  Hypernatremia , Grade 0, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Hypernatremia , Grade 0, Grade 3 | 0 | 0 | 0
  Hypernatremia , Grade 0, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Hypernatremia , Grade 0, Grade 4 | 0 | 0 | 0
  Hypernatremia , Grade 1, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Hypernatremia , Grade 1, Grade 0 | 0 | 0 | 0
  Hypernatremia , Grade 1, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Hypernatremia , Grade 1, Grade 2 | 0 | 0 | 0
  Hypernatremia , Grade 1, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Hypernatremia , Grade 1, Grade 3 | 0 | 0 | 0
  Hypernatremia , Grade 1, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Hypernatremia , Grade 1, Grade 4 | 0 | 0 | 0
  Hypernatremia , Grade 2, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Hypernatremia , Grade 2, Grade 0 | 0 | 0 | 0
  Hypernatremia , Grade 2, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Hypernatremia , Grade 2, Grade 1 | 0 | 0 | 0
  Hypernatremia , Grade 2, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Hypernatremia , Grade 2, Grade 3 | 0 | 0 | 0
  Hypernatremia , Grade 2, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Hypernatremia , Grade 2, Grade 4 | 0 | 0 | 0
  Hypernatremia , Grade 3, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Hypernatremia , Grade 3, Grade 0 | 0 | 0 | 0
  Hypernatremia , Grade 3, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Hypernatremia , Grade 3, Grade 1 | 0 | 0 | 0
  Hypernatremia , Grade 3, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Hypernatremia , Grade 3, Grade 2 | 0 | 0 | 0
  Hypernatremia , Grade 3, Grade 4: number analyzed (Participants) | 37 | 113 | 58
  Hypernatremia , Grade 3, Grade 4 | 0 | 0 | 0
  Hypernatremia , Grade 4, Grade 0: number analyzed (Participants) | 37 | 113 | 58
  Hypernatremia , Grade 4, Grade 0 | 0 | 0 | 0
  Hypernatremia , Grade 4, Grade 1: number analyzed (Participants) | 37 | 113 | 58
  Hypernatremia , Grade 4, Grade 1 | 0 | 0 | 0
  Hypernatremia , Grade 4, Grade 2: number analyzed (Participants) | 37 | 113 | 58
  Hypernatremia , Grade 4, Grade 2 | 0 | 0 | 0
  Hypernatremia , Grade 4, Grade 3: number analyzed (Participants) | 37 | 113 | 58
  Hypernatremia , Grade 4, Grade 3 | 0 | 0 | 0
  Hypocalcemia , Grade 0, Grade 1: number analyzed (Participants) | 37 | 112 | 58
  Hypocalcemia , Grade 0, Grade 1 | 1 | 9 | 3
  Hypocalcemia , Grade 0, Grade 2: number analyzed (Participants) | 37 | 112 | 58
  Hypocalcemia , Grade 0, Grade 2 | 1 | 0 | 0
  Hypocalcemia , Grade 0, Grade 3: number analyzed (Participants) | 37 | 112 | 58
  Hypocalcemia , Grade 0, Grade 3 | 0 | 2 | 1
  Hypocalcemia , Grade 0, Grade 4: number analyzed (Participants) | 37 | 112 | 58
  Hypocalcemia , Grade 0, Grade 4 | 2 | 1 | 0
  Hypocalcemia , Grade 1, Grade 0: number analyzed (Participants) | 37 | 112 | 58
  Hypocalcemia , Grade 1, Grade 0 | 0 | 2 | 2
  Hypocalcemia , Grade 1, Grade 2: number analyzed (Participants) | 37 | 112 | 58
  Hypocalcemia , Grade 1, Grade 2 | 0 | 0 | 0
  Hypocalcemia , Grade 1, Grade 3: number analyzed (Participants) | 37 | 112 | 58
  Hypocalcemia , Grade 1, Grade 3 | 0 | 0 | 0
  Hypocalcemia , Grade 1, Grade 4: number analyzed (Participants) | 37 | 112 | 58
  Hypocalcemia , Grade 1, Grade 4 | 0 | 0 | 0
  Hypocalcemia , Grade 2, Grade 0: number analyzed (Participants) | 37 | 112 | 58
  Hypocalcemia , Grade 2, Grade 0 | 0 | 1 | 0
  Hypocalcemia , Grade 2, Grade 1: number analyzed (Participants) | 37 | 112 | 58
  Hypocalcemia , Grade 2, Grade 1 | 0 | 1 | 0
  Hypocalcemia , Grade 2, Grade 3: number analyzed (Participants) | 37 | 112 | 58
  Hypocalcemia , Grade 2, Grade 3 | 0 | 0 | 0
  Hypocalcemia , Grade 2, Grade 4: number analyzed (Participants) | 37 | 112 | 58
  Hypocalcemia , Grade 2, Grade 4 | 0 | 0 | 0
  Hypocalcemia , Grade 3, Grade 0: number analyzed (Participants) | 37 | 112 | 58
  Hypocalcemia , Grade 3, Grade 0 | 0 | 0 | 0
  Hypocalcemia , Grade 3, Grade 1: number analyzed (Participants) | 37 | 112 | 58
  Hypocalcemia , Grade 3, Grade 1 | 0 | 0 | 0
  Hypocalcemia , Grade 3, Grade 2: number analyzed (Participants) | 37 | 112 | 58
  Hypocalcemia , Grade 3, Grade 2 | 0 | 0 | 0
  Hypocalcemia , Grade 3, Grade 4: number analyzed (Participants) | 37 | 112 | 58
  Hypocalcemia , Grade 3, Grade 4 | 0 | 0 | 0
  Hypocalcemia , Grade 4, Grade 0: number analyzed (Participants) | 37 | 112 | 58
  Hypocalcemia , Grade 4, Grade 0 | 0 | 0 | 0
  Hypocalcemia , Grade 4, Grade 1: number analyzed (Participants) | 37 | 112 | 58
  Hypocalcemia , Grade 4, Grade 1 | 0 | 0 | 0
  Hypocalcemia , Grade 4, Grade 2: number analyzed (Participants) | 37 | 112 | 58
  Hypocalcemia , Grade 4, Grade 2 | 0 | 0 | 0
  Hypocalcemia , Grade 4, Grade 3: number analyzed (Participants) | 37 | 112 | 58
  Hypocalcemia , Grade 4, Grade 3 | 0 | 0 | 0
  Hypocalcemia , Missing, Grade 0: number analyzed (Participants) | 0 | 112 | 0
  Hypocalcemia , Missing, Grade 0 |  | 1 |
  Hypocalcemia , Missing, Grade 1: number analyzed (Participants) | 0 | 112 | 0
  Hypocalcemia , Missing, Grade 1 |  | 0 |
  Hypocalcemia , Missing, Grade 2: number analyzed (Participants) | 0 | 112 | 0
  Hypocalcemia , Missing, Grade 2 |  | 0 |
  Hypocalcemia , Missing, Grade 3: number analyzed (Participants) | 0 | 112 | 0
  Hypocalcemia , Missing, Grade 3 |  | 0 |
  Hypocalcemia , Missing, Grade 4: number analyzed (Participants) | 0 | 112 | 0
  Hypocalcemia , Missing, Grade 4 |  | 0 |
  Hypercalcemia , Grade 0, Grade 1: number analyzed (Participants) | 37 | 112 | 58
  Hypercalcemia , Grade 0, Grade 1 | 5 | 5 | 6
  Hypercalcemia , Grade 0, Grade 2: number analyzed (Participants) | 37 | 112 | 58
  Hypercalcemia , Grade 0, Grade 2 | 0 | 0 | 1
  Hypercalcemia , Grade 0, Grade 3: number analyzed (Participants) | 37 | 112 | 58
  Hypercalcemia , Grade 0, Grade 3 | 0 | 1 | 1
  Hypercalcemia , Grade 0, Grade 4: number analyzed (Participants) | 37 | 112 | 58
  Hypercalcemia , Grade 0, Grade 4 | 0 | 1 | 0
  Hypercalcemia , Grade 1, Grade 0: number analyzed (Participants) | 37 | 112 | 58
  Hypercalcemia , Grade 1, Grade 0 | 0 | 0 | 0
  Hypercalcemia , Grade 1, Grade 2: number analyzed (Participants) | 37 | 112 | 58
  Hypercalcemia , Grade 1, Grade 2 | 0 | 2 | 0
  Hypercalcemia , Grade 1, Grade 3: number analyzed (Participants) | 37 | 112 | 58
  Hypercalcemia , Grade 1, Grade 3 | 0 | 1 | 1
  Hypercalcemia , Grade 1, Grade 4: number analyzed (Participants) | 37 | 112 | 58
  Hypercalcemia , Grade 1, Grade 4 | 0 | 0 | 0
  Hypercalcemia , Grade 2, Grade 0: number analyzed (Participants) | 37 | 112 | 58
  Hypercalcemia , Grade 2, Grade 0 | 0 | 0 | 1
  Hypercalcemia , Grade 2, Grade 1: number analyzed (Participants) | 37 | 112 | 58
  Hypercalcemia , Grade 2, Grade 1 | 0 | 0 | 0
  Hypercalcemia , Grade 2, Grade 3: number analyzed (Participants) | 37 | 112 | 58
  Hypercalcemia , Grade 2, Grade 3 | 0 | 0 | 1
  Hypercalcemia , Grade 2, Grade 4: number analyzed (Participants) | 37 | 112 | 58
  Hypercalcemia , Grade 2, Grade 4 | 0 | 0 | 0
  Hypercalcemia , Grade 3, Grade 0: number analyzed (Participants) | 37 | 112 | 58
  Hypercalcemia , Grade 3, Grade 0 | 0 | 0 | 0
  Hypercalcemia , Grade 3, Grade 1: number analyzed (Participants) | 37 | 112 | 58
  Hypercalcemia , Grade 3, Grade 1 | 0 | 0 | 0
  Hypercalcemia , Grade 3, Grade 2: number analyzed (Participants) | 37 | 112 | 58
  Hypercalcemia , Grade 3, Grade 2 | 0 | 0 | 0
  Hypercalcemia , Grade 3, Grade 4: number analyzed (Participants) | 37 | 112 | 58
  Hypercalcemia , Grade 3, Grade 4 | 1 | 0 | 0
  Hypercalcemia , Grade 4, Grade 0: number analyzed (Participants) | 37 | 112 | 58
  Hypercalcemia , Grade 4, Grade 0 | 0 | 0 | 0
  Hypercalcemia , Grade 4, Grade 1: number analyzed (Participants) | 37 | 112 | 58
  Hypercalcemia , Grade 4, Grade 1 | 0 | 0 | 0
  Hypercalcemia , Grade 4, Grade 2: number analyzed (Participants) | 37 | 112 | 58
  Hypercalcemia , Grade 4, Grade 2 | 0 | 0 | 0
  Hypercalcemia , Grade 4, Grade 3: number analyzed (Participants) | 37 | 112 | 58
  Hypercalcemia , Grade 4, Grade 3 | 0 | 0 | 0
  Hypercalcemia , Missing, Grade 0: number analyzed (Participants) | 0 | 112 | 0
  Hypercalcemia , Missing, Grade 0 |  | 1 |
  Hypercalcemia , Missing, Grade 1: number analyzed (Participants) | 0 | 112 | 0
  Hypercalcemia , Missing, Grade 1 |  | 0 |
  Hypercalcemia , Missing, Grade 2: number analyzed (Participants) | 0 | 112 | 0
  Hypercalcemia , Missing, Grade 2 |  | 0 |
  Hypercalcemia , Missing, Grade 3: number analyzed (Participants) | 0 | 112 | 0
  Hypercalcemia , Missing, Grade 3 |  | 0 |
  Hypercalcemia , Missing, Grade 4: number analyzed (Participants) | 0 | 112 | 0
  Hypercalcemia , Missing, Grade 4 |  | 0 |
  Chronic Kidney Disease , Grade 0, Grade 1: number analyzed (Participants) | 8 | 47 | 12
  Chronic Kidney Disease , Grade 0, Grade 1 | 0 | 0 | 0
  Chronic Kidney Disease , Grade 0, Grade 2: number analyzed (Participants) | 8 | 47 | 12
  Chronic Kidney Disease , Grade 0, Grade 2 | 1 | 4 | 0
  Chronic Kidney Disease , Grade 0, Grade 3: number analyzed (Participants) | 8 | 47 | 12
  Chronic Kidney Disease , Grade 0, Grade 3 | 0 | 0 | 0
  Chronic Kidney Disease , Grade 0, Grade 4: number analyzed (Participants) | 8 | 47 | 12
  Chronic Kidney Disease , Grade 0, Grade 4 | 0 | 1 | 3
  Chronic Kidney Disease , Grade 1, Grade 0: number analyzed (Participants) | 8 | 47 | 12
  Chronic Kidney Disease , Grade 1, Grade 0 | 0 | 1 | 0
  Chronic Kidney Disease , Grade 1, Grade 2: number analyzed (Participants) | 8 | 47 | 12
  Chronic Kidney Disease , Grade 1, Grade 2 | 0 | 2 | 0
  Chronic Kidney Disease , Grade 1, Grade 3: number analyzed (Participants) | 8 | 47 | 12
  Chronic Kidney Disease , Grade 1, Grade 3 | 0 | 0 | 0
  Chronic Kidney Disease , Grade 1, Grade 4: number analyzed (Participants) | 8 | 47 | 12
  Chronic Kidney Disease , Grade 1, Grade 4 | 0 | 0 | 0
  Chronic Kidney Disease , Grade 2, Grade 0: number analyzed (Participants) | 8 | 47 | 12
  Chronic Kidney Disease , Grade 2, Grade 0 | 0 | 0 | 0
  Chronic Kidney Disease , Grade 2, Grade 1: number analyzed (Participants) | 8 | 47 | 12
  Chronic Kidney Disease , Grade 2, Grade 1 | 0 | 1 | 0
  Chronic Kidney Disease , Grade 2, Grade 2: number analyzed (Participants) | 8 | 47 | 12
  Chronic Kidney Disease , Grade 2, Grade 2 | 1 | 7 | 2
  Chronic Kidney Disease , Grade 2, Grade 3: number analyzed (Participants) | 8 | 47 | 12
  Chronic Kidney Disease , Grade 2, Grade 3 | 0 | 1 | 0
  Chronic Kidney Disease , Grade 2, Grade 4: number analyzed (Participants) | 8 | 47 | 12
  Chronic Kidney Disease , Grade 2, Grade 4 | 0 | 0 | 0
  Chronic Kidney Disease , Grade 3, Grade 0: number analyzed (Participants) | 8 | 47 | 12
  Chronic Kidney Disease , Grade 3, Grade 0 | 0 | 0 | 0
  Chronic Kidney Disease , Grade 3, Grade 1: number analyzed (Participants) | 8 | 47 | 12
  Chronic Kidney Disease , Grade 3, Grade 1 | 0 | 0 | 0
  Chronic Kidney Disease , Grade 3, Grade 2: number analyzed (Participants) | 8 | 47 | 12
  Chronic Kidney Disease , Grade 3, Grade 2 | 0 | 0 | 0
  Chronic Kidney Disease , Grade 3, Grade 4: number analyzed (Participants) | 8 | 47 | 12
  Chronic Kidney Disease , Grade 3, Grade 4 | 0 | 0 | 0
  Chronic Kidney Disease , Grade 4, Grade 0: number analyzed (Participants) | 8 | 47 | 12
  Chronic Kidney Disease , Grade 4, Grade 0 | 0 | 0 | 0
  Chronic Kidney Disease , Grade 4, Grade 1: number analyzed (Participants) | 8 | 47 | 12
  Chronic Kidney Disease , Grade 4, Grade 1 | 0 | 0 | 0
  Chronic Kidney Disease , Grade 4, Grade 2: number analyzed (Participants) | 8 | 47 | 12
  Chronic Kidney Disease , Grade 4, Grade 2 | 0 | 0 | 0
  Chronic Kidney Disease , Grade 4, Grade 3: number analyzed (Participants) | 8 | 47 | 12
  Chronic Kidney Disease , Grade 4, Grade 3 | 0 | 0 | 0
  Chronic Kidney Disease , Missing, Grade 0: number analyzed (Participants) | 8 | 47 | 12
  Chronic Kidney Disease , Missing, Grade 0 | 1 | 2 | 0
  Chronic Kidney Disease , Missing, Grade 1: number analyzed (Participants) | 8 | 47 | 12
  Chronic Kidney Disease , Missing, Grade 1 | 1 | 4 | 3
  Chronic Kidney Disease , Missing, Grade 2: number analyzed (Participants) | 8 | 47 | 12
  Chronic Kidney Disease , Missing, Grade 2 | 0 | 1 | 1
  Chronic Kidney Disease , Missing, Grade 3: number analyzed (Participants) | 8 | 47 | 12
  Chronic Kidney Disease , Missing, Grade 3 | 0 | 0 | 0
  Chronic Kidney Disease , Missing, Grade 4: number analyzed (Participants) | 8 | 47 | 12
  Chronic Kidney Disease , Missing, Grade 4 | 0 | 1 | 0

19. Secondary Outcome: Part 1B: Number of Participants With Worst Case Chemistry Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: as for outcome 12
Time Frame: Up to approximately 367 weeks
Population: All Treated Population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1B: Fela 0.300 mg/kg | Part 1B: Fela 1.000 mg/kg | Part 1B: Fela 24 mg
Number analyzed (Participants) | 39 | 115 | 59
Participants
  Lactate Dehydrogenase (IU/L), To Low: number analyzed (Participants) | 1 | 0 | 4
  Lactate Dehydrogenase (IU/L), To Low | 0 |  | 0
  Lactate Dehydrogenase (IU/L), To Normal or No Change: number analyzed (Participants) | 1 | 0 | 4
  Lactate Dehydrogenase (IU/L), To Normal or No Change | 1 |  | 3
  Lactate Dehydrogenase (IU/L), To High: number analyzed (Participants) | 1 | 0 | 4
  Lactate Dehydrogenase (IU/L), To High | 0 |  | 1
  Protein (g/L), To Low: number analyzed (Participants) | 37 | 113 | 58
  Protein (g/L), To Low | 1 | 22 | 9
  Protein (g/L), To Normal or No Change: number analyzed (Participants) | 37 | 113 | 58
  Protein (g/L), To Normal or No Change | 34 | 80 | 45
  Protein (g/L), To High: number analyzed (Participants) | 37 | 113 | 58
  Protein (g/L), To High | 2 | 11 | 4
  Triiodothyronine, Free (pmol/L), To Low: number analyzed (Participants) | 30 | 104 | 51
  Triiodothyronine, Free (pmol/L), To Low | 5 | 15 | 10
  Triiodothyronine, Free (pmol/L), To Normal or No Change: number analyzed (Participants) | 30 | 104 | 51
  Triiodothyronine, Free (pmol/L), To Normal or No Change | 23 | 74 | 37
  Triiodothyronine, Free (pmol/L), To High: number analyzed (Participants) | 30 | 104 | 51
  Triiodothyronine, Free (pmol/L), To High | 2 | 16 | 4
  Thyroxine, Free (pmol/L), To Low: number analyzed (Participants) | 31 | 103 | 51
  Thyroxine, Free (pmol/L), To Low | 2 | 14 | 5
  Thyroxine, Free (pmol/L), To Normal or No Change: number analyzed (Participants) | 31 | 103 | 51
  Thyroxine, Free (pmol/L), To Normal or No Change | 27 | 78 | 44
  Thyroxine, Free (pmol/L), To High: number analyzed (Participants) | 31 | 103 | 51
  Thyroxine, Free (pmol/L), To High | 2 | 12 | 2
  Troponin I (ug/L), To Low: number analyzed (Participants) | 14 | 34 | 19
  Troponin I (ug/L), To Low | 0 | 1 | 0
  Troponin I (ug/L), To Normal or No Change: number analyzed (Participants) | 14 | 34 | 19
  Troponin I (ug/L), To Normal or No Change | 12 | 27 | 15
  Troponin I (ug/L), To High: number analyzed (Participants) | 14 | 34 | 19
  Troponin I (ug/L), To High | 2 | 6 | 4
  Troponin T (ug/L), To Low: number analyzed (Participants) | 19 | 43 | 32
  Troponin T (ug/L), To Low | 0 | 0 | 0
  Troponin T (ug/L), To Normal or No Change: number analyzed (Participants) | 19 | 43 | 32
  Troponin T (ug/L), To Normal or No Change | 18 | 35 | 30
  Troponin T (ug/L), To High: number analyzed (Participants) | 19 | 43 | 32
  Troponin T (ug/L), To High | 1 | 8 | 2
  Thyrotropin (mU/L), To Low: number analyzed (Participants) | 31 | 105 | 51
  Thyrotropin (mU/L), To Low | 3 | 4 | 1
  Thyrotropin (mU/L), To Normal or No Change: number analyzed (Participants) | 31 | 105 | 51
  Thyrotropin (mU/L), To Normal or No Change | 23 | 82 | 41
  Thyrotropin (mU/L), To High: number analyzed (Participants) | 31 | 105 | 51
  Thyrotropin (mU/L), To High | 5 | 19 | 9
  Urea (mmol/L), To Low: number analyzed (Participants) | 33 | 89 | 38
  Urea (mmol/L), To Low | 1 | 10 | 2
  Urea (mmol/L), To Normal or No Change: number analyzed (Participants) | 33 | 89 | 38
  Urea (mmol/L), To Normal or No Change | 26 | 53 | 28
  Urea (mmol/L), To High: number analyzed (Participants) | 33 | 89 | 38
  Urea (mmol/L), To High | 6 | 30 | 9

20. Secondary Outcome: Part 1B: Number of Participants With Worst-case Grade Change From Baseline in Hematology Parameters
Description: as for outcome 5
Time Frame: Baseline (Day 1) and up to approximately 367 weeks
Population: All Treated Population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1B: Fela 0.300 mg/kg | Part 1B: Fela 1.000 mg/kg | Part 1B: Fela 24 mg
Number analyzed (Participants) | 39 | 115 | 59
Participants
  Anemia , Grade 0, Grade 1: number analyzed (Participants) | 37 | 114 | 58
  Anemia , Grade 0, Grade 1 | 4 | 22 | 7
  Anemia , Grade 0, Grade 2: number analyzed (Participants) | 37 | 114 | 58
  Anemia , Grade 0, Grade 2 | 2 | 7 | 5
  Anemia , Grade 0, Grade 3: number analyzed (Participants) | 37 | 114 | 58
  Anemia , Grade 0, Grade 3 | 0 | 4 | 1
  Anemia , Grade 0, Grade 4: number analyzed (Participants) | 37 | 114 | 58
  Anemia , Grade 0, Grade 4 | 0 | 0 | 0
  Anemia , Grade 1, Grade 0: number analyzed (Participants) | 37 | 114 | 58
  Anemia , Grade 1, Grade 0 | 0 | 1 | 1
  Anemia , Grade 1, Grade 2: number analyzed (Participants) | 37 | 114 | 58
  Anemia , Grade 1, Grade 2 | 6 | 20 | 8
  Anemia , Grade 1, Grade 3: number analyzed (Participants) | 37 | 114 | 58
  Anemia , Grade 1, Grade 3 | 0 | 2 | 1
  Anemia , Grade 1, Grade 4: number analyzed (Participants) | 37 | 114 | 58
  Anemia , Grade 1, Grade 4 | 0 | 0 | 0
  Anemia , Grade 2, Grade 0: number analyzed (Participants) | 37 | 114 | 58
  Anemia , Grade 2, Grade 0 | 0 | 0 | 0
  Anemia , Grade 2, Grade 1: number analyzed (Participants) | 37 | 114 | 58
  Anemia , Grade 2, Grade 1 | 0 | 0 | 0
  Anemia , Grade 2, Grade 3: number analyzed (Participants) | 37 | 114 | 58
  Anemia , Grade 2, Grade 3 | 1 | 8 | 4
  Anemia , Grade 2, Grade 4: number analyzed (Participants) | 37 | 114 | 58
  Anemia , Grade 2, Grade 4 | 0 | 0 | 0
  Anemia , Grade 3, Grade 0: number analyzed (Participants) | 37 | 114 | 58
  Anemia , Grade 3, Grade 0 | 0 | 0 | 0
  Anemia , Grade 3, Grade 1: number analyzed (Participants) | 37 | 114 | 58
  Anemia , Grade 3, Grade 1 | 0 | 0 | 0
  Anemia , Grade 3, Grade 2: number analyzed (Participants) | 37 | 114 | 58
  Anemia , Grade 3, Grade 2 | 0 | 0 | 0
  Anemia , Grade 3, Grade 4: number analyzed (Participants) | 37 | 114 | 58
  Anemia , Grade 3, Grade 4 | 0 | 0 | 0
  Anemia , Grade 4, Grade 0: number analyzed (Participants) | 37 | 114 | 58
  Anemia , Grade 4, Grade 0 | 0 | 0 | 0
  Anemia , Grade 4, Grade 1: number analyzed (Participants) | 37 | 114 | 58
  Anemia , Grade 4, Grade 1 | 0 | 0 | 0
  Anemia , Grade 4, Grade 2: number analyzed (Participants) | 37 | 114 | 58
  Anemia , Grade 4, Grade 2 | 0 | 0 | 0
  Anemia , Grade 4, Grade 3: number analyzed (Participants) | 37 | 114 | 58
  Anemia , Grade 4, Grade 3 | 0 | 0 | 0
  Hemoglobin Increased, Grade 0, Grade 1: number analyzed (Participants) | 37 | 114 | 58
  Hemoglobin Increased, Grade 0, Grade 1 | 0 | 0 | 0
  Hemoglobin Increased, Grade 0, Grade 2: number analyzed (Participants) | 37 | 114 | 58
  Hemoglobin Increased, Grade 0, Grade 2 | 0 | 0 | 0
  Hemoglobin Increased, Grade 0, Grade 3: number analyzed (Participants) | 37 | 114 | 58
  Hemoglobin Increased, Grade 0, Grade 3 | 0 | 0 | 1
  Hemoglobin Increased, Grade 0, Grade 4: number analyzed (Participants) | 37 | 114 | 58
  Hemoglobin Increased, Grade 0, Grade 4 | 0 | 0 | 0
  Hemoglobin Increased, Grade 1, Grade 0: number analyzed (Participants) | 37 | 114 | 58
  Hemoglobin Increased, Grade 1, Grade 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 1, Grade 2: number analyzed (Participants) | 37 | 114 | 58
  Hemoglobin Increased, Grade 1, Grade 2 | 0 | 0 | 0
  Hemoglobin Increased, Grade 1, Grade 3: number analyzed (Participants) | 37 | 114 | 58
  Hemoglobin Increased, Grade 1, Grade 3 | 0 | 0 | 0
  Hemoglobin Increased, Grade 1, Grade 4: number analyzed (Participants) | 37 | 114 | 58
  Hemoglobin Increased, Grade 1, Grade 4 | 0 | 0 | 0
  Hemoglobin Increased, Grade 2, Grade 0: number analyzed (Participants) | 37 | 114 | 58
  Hemoglobin Increased, Grade 2, Grade 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 2, Grade 1: number analyzed (Participants) | 37 | 114 | 58
  Hemoglobin Increased, Grade 2, Grade 1 | 0 | 0 | 0
  Hemoglobin Increased, Grade 2, Grade 3: number analyzed (Participants) | 37 | 114 | 58
  Hemoglobin Increased, Grade 2, Grade 3 | 0 | 0 | 0
  Hemoglobin Increased, Grade 2, Grade 4: number analyzed (Participants) | 37 | 114 | 58
  Hemoglobin Increased, Grade 2, Grade 4 | 0 | 0 | 0
  Hemoglobin Increased, Grade 3, Grade 0: number analyzed (Participants) | 37 | 114 | 58
  Hemoglobin Increased, Grade 3, Grade 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 3, Grade 1: number analyzed (Participants) | 37 | 114 | 58
  Hemoglobin Increased, Grade 3, Grade 1 | 0 | 0 | 0
  Hemoglobin Increased, Grade 3, Grade 2: number analyzed (Participants) | 37 | 114 | 58
  Hemoglobin Increased, Grade 3, Grade 2 | 0 | 0 | 0
  Hemoglobin Increased, Grade 3, Grade 4: number analyzed (Participants) | 37 | 114 | 58
  Hemoglobin Increased, Grade 3, Grade 4 | 0 | 0 | 0
  Hemoglobin Increased, Grade 4, Grade 0: number analyzed (Participants) | 37 | 114 | 58
  Hemoglobin Increased, Grade 4, Grade 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 4, Grade 1: number analyzed (Participants) | 37 | 114 | 58
  Hemoglobin Increased, Grade 4, Grade 1 | 0 | 0 | 0
  Hemoglobin Increased, Grade 4, Grade 2: number analyzed (Participants) | 37 | 114 | 58
  Hemoglobin Increased, Grade 4, Grade 2 | 0 | 0 | 0
  Hemoglobin Increased, Grade 4, Grade 3: number analyzed (Participants) | 37 | 114 | 58
  Hemoglobin Increased, Grade 4, Grade 3 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 0, Grade 1: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Decreased, Grade 0, Grade 1 | 2 | 22 | 8
  Lymphocyte Count Decreased, Grade 0, Grade 2: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Decreased, Grade 0, Grade 2 | 1 | 10 | 6
  Lymphocyte Count Decreased, Grade 0, Grade 3: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Decreased, Grade 0, Grade 3 | 0 | 1 | 0
  Lymphocyte Count Decreased, Grade 0, Grade 4: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Decreased, Grade 0, Grade 4 | 0 | 1 | 0
  Lymphocyte Count Decreased, Grade 1, Grade 0: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Decreased, Grade 1, Grade 0 | 1 | 1 | 0
  Lymphocyte Count Decreased, Grade 1, Grade 2: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Decreased, Grade 1, Grade 2 | 5 | 15 | 7
  Lymphocyte Count Decreased, Grade 1, Grade 3: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Decreased, Grade 1, Grade 3 | 1 | 4 | 1
  Lymphocyte Count Decreased, Grade 1, Grade 4: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Decreased, Grade 1, Grade 4 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 2, Grade 0: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Decreased, Grade 2, Grade 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 2, Grade 1: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Decreased, Grade 2, Grade 1 | 1 | 0 | 0
  Lymphocyte Count Decreased, Grade 2, Grade 3: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Decreased, Grade 2, Grade 3 | 3 | 2 | 3
  Lymphocyte Count Decreased, Grade 2, Grade 4: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Decreased, Grade 2, Grade 4 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 3, Grade 0: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Decreased, Grade 3, Grade 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 3, Grade 1: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Decreased, Grade 3, Grade 1 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 3, Grade 2: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Decreased, Grade 3, Grade 2 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 3, Grade 4: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Decreased, Grade 3, Grade 4 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 4, Grade 0: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Decreased, Grade 4, Grade 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 4, Grade 1: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Decreased, Grade 4, Grade 1 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 4, Grade 2: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Decreased, Grade 4, Grade 2 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 4, Grade 3: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Decreased, Grade 4, Grade 3 | 0 | 0 | 0
  Lymphocyte Count Decreased, Missing, Grade 0: number analyzed (Participants) | 0 | 114 | 0
  Lymphocyte Count Decreased, Missing, Grade 0 |  | 0 |
  Lymphocyte Count Decreased, Missing, Grade 1: number analyzed (Participants) | 0 | 114 | 0
  Lymphocyte Count Decreased, Missing, Grade 1 |  | 1 |
  Lymphocyte Count Decreased, Missing, Grade 2: number analyzed (Participants) | 0 | 114 | 0
  Lymphocyte Count Decreased, Missing, Grade 2 |  | 3 |
  Lymphocyte Count Decreased, Missing, Grade 3: number analyzed (Participants) | 0 | 114 | 0
  Lymphocyte Count Decreased, Missing, Grade 3 |  | 0 |
  Lymphocyte Count Decreased, Missing, Grade 4: number analyzed (Participants) | 0 | 114 | 0
  Lymphocyte Count Decreased, Missing, Grade 4 |  | 0 |
  Lymphocyte Count Increased, Grade 0, Grade 1: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Increased, Grade 0, Grade 1 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 0, Grade 2: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Increased, Grade 0, Grade 2 | 0 | 4 | 0
  Lymphocyte Count Increased, Grade 0, Grade 3: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Increased, Grade 0, Grade 3 | 0 | 1 | 1
  Lymphocyte Count Increased, Grade 0, Grade 4: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Increased, Grade 0, Grade 4 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 1, Grade 0: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Increased, Grade 1, Grade 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 1, Grade 2: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Increased, Grade 1, Grade 2 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 1, Grade 3: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Increased, Grade 1, Grade 3 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 1, Grade 4: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Increased, Grade 1, Grade 4 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 2, Grade 0: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Increased, Grade 2, Grade 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 2, Grade 1: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Increased, Grade 2, Grade 1 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 2, Grade 3: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Increased, Grade 2, Grade 3 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 2, Grade 4: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Increased, Grade 2, Grade 4 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 3, Grade 0: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Increased, Grade 3, Grade 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 3, Grade 1: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Increased, Grade 3, Grade 1 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 3, Grade 2: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Increased, Grade 3, Grade 2 | 0 | 1 | 0
  Lymphocyte Count Increased, Grade 3, Grade 4: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Increased, Grade 3, Grade 4 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 4, Grade 0: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Increased, Grade 4, Grade 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 4, Grade 1: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Increased, Grade 4, Grade 1 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 4, Grade 2: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Increased, Grade 4, Grade 2 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 4, Grade 3: number analyzed (Participants) | 37 | 114 | 58
  Lymphocyte Count Increased, Grade 4, Grade 3 | 0 | 0 | 0
  Lymphocyte Count Increased, Missing, Grade 0: number analyzed (Participants) | 0 | 114 | 0
  Lymphocyte Count Increased, Missing, Grade 0 |  | 3 |
  Lymphocyte Count Increased, Missing, Grade 1: number analyzed (Participants) | 0 | 114 | 0
  Lymphocyte Count Increased, Missing, Grade 1 |  | 0 |
  Lymphocyte Count Increased, Missing, Grade 2: number analyzed (Participants) | 0 | 114 | 0
  Lymphocyte Count Increased, Missing, Grade 2 |  | 1 |
  Lymphocyte Count Increased, Missing, Grade 3: number analyzed (Participants) | 0 | 114 | 0
  Lymphocyte Count Increased, Missing, Grade 3 |  | 0 |
  Lymphocyte Count Increased, Missing, Grade 4: number analyzed (Participants) | 0 | 114 | 0
  Lymphocyte Count Increased, Missing, Grade 4 |  | 0 |
  Neutrophil Count Decreased, Grade 0, Grade 1: number analyzed (Participants) | 36 | 114 | 58
  Neutrophil Count Decreased, Grade 0, Grade 1 | 1 | 4 | 2
  Neutrophil Count Decreased, Grade 0, Grade 2: number analyzed (Participants) | 36 | 114 | 58
  Neutrophil Count Decreased, Grade 0, Grade 2 | 0 | 0 | 3
  Neutrophil Count Decreased, Grade 0, Grade 3: number analyzed (Participants) | 36 | 114 | 58
  Neutrophil Count Decreased, Grade 0, Grade 3 | 0 | 1 | 0
  Neutrophil Count Decreased, Grade 0, Grade 4: number analyzed (Participants) | 36 | 114 | 58
  Neutrophil Count Decreased, Grade 0, Grade 4 | 0 | 1 | 0
  Neutrophil Count Decreased, Grade 1, Grade 0: number analyzed (Participants) | 36 | 114 | 58
  Neutrophil Count Decreased, Grade 1, Grade 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 1, Grade 2: number analyzed (Participants) | 36 | 114 | 58
  Neutrophil Count Decreased, Grade 1, Grade 2 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 1, Grade 3: number analyzed (Participants) | 36 | 114 | 58
  Neutrophil Count Decreased, Grade 1, Grade 3 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 1, Grade 4: number analyzed (Participants) | 36 | 114 | 58
  Neutrophil Count Decreased, Grade 1, Grade 4 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 2, Grade 0: number analyzed (Participants) | 36 | 114 | 58
  Neutrophil Count Decreased, Grade 2, Grade 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 2, Grade 1: number analyzed (Participants) | 36 | 114 | 58
  Neutrophil Count Decreased, Grade 2, Grade 1 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 2, Grade 3: number analyzed (Participants) | 36 | 114 | 58
  Neutrophil Count Decreased, Grade 2, Grade 3 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 2, Grade 4: number analyzed (Participants) | 36 | 114 | 58
  Neutrophil Count Decreased, Grade 2, Grade 4 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 3, Grade 0: number analyzed (Participants) | 36 | 114 | 58
  Neutrophil Count Decreased, Grade 3, Grade 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 3, Grade 1: number analyzed (Participants) | 36 | 114 | 58
  Neutrophil Count Decreased, Grade 3, Grade 1 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 3, Grade 2: number analyzed (Participants) | 36 | 114 | 58
  Neutrophil Count Decreased, Grade 3, Grade 2 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 3, Grade 4: number analyzed (Participants) | 36 | 114 | 58
  Neutrophil Count Decreased, Grade 3, Grade 4 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 4, Grade 0: number analyzed (Participants) | 36 | 114 | 58
  Neutrophil Count Decreased, Grade 4, Grade 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 4, Grade 1: number analyzed (Participants) | 36 | 114 | 58
  Neutrophil Count Decreased, Grade 4, Grade 1 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 4, Grade 2: number analyzed (Participants) | 36 | 114 | 58
  Neutrophil Count Decreased, Grade 4, Grade 2 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 4, Grade 3: number analyzed (Participants) | 36 | 114 | 58
  Neutrophil Count Decreased, Grade 4, Grade 3 | 0 | 0 | 0
  Neutrophil Count Decreased, Missing, Grade 0: number analyzed (Participants) | 0 | 114 | 0
  Neutrophil Count Decreased, Missing, Grade 0 |  | 6 |
  Neutrophil Count Decreased, Missing, Grade 1: number analyzed (Participants) | 0 | 114 | 0
  Neutrophil Count Decreased, Missing, Grade 1 |  | 0 |
  Neutrophil Count Decreased, Missing, Grade 2: number analyzed (Participants) | 0 | 114 | 0
  Neutrophil Count Decreased, Missing, Grade 2 |  | 0 |
  Neutrophil Count Decreased, Missing, Grade 3: number analyzed (Participants) | 0 | 114 | 0
  Neutrophil Count Decreased, Missing, Grade 3 |  | 0 |
  Neutrophil Count Decreased, Missing, Grade 4: number analyzed (Participants) | 0 | 114 | 0
  Neutrophil Count Decreased, Missing, Grade 4 |  | 0 |
  Platelet Count Decreased, Grade 0, Grade 1: number analyzed (Participants) | 37 | 114 | 58
  Platelet Count Decreased, Grade 0, Grade 1 | 0 | 6 | 2
  Platelet Count Decreased, Grade 0, Grade 2: number analyzed (Participants) | 37 | 114 | 58
  Platelet Count Decreased, Grade 0, Grade 2 | 0 | 0 | 0
  Platelet Count Decreased, Grade 0, Grade 3: number analyzed (Participants) | 37 | 114 | 58
  Platelet Count Decreased, Grade 0, Grade 3 | 0 | 1 | 0
  Platelet Count Decreased, Grade 0, Grade 4: number analyzed (Participants) | 37 | 114 | 58
  Platelet Count Decreased, Grade 0, Grade 4 | 0 | 0 | 1
  Platelet Count Decreased, Grade 1, Grade 0: number analyzed (Participants) | 37 | 114 | 58
  Platelet Count Decreased, Grade 1, Grade 0 | 0 | 1 | 0
  Platelet Count Decreased, Grade 1, Grade 2: number analyzed (Participants) | 37 | 114 | 58
  Platelet Count Decreased, Grade 1, Grade 2 | 0 | 0 | 0
  Platelet Count Decreased, Grade 1, Grade 3: number analyzed (Participants) | 37 | 114 | 58
  Platelet Count Decreased, Grade 1, Grade 3 | 0 | 0 | 0
  Platelet Count Decreased, Grade 1, Grade 4: number analyzed (Participants) | 37 | 114 | 58
  Platelet Count Decreased, Grade 1, Grade 4 | 0 | 0 | 0
  Platelet Count Decreased, Grade 2, Grade 0: number analyzed (Participants) | 37 | 114 | 58
  Platelet Count Decreased, Grade 2, Grade 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 2, Grade 1: number analyzed (Participants) | 37 | 114 | 58
  Platelet Count Decreased, Grade 2, Grade 1 | 0 | 0 | 0
  Platelet Count Decreased, Grade 2, Grade 3: number analyzed (Participants) | 37 | 114 | 58
  Platelet Count Decreased, Grade 2, Grade 3 | 0 | 0 | 0
  Platelet Count Decreased, Grade 2, Grade 4: number analyzed (Participants) | 37 | 114 | 58
  Platelet Count Decreased, Grade 2, Grade 4 | 0 | 0 | 0
  Platelet Count Decreased, Grade 3, Grade 0: number analyzed (Participants) | 37 | 114 | 58
  Platelet Count Decreased, Grade 3, Grade 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 3, Grade 1: number analyzed (Participants) | 37 | 114 | 58
  Platelet Count Decreased, Grade 3, Grade 1 | 0 | 0 | 0
  Platelet Count Decreased, Grade 3, Grade 2: number analyzed (Participants) | 37 | 114 | 58
  Platelet Count Decreased, Grade 3, Grade 2 | 0 | 0 | 0
  Platelet Count Decreased, Grade 3, Grade 4: number analyzed (Participants) | 37 | 114 | 58
  Platelet Count Decreased, Grade 3, Grade 4 | 0 | 0 | 0
  Platelet Count Decreased, Grade 4, Grade 0: number analyzed (Participants) | 37 | 114 | 58
  Platelet Count Decreased, Grade 4, Grade 0 | 1 | 0 | 0
  Platelet Count Decreased, Grade 4, Grade 1: number analyzed (Participants) | 37 | 114 | 58
  Platelet Count Decreased, Grade 4, Grade 1 | 0 | 0 | 0
  Platelet Count Decreased, Grade 4, Grade 2: number analyzed (Participants) | 37 | 114 | 58
  Platelet Count Decreased, Grade 4, Grade 2 | 0 | 0 | 0
  Platelet Count Decreased, Grade 4, Grade 3: number analyzed (Participants) | 37 | 114 | 58
  Platelet Count Decreased, Grade 4, Grade 3 | 0 | 0 | 0
  Platelet Count Decreased, Missing, Grade 0: number analyzed (Participants) | 0 | 114 | 0
  Platelet Count Decreased, Missing, Grade 0 |  | 2 |
  Platelet Count Decreased, Missing, Grade 1: number analyzed (Participants) | 0 | 114 | 0
  Platelet Count Decreased, Missing, Grade 1 |  | 0 |
  Platelet Count Decreased, Missing, Grade 2: number analyzed (Participants) | 0 | 114 | 0
  Platelet Count Decreased, Missing, Grade 2 |  | 0 |
  Platelet Count Decreased, Missing, Grade 3: number analyzed (Participants) | 0 | 114 | 0
  Platelet Count Decreased, Missing, Grade 3 |  | 0 |
  Platelet Count Decreased, Missing, Grade 4: number analyzed (Participants) | 0 | 114 | 0
  Platelet Count Decreased, Missing, Grade 4 |  | 0 |
  White Blood Cell Decreased, Grade 0, Grade 1: number analyzed (Participants) | 37 | 114 | 58
  White Blood Cell Decreased, Grade 0, Grade 1 | 4 | 9 | 3
  White Blood Cell Decreased, Grade 0, Grade 2: number analyzed (Participants) | 37 | 114 | 58
  White Blood Cell Decreased, Grade 0, Grade 2 | 0 | 1 | 2
  White Blood Cell Decreased, Grade 0, Grade 3: number analyzed (Participants) | 37 | 114 | 58
  White Blood Cell Decreased, Grade 0, Grade 3 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 0, Grade 4: number analyzed (Participants) | 37 | 114 | 58
  White Blood Cell Decreased, Grade 0, Grade 4 | 0 | 2 | 0
  White Blood Cell Decreased, Grade 1, Grade 0: number analyzed (Participants) | 37 | 114 | 58
  White Blood Cell Decreased, Grade 1, Grade 0 | 0 | 1 | 0
  White Blood Cell Decreased, Grade 1, Grade 2: number analyzed (Participants) | 37 | 114 | 58
  White Blood Cell Decreased, Grade 1, Grade 2 | 1 | 2 | 2
  White Blood Cell Decreased, Grade 1, Grade 3: number analyzed (Participants) | 37 | 114 | 58
  White Blood Cell Decreased, Grade 1, Grade 3 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 1, Grade 4: number analyzed (Participants) | 37 | 114 | 58
  White Blood Cell Decreased, Grade 1, Grade 4 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 2, Grade 0: number analyzed (Participants) | 37 | 114 | 58
  White Blood Cell Decreased, Grade 2, Grade 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 2, Grade 1: number analyzed (Participants) | 37 | 114 | 58
  White Blood Cell Decreased, Grade 2, Grade 1 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 2, Grade 3: number analyzed (Participants) | 37 | 114 | 58
  White Blood Cell Decreased, Grade 2, Grade 3 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 2, Grade 4: number analyzed (Participants) | 37 | 114 | 58
  White Blood Cell Decreased, Grade 2, Grade 4 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 3, Grade 0: number analyzed (Participants) | 37 | 114 | 58
  White Blood Cell Decreased, Grade 3, Grade 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 3, Grade 1: number analyzed (Participants) | 37 | 114 | 58
  White Blood Cell Decreased, Grade 3, Grade 1 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 3, Grade 2: number analyzed (Participants) | 37 | 114 | 58
  White Blood Cell Decreased, Grade 3, Grade 2 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 3, Grade 4: number analyzed (Participants) | 37 | 114 | 58
  White Blood Cell Decreased, Grade 3, Grade 4 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 4, Grade 0: number analyzed (Participants) | 37 | 114 | 58
  White Blood Cell Decreased, Grade 4, Grade 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 4, Grade 1: number analyzed (Participants) | 37 | 114 | 58
  White Blood Cell Decreased, Grade 4, Grade 1 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 4, Grade 2: number analyzed (Participants) | 37 | 114 | 58
  White Blood Cell Decreased, Grade 4, Grade 2 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 4, Grade 3: number analyzed (Participants) | 37 | 114 | 58
  White Blood Cell Decreased, Grade 4, Grade 3 | 0 | 0 | 0
  Leukocytosis , Grade 0, Grade 1: number analyzed (Participants) | 37 | 114 | 58
  Leukocytosis , Grade 0, Grade 1 | 0 | 0 | 0
  Leukocytosis , Grade 0, Grade 2: number analyzed (Participants) | 37 | 114 | 58
  Leukocytosis , Grade 0, Grade 2 | 0 | 0 | 0
  Leukocytosis , Grade 0, Grade 3: number analyzed (Participants) | 37 | 114 | 58
  Leukocytosis , Grade 0, Grade 3 | 0 | 0 | 0
  Leukocytosis , Grade 0, Grade 4: number analyzed (Participants) | 37 | 114 | 58
  Leukocytosis , Grade 0, Grade 4 | 0 | 0 | 0
  Leukocytosis , Grade 1, Grade 0: number analyzed (Participants) | 37 | 114 | 58
  Leukocytosis , Grade 1, Grade 0 | 0 | 0 | 0
  Leukocytosis , Grade 1, Grade 2: number analyzed (Participants) | 37 | 114 | 58
  Leukocytosis , Grade 1, Grade 2 | 0 | 0 | 0
  Leukocytosis , Grade 1, Grade 3: number analyzed (Participants) | 37 | 114 | 58
  Leukocytosis , Grade 1, Grade 3 | 0 | 0 | 0
  Leukocytosis , Grade 1, Grade 4: number analyzed (Participants) | 37 | 114 | 58
  Leukocytosis , Grade 1, Grade 4 | 0 | 0 | 0
  Leukocytosis , Grade 2, Grade 0: number analyzed (Participants) | 37 | 114 | 58
  Leukocytosis , Grade 2, Grade 0 | 0 | 0 | 0
  Leukocytosis , Grade 2, Grade 1: number analyzed (Participants) | 37 | 114 | 58
  Leukocytosis , Grade 2, Grade 1 | 0 | 0 | 0
  Leukocytosis , Grade 2, Grade 3: number analyzed (Participants) | 37 | 114 | 58
  Leukocytosis , Grade 2, Grade 3 | 0 | 0 | 0
  Leukocytosis , Grade 2, Grade 4: number analyzed (Participants) | 37 | 114 | 58
  Leukocytosis , Grade 2, Grade 4 | 0 | 0 | 0
  Leukocytosis , Grade 3, Grade 0: number analyzed (Participants) | 37 | 114 | 58
  Leukocytosis , Grade 3, Grade 0 | 0 | 0 | 0
  Leukocytosis , Grade 3, Grade 1: number analyzed (Participants) | 37 | 114 | 58
  Leukocytosis , Grade 3, Grade 1 | 0 | 0 | 0
  Leukocytosis , Grade 3, Grade 2: number analyzed (Participants) | 37 | 114 | 58
  Leukocytosis , Grade 3, Grade 2 | 0 | 0 | 0
  Leukocytosis , Grade 3, Grade 4: number analyzed (Participants) | 37 | 114 | 58
  Leukocytosis , Grade 3, Grade 4 | 0 | 0 | 0
  Leukocytosis , Grade 4, Grade 0: number analyzed (Participants) | 37 | 114 | 58
  Leukocytosis , Grade 4, Grade 0 | 0 | 0 | 0
  Leukocytosis , Grade 4, Grade 1: number analyzed (Participants) | 37 | 114 | 58
  Leukocytosis , Grade 4, Grade 1 | 0 | 0 | 0
  Leukocytosis , Grade 4, Grade 2: number analyzed (Participants) | 37 | 114 | 58
  Leukocytosis , Grade 4, Grade 2 | 0 | 0 | 0
  Leukocytosis , Grade 4, Grade 3: number analyzed (Participants) | 37 | 114 | 58
  Leukocytosis , Grade 4, Grade 3 | 0 | 0 | 0

21. Secondary Outcome: Part 1B: Number of Participants With Worst Case Hematology Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Normal ranges were 0.01 to 0.3*10^9 cells/L (basophils), 0 to 500 cells /L (eosinophils), 41 to 50 percentage of RBC in blood (hematocrit), 2 to 8 percentage of WBC (monocytes), and Women: 4.2 to 5.4 million RBC/ mcL of blood and Men: 4.7 to 6.1 million RBC/ mcL (erythrocyte count). Participants were counted in worst case category that their value changes to low, normal or no change [NC] or high), unless there is NC in their category. Participants whose laboratory value category was unchanged (e.g. High to High) or whose value became normal, were recorded in "To Normal or No Change" category. Participants were counted twice if participant had values that changed To Low and To High, so percentages may not add to 100%.
Time Frame: Up to approximately 367 weeks
Population: All Treated Population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1B: Fela 0.300 mg/kg | Part 1B: Fela 1.000 mg/kg | Part 1B: Fela 24 mg
Number analyzed (Participants) | 39 | 115 | 59
Participants
  Basophils, To Low: number analyzed (Participants) | 36 | 107 | 58
  Basophils, To Low | 1 | 3 | 1
  Basophils, To Normal or No Change: number analyzed (Participants) | 36 | 107 | 58
  Basophils, To Normal or No Change | 35 | 101 | 55
  Basophils, To High: number analyzed (Participants) | 36 | 107 | 58
  Basophils, To High | 0 | 3 | 2
  Eosinophils, To Low: number analyzed (Participants) | 37 | 113 | 58
  Eosinophils, To Low | 5 | 11 | 7
  Eosinophils, To Normal or No Change: number analyzed (Participants) | 37 | 113 | 58
  Eosinophils, To Normal or No Change | 27 | 85 | 46
  Eosinophils, To High: number analyzed (Participants) | 37 | 113 | 58
  Eosinophils, To High | 7 | 18 | 6
  Hematocrit, To Low: number analyzed (Participants) | 37 | 114 | 58
  Hematocrit, To Low | 8 | 33 | 20
  Hematocrit, To Normal or No Change: number analyzed (Participants) | 37 | 114 | 58
  Hematocrit, To Normal or No Change | 28 | 74 | 38
  Hematocrit, To High: number analyzed (Participants) | 37 | 114 | 58
  Hematocrit, To High | 2 | 7 | 0
  Monocytes, To Low: number analyzed (Participants) | 37 | 114 | 58
  Monocytes, To Low | 0 | 3 | 0
  Monocytes, To Normal or No Change: number analyzed (Participants) | 37 | 114 | 58
  Monocytes, To Normal or No Change | 29 | 92 | 43
  Monocytes, To High: number analyzed (Participants) | 37 | 114 | 58
  Monocytes, To High | 8 | 20 | 15
  Erythrocytes, To Low: number analyzed (Participants) | 37 | 114 | 58
  Erythrocytes, To Low | 8 | 25 | 12
  Erythrocytes, To Normal or No Change: number analyzed (Participants) | 37 | 114 | 58
  Erythrocytes, To Normal or No Change | 29 | 85 | 45
  Erythrocytes, To High: number analyzed (Participants) | 37 | 114 | 58
  Erythrocytes, To High | 0 | 4 | 1

22. Secondary Outcome: Part 1B: Number of Participants With Worst Case Urinalysis Results Post-Baseline Relative to Baseline
Description: as for outcome 7
Time Frame: Up to approximately 367 weeks
Population: All treated population. Only those participants with data available at specified categories have been analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1B: Fela 0.300 mg/kg | Part 1B: Fela 1.000 mg/kg | Part 1B: Fela 24 mg
Number analyzed (Participants) | 38 | 113 | 58
Participants
  Glucose, No Change/Decreased | 36 | 104 | 56
  Glucose, Any Increase | 2 | 9 | 2
  Ketones, No Change/Decreased | 29 | 76 | 46
  Ketones, Any Increase | 9 | 37 | 12
  Occult Blood, No Change/Decreased: number analyzed (Participants) | 36 | 110 | 58
  Occult Blood, No Change/Decreased | 24 | 70 | 39
  Occult Blood, Any Increase: number analyzed (Participants) | 36 | 110 | 58
  Occult Blood, Any Increase | 12 | 40 | 19

23. Secondary Outcome: Part 1B: Number of Participants With Dose Modifications of Feladilimab
Description: Number of participants with dose modifications (including dose delays, dose escalation and infusion interruptions) were reported for Feladilimab.
Time Frame: Up to approximately 367 weeks
Population: All treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1B: Fela 0.300 mg/kg | Part 1B: Fela 1.000 mg/kg | Part 1B: Fela 24 mg
Number analyzed (Participants) | 39 | 115 | 59
Participants
  Dose delays | 4 | 17 | 5
  Dose escalations | 4 | 3 | 0
  Infusion interruptions | 0 | 1 | 0

24. Secondary Outcome: Part 2B: Number of Participants With Any Adverse Event(s) (AEs) and Serious Adverse Event(s) (SAEs)
Description: as for outcome 9
Time Frame: Up to approximately 367 weeks
Population: All Treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B: Fela 0.100 mg/kg + Pembro 200 mg | Part 2B: Fela 0.300 mg/kg + Pembro 200 mg | Part 2B: Fela 1.000 mg/kg + Pembro 200 mg | Part 2B: Fela 3.000 mg/kg + Pembro 200 mg | Part 2B: Fela 24 mg + Pembro 200 mg | Part 2B: Fela 48 mg + Pembro 400 mg | Part 2B: Fela 160 mg + Pembro 400 mg | Part 2B: Fela 80 mg + Pembro 200 mg
Number analyzed (Participants) | 14 | 255 | 44 | 23 | 4 | 6 | 5 | 1
Participants
  Any AEs | 13 | 250 | 43 | 23 | 4 | 5 | 4 | 1
  Any SAEs | 3 | 126 | 17 | 7 | 1 | 2 | 2 | 1

25. Secondary Outcome: Part 2B: Number of Participants With Worst-case Grade Change From Baseline in Clinical Chemistry Parameters
Description: as for outcome 3
Time Frame: Baseline (Day 1) and up to approximately 367 weeks
Population: All Treated Population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B: Fela 0.100 mg/kg + Pembro 200 mg | Part 2B: Fela 0.300 mg/kg + Pembro 200 mg | Part 2B: Fela 1.000 mg/kg + Pembro 200 mg | Part 2B: Fela 3.000 mg/kg + Pembro 200 mg | Part 2B: Fela 24 mg + Pembro 200 mg | Part 2B: Fela 48 mg + Pembro 400 mg | Part 2B: Fela 160 mg + Pembro 400 mg | Part 2B: Fela 80 mg + Pembro 200 mg
Number analyzed (Participants) | 14 | 255 | 44 | 23 | 4 | 6 | 5 | 1
Participants
  Hypoglycemia , Grade 0, Grade 1: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hypoglycemia , Grade 0, Grade 1 | 0 | 18 | 5 | 1 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 0, Grade 2: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hypoglycemia , Grade 0, Grade 2 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 0, Grade 3: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hypoglycemia , Grade 0, Grade 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 0, Grade 4: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hypoglycemia , Grade 0, Grade 4 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 1, Grade 0: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hypoglycemia , Grade 1, Grade 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Hypoglycemia , Grade 1, Grade 2: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hypoglycemia , Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 1, Grade 3: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hypoglycemia , Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 1, Grade 4: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hypoglycemia , Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 2, Grade 0: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hypoglycemia , Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 2, Grade 1: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hypoglycemia , Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 2, Grade 3: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hypoglycemia , Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 2, Grade 4: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hypoglycemia , Grade 2, Grade 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 3, Grade 0: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hypoglycemia , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 3, Grade 1: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hypoglycemia , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 3, Grade 2: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hypoglycemia , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 3, Grade 4: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hypoglycemia , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 4, Grade 0: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hypoglycemia , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 4, Grade 1: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hypoglycemia , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 4, Grade 2: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hypoglycemia , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Grade 4, Grade 3: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hypoglycemia , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Missing, Grade 0: number analyzed (Participants) | 0 | 252 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Missing, Grade 0 |  | 1 |  |  |  |  |  |
  Hypoglycemia , Missing, Grade 1: number analyzed (Participants) | 0 | 252 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Missing, Grade 1 |  | 0 |  |  |  |  |  |
  Hypoglycemia , Missing, Grade 2: number analyzed (Participants) | 0 | 252 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Missing, Grade 2 |  | 0 |  |  |  |  |  |
  Hypoglycemia , Missing, Grade 3: number analyzed (Participants) | 0 | 252 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Missing, Grade 3 |  | 0 |  |  |  |  |  |
  Hypoglycemia , Missing, Grade 4: number analyzed (Participants) | 0 | 252 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia , Missing, Grade 4 |  | 0 |  |  |  |  |  |
  Hyperglycemia , Grade 0, Grade 1: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hyperglycemia , Grade 0, Grade 1 | 4 | 91 | 12 | 6 | 1 | 2 | 2 | 0
  Hyperglycemia , Grade 0, Grade 2: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hyperglycemia , Grade 0, Grade 2 | 0 | 13 | 0 | 2 | 1 | 1 | 0 | 0
  Hyperglycemia , Grade 0, Grade 3: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hyperglycemia , Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 0, Grade 4: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hyperglycemia , Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 1, Grade 0: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hyperglycemia , Grade 1, Grade 0 | 0 | 5 | 2 | 0 | 0 | 0 | 1 | 0
  Hyperglycemia , Grade 1, Grade 2: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hyperglycemia , Grade 1, Grade 2 | 1 | 22 | 3 | 1 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 1, Grade 3: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hyperglycemia , Grade 1, Grade 3 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 1, Grade 4: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hyperglycemia , Grade 1, Grade 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 2, Grade 0: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hyperglycemia , Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 2, Grade 1: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hyperglycemia , Grade 2, Grade 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 2, Grade 3: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hyperglycemia , Grade 2, Grade 3 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Hyperglycemia , Grade 2, Grade 4: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hyperglycemia , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 3, Grade 0: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hyperglycemia , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 3, Grade 1: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hyperglycemia , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 3, Grade 2: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hyperglycemia , Grade 3, Grade 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 3, Grade 4: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hyperglycemia , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 4, Grade 0: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hyperglycemia , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 4, Grade 1: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hyperglycemia , Grade 4, Grade 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 4, Grade 2: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hyperglycemia , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Grade 4, Grade 3: number analyzed (Participants) | 14 | 252 | 42 | 22 | 4 | 6 | 5 | 1
  Hyperglycemia , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Missing, Grade 0: number analyzed (Participants) | 0 | 252 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Missing, Grade 0 |  | 1 |  |  |  |  |  |
  Hyperglycemia , Missing, Grade 1: number analyzed (Participants) | 0 | 252 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Missing, Grade 1 |  | 0 |  |  |  |  |  |
  Hyperglycemia , Missing, Grade 2: number analyzed (Participants) | 0 | 252 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Missing, Grade 2 |  | 0 |  |  |  |  |  |
  Hyperglycemia , Missing, Grade 3: number analyzed (Participants) | 0 | 252 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Missing, Grade 3 |  | 0 |  |  |  |  |  |
  Hyperglycemia , Missing, Grade 4: number analyzed (Participants) | 0 | 252 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia , Missing, Grade 4 |  | 0 |  |  |  |  |  |
  Hypoalbuminemia , Grade 0, Grade 1: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Hypoalbuminemia , Grade 0, Grade 1 | 6 | 47 | 7 | 6 | 1 | 2 | 0 | 0
  Hypoalbuminemia , Grade 0, Grade 2: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Hypoalbuminemia , Grade 0, Grade 2 | 1 | 12 | 2 | 1 | 0 | 2 | 2 | 0
  Hypoalbuminemia , Grade 0, Grade 3: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Hypoalbuminemia , Grade 0, Grade 3 | 0 | 5 | 1 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 0, Grade 4: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Hypoalbuminemia , Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 1, Grade 0: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Hypoalbuminemia , Grade 1, Grade 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 1, Grade 2: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Hypoalbuminemia , Grade 1, Grade 2 | 1 | 11 | 6 | 2 | 0 | 1 | 0 | 0
  Hypoalbuminemia , Grade 1, Grade 3: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Hypoalbuminemia , Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 1, Grade 4: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Hypoalbuminemia , Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 2, Grade 0: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Hypoalbuminemia , Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 2, Grade 1: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Hypoalbuminemia , Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 2, Grade 3: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Hypoalbuminemia , Grade 2, Grade 3 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 2, Grade 4: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Hypoalbuminemia , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 3, Grade 0: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Hypoalbuminemia , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 3, Grade 1: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Hypoalbuminemia , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 3, Grade 2: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Hypoalbuminemia , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 3, Grade 4: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Hypoalbuminemia , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 4, Grade 0: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Hypoalbuminemia , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 4, Grade 1: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Hypoalbuminemia , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 4, Grade 2: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Hypoalbuminemia , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Grade 4, Grade 3: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Hypoalbuminemia , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Missing, Grade 0: number analyzed (Participants) | 0 | 252 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Missing, Grade 0 |  | 0 |  |  |  |  |  |
  Hypoalbuminemia , Missing, Grade 1: number analyzed (Participants) | 0 | 252 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Missing, Grade 1 |  | 1 |  |  |  |  |  |
  Hypoalbuminemia , Missing, Grade 2: number analyzed (Participants) | 0 | 252 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Missing, Grade 2 |  | 0 |  |  |  |  |  |
  Hypoalbuminemia , Missing, Grade 3: number analyzed (Participants) | 0 | 252 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Missing, Grade 3 |  | 0 |  |  |  |  |  |
  Hypoalbuminemia , Missing, Grade 4: number analyzed (Participants) | 0 | 252 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia , Missing, Grade 4 |  | 0 |  |  |  |  |  |
  AP Increased, Grade 0, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AP Increased, Grade 0, Grade 1 | 3 | 50 | 11 | 2 | 0 | 1 | 2 | 0
  AP Increased, Grade 0, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AP Increased, Grade 0, Grade 2 | 0 | 7 | 1 | 0 | 0 | 1 | 0 | 0
  AP Increased, Grade 0, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AP Increased, Grade 0, Grade 3 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 0, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AP Increased, Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 1, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AP Increased, Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 1, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AP Increased, Grade 1, Grade 2 | 1 | 10 | 3 | 2 | 0 | 0 | 1 | 0
  AP Increased, Grade 1, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AP Increased, Grade 1, Grade 3 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
  AP Increased, Grade 1, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AP Increased, Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 2, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AP Increased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 2, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AP Increased, Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 2, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AP Increased, Grade 2, Grade 3 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0
  AP Increased, Grade 2, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AP Increased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 3, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AP Increased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 3, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AP Increased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 3, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AP Increased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 3, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AP Increased, Grade 3, Grade 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 4, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AP Increased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 4, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AP Increased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 4, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AP Increased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP Increased, Grade 4, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AP Increased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 0, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  ALT Increased, Grade 0, Grade 1 | 2 | 50 | 8 | 4 | 0 | 1 | 2 | 0
  ALT Increased, Grade 0, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  ALT Increased, Grade 0, Grade 2 | 1 | 6 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 0, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  ALT Increased, Grade 0, Grade 3 | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 0
  ALT Increased, Grade 0, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  ALT Increased, Grade 0, Grade 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 1, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  ALT Increased, Grade 1, Grade 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 1, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  ALT Increased, Grade 1, Grade 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  ALT Increased, Grade 1, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  ALT Increased, Grade 1, Grade 3 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
  ALT Increased, Grade 1, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  ALT Increased, Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 2, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  ALT Increased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 2, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  ALT Increased, Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 2, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  ALT Increased, Grade 2, Grade 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 2, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  ALT Increased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 3, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  ALT Increased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 3, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  ALT Increased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 3, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  ALT Increased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 3, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  ALT Increased, Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 4, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  ALT Increased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 4, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  ALT Increased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 4, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  ALT Increased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Increased, Grade 4, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  ALT Increased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 0, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AST Increased, Grade 0, Grade 1 | 4 | 65 | 8 | 4 | 0 | 0 | 2 | 0
  AST Increased, Grade 0, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AST Increased, Grade 0, Grade 2 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
  AST Increased, Grade 0, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AST Increased, Grade 0, Grade 3 | 0 | 4 | 2 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 0, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AST Increased, Grade 0, Grade 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 1, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AST Increased, Grade 1, Grade 0 | 0 | 5 | 3 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 1, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AST Increased, Grade 1, Grade 2 | 0 | 7 | 1 | 2 | 0 | 0 | 0 | 0
  AST Increased, Grade 1, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AST Increased, Grade 1, Grade 3 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  AST Increased, Grade 1, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AST Increased, Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 2, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AST Increased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 2, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AST Increased, Grade 2, Grade 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 2, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AST Increased, Grade 2, Grade 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 2, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AST Increased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 3, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AST Increased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 3, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AST Increased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 3, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AST Increased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 3, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AST Increased, Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 4, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AST Increased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 4, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AST Increased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 4, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AST Increased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Increased, Grade 4, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  AST Increased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 0, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Blood Bilirubin Increased, Grade 0, Grade 1 | 0 | 12 | 4 | 1 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 0, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Blood Bilirubin Increased, Grade 0, Grade 2 | 0 | 7 | 1 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 0, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Blood Bilirubin Increased, Grade 0, Grade 3 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 0, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Blood Bilirubin Increased, Grade 0, Grade 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 1, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Blood Bilirubin Increased, Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 1, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Blood Bilirubin Increased, Grade 1, Grade 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 1, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Blood Bilirubin Increased, Grade 1, Grade 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 1, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Blood Bilirubin Increased, Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 2, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Blood Bilirubin Increased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 2, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Blood Bilirubin Increased, Grade 2, Grade 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 2, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Blood Bilirubin Increased, Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 2, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Blood Bilirubin Increased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 3, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Blood Bilirubin Increased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 3, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Blood Bilirubin Increased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 3, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Blood Bilirubin Increased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 3, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Blood Bilirubin Increased, Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 4, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Blood Bilirubin Increased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 4, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Blood Bilirubin Increased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 4, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Blood Bilirubin Increased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Grade 4, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Blood Bilirubin Increased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Missing, Grade 0: number analyzed (Participants) | 0 | 253 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Missing, Grade 0 |  | 1 |  |  |  |  |  |
  Blood Bilirubin Increased, Missing, Grade 1: number analyzed (Participants) | 0 | 253 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Missing, Grade 1 |  | 0 |  |  |  |  |  |
  Blood Bilirubin Increased, Missing, Grade 2: number analyzed (Participants) | 0 | 253 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Missing, Grade 2 |  | 0 |  |  |  |  |  |
  Blood Bilirubin Increased, Missing, Grade 3: number analyzed (Participants) | 0 | 253 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Missing, Grade 3 |  | 0 |  |  |  |  |  |
  Blood Bilirubin Increased, Missing, Grade 4: number analyzed (Participants) | 0 | 253 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased, Missing, Grade 4 |  | 0 |  |  |  |  |  |
  Cpk Increased, Grade 0, Grade 1: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cpk Increased, Grade 0, Grade 1 |  |  | 0 |  |  |  |  |
  Cpk Increased, Grade 0, Grade 2: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cpk Increased, Grade 0, Grade 2 |  |  | 0 |  |  |  |  |
  Cpk Increased, Grade 0, Grade 3: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cpk Increased, Grade 0, Grade 3 |  |  | 0 |  |  |  |  |
  Cpk Increased, Grade 0, Grade 4: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cpk Increased, Grade 0, Grade 4 |  |  | 0 |  |  |  |  |
  Cpk Increased, Grade 1, Grade 0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cpk Increased, Grade 1, Grade 0 |  |  | 0 |  |  |  |  |
  Cpk Increased, Grade 1, Grade 2: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cpk Increased, Grade 1, Grade 2 |  |  | 0 |  |  |  |  |
  Cpk Increased, Grade 1, Grade 3: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cpk Increased, Grade 1, Grade 3 |  |  | 0 |  |  |  |  |
  Cpk Increased, Grade 1, Grade 4: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cpk Increased, Grade 1, Grade 4 |  |  | 0 |  |  |  |  |
  Cpk Increased, Grade 2, Grade 0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cpk Increased, Grade 2, Grade 0 |  |  | 0 |  |  |  |  |
  Cpk Increased, Grade 2, Grade 1: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cpk Increased, Grade 2, Grade 1 |  |  | 0 |  |  |  |  |
  Cpk Increased, Grade 2, Grade 3: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cpk Increased, Grade 2, Grade 3 |  |  | 0 |  |  |  |  |
  Cpk Increased, Grade 2, Grade 4: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cpk Increased, Grade 2, Grade 4 |  |  | 0 |  |  |  |  |
  Cpk Increased, Grade 3, Grade 0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cpk Increased, Grade 3, Grade 0 |  |  | 0 |  |  |  |  |
  Cpk Increased, Grade 3, Grade 1: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cpk Increased, Grade 3, Grade 1 |  |  | 0 |  |  |  |  |
  Cpk Increased, Grade 3, Grade 2: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cpk Increased, Grade 3, Grade 2 |  |  | 0 |  |  |  |  |
  Cpk Increased, Grade 3, Grade 4: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cpk Increased, Grade 3, Grade 4 |  |  | 0 |  |  |  |  |
  Cpk Increased, Grade 4, Grade 0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cpk Increased, Grade 4, Grade 0 |  |  | 0 |  |  |  |  |
  Cpk Increased, Grade 4, Grade 1: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cpk Increased, Grade 4, Grade 1 |  |  | 0 |  |  |  |  |
  Cpk Increased, Grade 4, Grade 2: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cpk Increased, Grade 4, Grade 2 |  |  | 0 |  |  |  |  |
  Cpk Increased, Grade 4, Grade 3: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cpk Increased, Grade 4, Grade 3 |  |  | 0 |  |  |  |  |
  Cpk Increased, Missing, Grade 0: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cpk Increased, Missing, Grade 0 |  |  | 1 |  |  |  |  |
  Cpk Increased, Missing, Grade 1: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cpk Increased, Missing, Grade 1 |  |  | 0 |  |  |  |  |
  Cpk Increased, Missing, Grade 2: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cpk Increased, Missing, Grade 2 |  |  | 0 |  |  |  |  |
  Cpk Increased, Missing, Grade 3: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cpk Increased, Missing, Grade 3 |  |  | 0 |  |  |  |  |
  Cpk Increased, Missing, Grade 4: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cpk Increased, Missing, Grade 4 |  |  | 0 |  |  |  |  |
  Creatinine Increased, Grade 0, Grade 1: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Creatinine Increased, Grade 0, Grade 1 | 2 | 24 | 4 | 6 | 0 | 1 | 0 | 1
  Creatinine Increased, Grade 0, Grade 2: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Creatinine Increased, Grade 0, Grade 2 | 0 | 9 | 1 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 0, Grade 3: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Creatinine Increased, Grade 0, Grade 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 0, Grade 4: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Creatinine Increased, Grade 0, Grade 4 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 1, Grade 0: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Creatinine Increased, Grade 1, Grade 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 1, Grade 2: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Creatinine Increased, Grade 1, Grade 2 | 0 | 12 | 0 | 0 | 0 | 0 | 1 | 0
  Creatinine Increased, Grade 1, Grade 3: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Creatinine Increased, Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 1, Grade 4: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Creatinine Increased, Grade 1, Grade 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 2, Grade 0: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Creatinine Increased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 2, Grade 1: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Creatinine Increased, Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 2, Grade 3: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Creatinine Increased, Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 2, Grade 4: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Creatinine Increased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 3, Grade 0: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Creatinine Increased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 3, Grade 1: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Creatinine Increased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 3, Grade 2: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Creatinine Increased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 3, Grade 4: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Creatinine Increased, Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 4, Grade 0: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Creatinine Increased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 4, Grade 1: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Creatinine Increased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 4, Grade 2: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Creatinine Increased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased, Grade 4, Grade 3: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Creatinine Increased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 0, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypokalemia , Grade 0, Grade 1 | 1 | 30 | 7 | 2 | 1 | 1 | 0 | 0
  Hypokalemia , Grade 0, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypokalemia , Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 0, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypokalemia , Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 0, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypokalemia , Grade 0, Grade 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 1, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypokalemia , Grade 1, Grade 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 1, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypokalemia , Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 1, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypokalemia , Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 1, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypokalemia , Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 2, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypokalemia , Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 2, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypokalemia , Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 2, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypokalemia , Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 2, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypokalemia , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 3, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypokalemia , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 3, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypokalemia , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 3, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypokalemia , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 3, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypokalemia , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 4, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypokalemia , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 4, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypokalemia , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 4, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypokalemia , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia , Grade 4, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypokalemia , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 0, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyperkalemia , Grade 0, Grade 1 | 1 | 45 | 6 | 4 | 0 | 2 | 0 | 1
  Hyperkalemia , Grade 0, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyperkalemia , Grade 0, Grade 2 | 0 | 8 | 3 | 1 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 0, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyperkalemia , Grade 0, Grade 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 0, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyperkalemia , Grade 0, Grade 4 | 0 | 4 | 1 | 3 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 1, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyperkalemia , Grade 1, Grade 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Hyperkalemia , Grade 1, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyperkalemia , Grade 1, Grade 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 1, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyperkalemia , Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 1, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyperkalemia , Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 2, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyperkalemia , Grade 2, Grade 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 2, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyperkalemia , Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 2, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyperkalemia , Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 2, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyperkalemia , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 3, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyperkalemia , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 3, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyperkalemia , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 3, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyperkalemia , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 3, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyperkalemia , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 4, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyperkalemia , Grade 4, Grade 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 4, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyperkalemia , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 4, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyperkalemia , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia , Grade 4, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyperkalemia , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 0, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyponatremia , Grade 0, Grade 1 | 4 | 52 | 5 | 8 | 0 | 3 | 1 | 0
  Hyponatremia , Grade 0, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyponatremia , Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 0, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyponatremia , Grade 0, Grade 3 | 0 | 10 | 3 | 2 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 0, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyponatremia , Grade 0, Grade 4 | 0 | 9 | 1 | 1 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 1, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyponatremia , Grade 1, Grade 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 1, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyponatremia , Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 1, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyponatremia , Grade 1, Grade 3 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0
  Hyponatremia , Grade 1, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyponatremia , Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 2, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyponatremia , Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 2, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyponatremia , Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 2, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyponatremia , Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 2, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyponatremia , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 3, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyponatremia , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 3, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyponatremia , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 3, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyponatremia , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 3, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyponatremia , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 4, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyponatremia , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 4, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyponatremia , Grade 4, Grade 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 4, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyponatremia , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia , Grade 4, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hyponatremia , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 0, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypernatremia , Grade 0, Grade 1 | 0 | 9 | 3 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 0, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypernatremia , Grade 0, Grade 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 0, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypernatremia , Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 0, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypernatremia , Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 1, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypernatremia , Grade 1, Grade 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 1, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypernatremia , Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 1, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypernatremia , Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 1, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypernatremia , Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 2, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypernatremia , Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 2, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypernatremia , Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 2, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypernatremia , Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 2, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypernatremia , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 3, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypernatremia , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 3, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypernatremia , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 3, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypernatremia , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 3, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypernatremia , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 4, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypernatremia , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 4, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypernatremia , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 4, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypernatremia , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia , Grade 4, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hypernatremia , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 0, Grade 1: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypocalcemia , Grade 0, Grade 1 | 1 | 26 | 2 | 2 | 0 | 1 | 0 | 0
  Hypocalcemia , Grade 0, Grade 2: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypocalcemia , Grade 0, Grade 2 | 0 | 5 | 0 | 0 | 1 | 0 | 0 | 0
  Hypocalcemia , Grade 0, Grade 3: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypocalcemia , Grade 0, Grade 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 0, Grade 4: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypocalcemia , Grade 0, Grade 4 | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 1, Grade 0: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypocalcemia , Grade 1, Grade 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 1
  Hypocalcemia , Grade 1, Grade 2: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypocalcemia , Grade 1, Grade 2 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 1, Grade 3: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypocalcemia , Grade 1, Grade 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 1, Grade 4: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypocalcemia , Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 2, Grade 0: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypocalcemia , Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 2, Grade 1: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypocalcemia , Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 2, Grade 3: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypocalcemia , Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 2, Grade 4: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypocalcemia , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 3, Grade 0: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypocalcemia , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 3, Grade 1: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypocalcemia , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 3, Grade 2: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypocalcemia , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 3, Grade 4: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypocalcemia , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 4, Grade 0: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypocalcemia , Grade 4, Grade 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 4, Grade 1: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypocalcemia , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 4, Grade 2: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypocalcemia , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Grade 4, Grade 3: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypocalcemia , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Missing, Grade 0: number analyzed (Participants) | 0 | 251 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Missing, Grade 0 |  | 0 |  |  |  |  |  |
  Hypocalcemia , Missing, Grade 1: number analyzed (Participants) | 0 | 251 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Missing, Grade 1 |  | 0 |  |  |  |  |  |
  Hypocalcemia , Missing, Grade 2: number analyzed (Participants) | 0 | 251 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Missing, Grade 2 |  | 0 |  |  |  |  |  |
  Hypocalcemia , Missing, Grade 3: number analyzed (Participants) | 0 | 251 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Missing, Grade 3 |  | 0 |  |  |  |  |  |
  Hypocalcemia , Missing, Grade 4: number analyzed (Participants) | 0 | 251 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia , Missing, Grade 4 |  | 1 |  |  |  |  |  |
  Hypercalcemia , Grade 0, Grade 1: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypercalcemia , Grade 0, Grade 1 | 2 | 34 | 7 | 9 | 0 | 0 | 2 | 0
  Hypercalcemia , Grade 0, Grade 2: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypercalcemia , Grade 0, Grade 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 0, Grade 3: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypercalcemia , Grade 0, Grade 3 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 0, Grade 4: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypercalcemia , Grade 0, Grade 4 | 0 | 10 | 1 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 1, Grade 0: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypercalcemia , Grade 1, Grade 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
  Hypercalcemia , Grade 1, Grade 2: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypercalcemia , Grade 1, Grade 2 | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 1, Grade 3: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypercalcemia , Grade 1, Grade 3 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 1, Grade 4: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypercalcemia , Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 2, Grade 0: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypercalcemia , Grade 2, Grade 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 2, Grade 1: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypercalcemia , Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 2, Grade 3: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypercalcemia , Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Hypercalcemia , Grade 2, Grade 4: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypercalcemia , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 3, Grade 0: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypercalcemia , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 3, Grade 1: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypercalcemia , Grade 3, Grade 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 3, Grade 2: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypercalcemia , Grade 3, Grade 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 3, Grade 4: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypercalcemia , Grade 3, Grade 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 4, Grade 0: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypercalcemia , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 4, Grade 1: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypercalcemia , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 4, Grade 2: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypercalcemia , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Grade 4, Grade 3: number analyzed (Participants) | 14 | 251 | 42 | 23 | 4 | 6 | 5 | 1
  Hypercalcemia , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Missing, Grade 0: number analyzed (Participants) | 0 | 251 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Missing, Grade 0 |  | 0 |  |  |  |  |  |
  Hypercalcemia , Missing, Grade 1: number analyzed (Participants) | 0 | 251 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Missing, Grade 1 |  | 0 |  |  |  |  |  |
  Hypercalcemia , Missing, Grade 2: number analyzed (Participants) | 0 | 251 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Missing, Grade 2 |  | 0 |  |  |  |  |  |
  Hypercalcemia , Missing, Grade 3: number analyzed (Participants) | 0 | 251 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Missing, Grade 3 |  | 0 |  |  |  |  |  |
  Hypercalcemia , Missing, Grade 4: number analyzed (Participants) | 0 | 251 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia , Missing, Grade 4 |  | 1 |  |  |  |  |  |
  Chronic Kidney Disease , Grade 0, Grade 1: number analyzed (Participants) | 5 | 98 | 10 | 13 | 1 | 1 | 3 | 0
  Chronic Kidney Disease , Grade 0, Grade 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 |
  Chronic Kidney Disease , Grade 0, Grade 2: number analyzed (Participants) | 5 | 98 | 10 | 13 | 1 | 1 | 3 | 0
  Chronic Kidney Disease , Grade 0, Grade 2 | 0 | 5 | 0 | 1 | 0 | 0 | 0 |
  Chronic Kidney Disease , Grade 0, Grade 3: number analyzed (Participants) | 5 | 98 | 10 | 13 | 1 | 1 | 3 | 0
  Chronic Kidney Disease , Grade 0, Grade 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 |
  Chronic Kidney Disease , Grade 0, Grade 4: number analyzed (Participants) | 5 | 98 | 10 | 13 | 1 | 1 | 3 | 0
  Chronic Kidney Disease , Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Chronic Kidney Disease , Grade 1, Grade 0: number analyzed (Participants) | 5 | 98 | 10 | 13 | 1 | 1 | 3 | 0
  Chronic Kidney Disease , Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Chronic Kidney Disease , Grade 1, Grade 2: number analyzed (Participants) | 5 | 98 | 10 | 13 | 1 | 1 | 3 | 0
  Chronic Kidney Disease , Grade 1, Grade 2 | 0 | 11 | 0 | 0 | 0 | 0 | 0 |
  Chronic Kidney Disease , Grade 1, Grade 3: number analyzed (Participants) | 5 | 98 | 10 | 13 | 1 | 1 | 3 | 0
  Chronic Kidney Disease , Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Chronic Kidney Disease , Grade 1, Grade 4: number analyzed (Participants) | 5 | 98 | 10 | 13 | 1 | 1 | 3 | 0
  Chronic Kidney Disease , Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Chronic Kidney Disease , Grade 2, Grade 0: number analyzed (Participants) | 5 | 98 | 10 | 13 | 1 | 1 | 3 | 0
  Chronic Kidney Disease , Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Chronic Kidney Disease , Grade 2, Grade 1: number analyzed (Participants) | 5 | 98 | 10 | 13 | 1 | 1 | 3 | 0
  Chronic Kidney Disease , Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Chronic Kidney Disease , Grade 2, Grade 3: number analyzed (Participants) | 5 | 98 | 10 | 13 | 1 | 1 | 3 | 0
  Chronic Kidney Disease , Grade 2, Grade 3 | 0 | 4 | 0 | 0 | 0 | 0 | 0 |
  Chronic Kidney Disease , Grade 2, Grade 4: number analyzed (Participants) | 5 | 98 | 10 | 13 | 1 | 1 | 3 | 0
  Chronic Kidney Disease , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Chronic Kidney Disease , Grade 3, Grade 0: number analyzed (Participants) | 5 | 98 | 10 | 13 | 1 | 1 | 3 | 0
  Chronic Kidney Disease , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Chronic Kidney Disease , Grade 3, Grade 1: number analyzed (Participants) | 5 | 98 | 10 | 13 | 1 | 1 | 3 | 0
  Chronic Kidney Disease , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Chronic Kidney Disease , Grade 3, Grade 2: number analyzed (Participants) | 5 | 98 | 10 | 13 | 1 | 1 | 3 | 0
  Chronic Kidney Disease , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Chronic Kidney Disease , Grade 3, Grade 4: number analyzed (Participants) | 5 | 98 | 10 | 13 | 1 | 1 | 3 | 0
  Chronic Kidney Disease , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Chronic Kidney Disease , Grade 4, Grade 0: number analyzed (Participants) | 5 | 98 | 10 | 13 | 1 | 1 | 3 | 0
  Chronic Kidney Disease , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Chronic Kidney Disease , Grade 4, Grade 1: number analyzed (Participants) | 5 | 98 | 10 | 13 | 1 | 1 | 3 | 0
  Chronic Kidney Disease , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Chronic Kidney Disease , Grade 4, Grade 2: number analyzed (Participants) | 5 | 98 | 10 | 13 | 1 | 1 | 3 | 0
  Chronic Kidney Disease , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Chronic Kidney Disease , Grade 4, Grade 3: number analyzed (Participants) | 5 | 98 | 10 | 13 | 1 | 1 | 3 | 0
  Chronic Kidney Disease , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Chronic Kidney Disease , Missing, Grade 0: number analyzed (Participants) | 5 | 98 | 10 | 13 | 0 | 0 | 3 | 0
  Chronic Kidney Disease , Missing, Grade 0 | 0 | 6 | 1 | 1 |  |  | 1 |
  Chronic Kidney Disease , Missing, Grade 1: number analyzed (Participants) | 5 | 98 | 10 | 13 | 0 | 0 | 3 | 0
  Chronic Kidney Disease , Missing, Grade 1 | 2 | 9 | 0 | 1 |  |  | 0 |
  Chronic Kidney Disease , Missing, Grade 2: number analyzed (Participants) | 5 | 98 | 10 | 13 | 0 | 0 | 3 | 0
  Chronic Kidney Disease , Missing, Grade 2 | 1 | 10 | 3 | 4 |  |  | 0 |
  Chronic Kidney Disease , Missing, Grade 3: number analyzed (Participants) | 5 | 98 | 10 | 13 | 0 | 0 | 3 | 0
  Chronic Kidney Disease , Missing, Grade 3 | 0 | 0 | 0 | 0 |  |  | 0 |
  Chronic Kidney Disease , Missing, Grade 4: number analyzed (Participants) | 5 | 98 | 10 | 13 | 0 | 0 | 3 | 0
  Chronic Kidney Disease , Missing, Grade 4 | 0 | 6 | 0 | 1 |  |  | 0 |

26. Secondary Outcome: Part 2B: Number of Participants With Worst Case Chemistry Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Normal ranges were 0.1 to 0.3 micromoles (umol)/liter (L) (direct bilirubin); 6 to 8.3 grams/L (protein); 100 to 250 international units (IU)/L (Lactate Dehydrogenase(LDH)); 2.3 - 4.1 picomoles/L (Free Triiodothyronine(T3)); 4.6 to 11.2 picomoles/L (Free Thyroxine(T4)); 0 and 0.04 microgram (ug)/L (Troponin I); 0 - 0.01 ug/L (Troponin T); 0.45 to 4.5 milliunits (Mu)/L (Thyrotropin(TSH)); 24-204 ug/L (creatine kinase); and 6 to 24 millimoles/L (Urea). Participants were counted in worst case category that their value changes to low, normal or no change [NC] or high), unless there is NC in their category. Participants whose laboratory value category was unchanged (e.g. High to High) or whose value became normal, were recorded in "To Normal or No Change" category. Participants were counted twice if participant had values that changed To Low and To High, so percentages may not add to 100%.
Time Frame: Up to approximately 367 weeks
Population: All Treated Population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B: Fela 0.100 mg/kg + Pembro 200 mg | Part 2B: Fela 0.300 mg/kg + Pembro 200 mg | Part 2B: Fela 1.000 mg/kg + Pembro 200 mg | Part 2B: Fela 3.000 mg/kg + Pembro 200 mg | Part 2B: Fela 24 mg + Pembro 200 mg | Part 2B: Fela 48 mg + Pembro 400 mg | Part 2B: Fela 160 mg + Pembro 400 mg | Part 2B: Fela 80 mg + Pembro 200 mg
Number analyzed (Participants) | 14 | 255 | 44 | 23 | 4 | 6 | 5 | 1
Participants
  Direct Bilirubin (umol/L), To Low: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin (umol/L), To Low |  |  | 0 |  |  |  |  |
  Direct Bilirubin (umol/L), To Normal or No Change: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin (umol/L), To Normal or No Change |  |  | 0 |  |  |  |  |
  Direct Bilirubin (umol/L), To High: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin (umol/L), To High |  |  | 1 |  |  |  |  |
  Creatine Kinase MB (ug/L), To Low: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Creatine Kinase MB (ug/L), To Low |  |  | 0 |  |  |  |  |
  Creatine Kinase MB (ug/L), To Normal or No Change: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Creatine Kinase MB (ug/L), To Normal or No Change |  |  | 1 |  |  |  |  |
  Creatine Kinase MB (ug/L), To High: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Creatine Kinase MB (ug/L), To High |  |  | 0 |  |  |  |  |
  Lactate Dehydrogenase (IU/L), To Low: number analyzed (Participants) | 0 | 2 | 4 | 1 | 0 | 0 | 0 | 0
  Lactate Dehydrogenase (IU/L), To Low |  | 0 | 0 | 1 |  |  |  |
  Lactate Dehydrogenase (IU/L), To Normal or No Change: number analyzed (Participants) | 0 | 2 | 4 | 1 | 0 | 0 | 0 | 0
  Lactate Dehydrogenase (IU/L), To Normal or No Change |  | 0 | 2 | 0 |  |  |  |
  Lactate Dehydrogenase (IU/L), To High: number analyzed (Participants) | 0 | 2 | 4 | 1 | 0 | 0 | 0 | 0
  Lactate Dehydrogenase (IU/L), To High |  | 2 | 2 | 0 |  |  |  |
  Protein (g/L), To Low: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Protein (g/L), To Low | 1 | 37 | 9 | 2 | 3 | 1 | 1 | 0
  Protein (g/L), To Normal or No Change: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Protein (g/L), To Normal or No Change | 11 | 183 | 27 | 18 | 1 | 4 | 2 | 1
  Protein (g/L), To High: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Protein (g/L), To High | 2 | 38 | 7 | 4 | 0 | 1 | 2 | 0
  Triiodothyronine, Free (pmol/L), To Low: number analyzed (Participants) | 13 | 226 | 38 | 20 | 4 | 5 | 4 | 0
  Triiodothyronine, Free (pmol/L), To Low | 3 | 41 | 7 | 5 | 0 | 0 | 2 |
  Triiodothyronine, Free (pmol/L), To Normal or No Change: number analyzed (Participants) | 13 | 226 | 38 | 20 | 4 | 5 | 4 | 0
  Triiodothyronine, Free (pmol/L), To Normal or No Change | 10 | 160 | 29 | 12 | 3 | 5 | 2 |
  Triiodothyronine, Free (pmol/L), To High: number analyzed (Participants) | 13 | 226 | 38 | 20 | 4 | 5 | 4 | 0
  Triiodothyronine, Free (pmol/L), To High | 0 | 31 | 2 | 3 | 1 | 0 | 0 |
  Thyroxine, Free (pmol/L), To Low: number analyzed (Participants) | 13 | 229 | 38 | 20 | 4 | 3 | 4 | 0
  Thyroxine, Free (pmol/L), To Low | 2 | 30 | 6 | 3 | 1 | 0 | 0 |
  Thyroxine, Free (pmol/L), To Normal or No Change: number analyzed (Participants) | 13 | 229 | 38 | 20 | 4 | 3 | 4 | 0
  Thyroxine, Free (pmol/L), To Normal or No Change | 10 | 180 | 30 | 16 | 2 | 3 | 4 |
  Thyroxine, Free (pmol/L), To High: number analyzed (Participants) | 13 | 229 | 38 | 20 | 4 | 3 | 4 | 0
  Thyroxine, Free (pmol/L), To High | 1 | 25 | 2 | 1 | 1 | 0 | 0 |
  Troponin I (ug/L), To Low: number analyzed (Participants) | 8 | 125 | 21 | 16 | 3 | 2 | 3 | 0
  Troponin I (ug/L), To Low | 0 | 1 | 0 | 2 | 0 | 0 | 0 |
  Troponin I (ug/L), To Normal or No Change: number analyzed (Participants) | 8 | 125 | 21 | 16 | 3 | 2 | 3 | 0
  Troponin I (ug/L), To Normal or No Change | 7 | 109 | 18 | 12 | 3 | 2 | 3 |
  Troponin I (ug/L), To High: number analyzed (Participants) | 8 | 125 | 21 | 16 | 3 | 2 | 3 | 0
  Troponin I (ug/L), To High | 1 | 15 | 3 | 2 | 0 | 0 | 0 |
  Troponin T (ug/L), To Low: number analyzed (Participants) | 0 | 57 | 7 | 5 | 1 | 1 | 0 | 0
  Troponin T (ug/L), To Low |  | 0 | 0 | 0 | 0 | 0 |  |
  Troponin T (ug/L), To Normal or No Change: number analyzed (Participants) | 0 | 57 | 7 | 5 | 1 | 1 | 0 | 0
  Troponin T (ug/L), To Normal or No Change |  | 44 | 6 | 4 | 1 | 1 |  |
  Troponin T (ug/L), To High: number analyzed (Participants) | 0 | 57 | 7 | 5 | 1 | 1 | 0 | 0
  Troponin T (ug/L), To High |  | 13 | 1 | 1 | 0 | 0 |  |
  Thyrotropin (mU/L), To Low: number analyzed (Participants) | 13 | 229 | 38 | 20 | 3 | 5 | 4 | 0
  Thyrotropin (mU/L), To Low | 0 | 22 | 1 | 2 | 0 | 1 | 1 |
  Thyrotropin (mU/L), To Normal or No Change: number analyzed (Participants) | 13 | 229 | 38 | 20 | 3 | 5 | 4 | 0
  Thyrotropin (mU/L), To Normal or No Change | 12 | 179 | 29 | 12 | 3 | 4 | 3 |
  Thyrotropin (mU/L), To High: number analyzed (Participants) | 13 | 229 | 38 | 20 | 3 | 5 | 4 | 0
  Thyrotropin (mU/L), To High | 1 | 34 | 8 | 6 | 0 | 1 | 0 |
  Urea (mmol/L), To Low: number analyzed (Participants) | 12 | 223 | 36 | 19 | 0 | 3 | 5 | 0
  Urea (mmol/L), To Low | 2 | 33 | 3 | 5 |  | 0 | 1 |
  Urea (mmol/L), To Normal or No Change: number analyzed (Participants) | 12 | 223 | 36 | 19 | 0 | 3 | 5 | 0
  Urea (mmol/L), To Normal or No Change | 9 | 137 | 27 | 10 |  | 1 | 3 |
  Urea (mmol/L), To High: number analyzed (Participants) | 12 | 223 | 36 | 19 | 0 | 3 | 5 | 0
  Urea (mmol/L), To High | 1 | 53 | 6 | 4 |  | 2 | 1 |

27. Secondary Outcome: Part 2B: Number of Participants With Worst-case Grade Change From Baseline in Hematology Parameters
Description: as for outcome 5
Time Frame: Baseline (Day 1) and up to approximately 367 weeks
Population: All Treated Population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B: Fela 0.100 mg/kg + Pembro 200 mg | Part 2B: Fela 0.300 mg/kg + Pembro 200 mg | Part 2B: Fela 1.000 mg/kg + Pembro 200 mg | Part 2B: Fela 3.000 mg/kg + Pembro 200 mg | Part 2B: Fela 24 mg + Pembro 200 mg | Part 2B: Fela 48 mg + Pembro 400 mg | Part 2B: Fela 160 mg + Pembro 400 mg | Part 2B: Fela 80 mg + Pembro 200 mg
Number analyzed (Participants) | 14 | 255 | 44 | 23 | 4 | 6 | 5 | 1
Participants
  Anemia , Grade 0, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Anemia , Grade 0, Grade 1 | 4 | 71 | 13 | 5 | 1 | 2 | 0 | 0
  Anemia , Grade 0, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Anemia , Grade 0, Grade 2 | 1 | 9 | 4 | 2 | 0 | 0 | 0 | 0
  Anemia , Grade 0, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Anemia , Grade 0, Grade 3 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 0, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Anemia , Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 1, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Anemia , Grade 1, Grade 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 1, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Anemia , Grade 1, Grade 2 | 3 | 44 | 7 | 4 | 0 | 0 | 2 | 0
  Anemia , Grade 1, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Anemia , Grade 1, Grade 3 | 0 | 10 | 0 | 1 | 0 | 1 | 0 | 0
  Anemia , Grade 1, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Anemia , Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 2, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Anemia , Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 2, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Anemia , Grade 2, Grade 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Anemia , Grade 2, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Anemia , Grade 2, Grade 3 | 0 | 5 | 1 | 1 | 0 | 0 | 0 | 0
  Anemia , Grade 2, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Anemia , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 3, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Anemia , Grade 3, Grade 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 3, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Anemia , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 3, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Anemia , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 3, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Anemia , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 4, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Anemia , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 4, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Anemia , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 4, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Anemia , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia , Grade 4, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Anemia , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 0, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hemoglobin Increased, Grade 0, Grade 1 | 0 | 5 | 2 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 0, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hemoglobin Increased, Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 0, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hemoglobin Increased, Grade 0, Grade 3 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 0, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hemoglobin Increased, Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 1, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hemoglobin Increased, Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 1, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hemoglobin Increased, Grade 1, Grade 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 1, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hemoglobin Increased, Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 1, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hemoglobin Increased, Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 2, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hemoglobin Increased, Grade 2, Grade 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 2, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hemoglobin Increased, Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 2, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hemoglobin Increased, Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 2, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hemoglobin Increased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 3, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hemoglobin Increased, Grade 3, Grade 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 3, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hemoglobin Increased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 3, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hemoglobin Increased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 3, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hemoglobin Increased, Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 4, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hemoglobin Increased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 4, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hemoglobin Increased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 4, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hemoglobin Increased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin Increased, Grade 4, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Hemoglobin Increased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 0, Grade 1: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Decreased, Grade 0, Grade 1 | 3 | 40 | 7 | 1 | 2 | 1 | 1 | 0
  Lymphocyte Count Decreased, Grade 0, Grade 2: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Decreased, Grade 0, Grade 2 | 1 | 24 | 3 | 4 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 0, Grade 3: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Decreased, Grade 0, Grade 3 | 1 | 6 | 1 | 1 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 0, Grade 4: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Decreased, Grade 0, Grade 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 1, Grade 0: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Decreased, Grade 1, Grade 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 1, Grade 2: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Decreased, Grade 1, Grade 2 | 3 | 42 | 9 | 5 | 1 | 2 | 0 | 0
  Lymphocyte Count Decreased, Grade 1, Grade 3: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Decreased, Grade 1, Grade 3 | 0 | 16 | 1 | 2 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 1, Grade 4: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Decreased, Grade 1, Grade 4 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 2, Grade 0: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Decreased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 2, Grade 1: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Decreased, Grade 2, Grade 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Lymphocyte Count Decreased, Grade 2, Grade 3: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Decreased, Grade 2, Grade 3 | 0 | 7 | 1 | 3 | 0 | 1 | 2 | 0
  Lymphocyte Count Decreased, Grade 2, Grade 4: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Decreased, Grade 2, Grade 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 3, Grade 0: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Decreased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 3, Grade 1: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Decreased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 3, Grade 2: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Decreased, Grade 3, Grade 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 3, Grade 4: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Decreased, Grade 3, Grade 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 4, Grade 0: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Decreased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 4, Grade 1: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Decreased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 4, Grade 2: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Decreased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Grade 4, Grade 3: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Decreased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased, Missing, Grade 0: number analyzed (Participants) | 0 | 252 | 0 | 0 | 0 | 6 | 0 | 0
  Lymphocyte Count Decreased, Missing, Grade 0 |  | 1 |  |  |  | 0 |  |
  Lymphocyte Count Decreased, Missing, Grade 1: number analyzed (Participants) | 0 | 252 | 0 | 0 | 0 | 6 | 0 | 0
  Lymphocyte Count Decreased, Missing, Grade 1 |  | 0 |  |  |  | 0 |  |
  Lymphocyte Count Decreased, Missing, Grade 2: number analyzed (Participants) | 0 | 252 | 0 | 0 | 0 | 6 | 0 | 0
  Lymphocyte Count Decreased, Missing, Grade 2 |  | 1 |  |  |  | 1 |  |
  Lymphocyte Count Decreased, Missing, Grade 3: number analyzed (Participants) | 0 | 252 | 0 | 0 | 0 | 6 | 0 | 0
  Lymphocyte Count Decreased, Missing, Grade 3 |  | 0 |  |  |  | 0 |  |
  Lymphocyte Count Decreased, Missing, Grade 4: number analyzed (Participants) | 0 | 252 | 0 | 0 | 0 | 6 | 0 | 0
  Lymphocyte Count Decreased, Missing, Grade 4 |  | 0 |  |  |  | 0 |  |
  Lymphocyte Count Increased, Grade 0, Grade 1: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Increased, Grade 0, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 0, Grade 2: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Increased, Grade 0, Grade 2 | 1 | 9 | 3 | 1 | 0 | 0 | 1 | 0
  Lymphocyte Count Increased, Grade 0, Grade 3: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Increased, Grade 0, Grade 3 | 0 | 4 | 1 | 1 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 0, Grade 4: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Increased, Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 1, Grade 0: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Increased, Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 1, Grade 2: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Increased, Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 1, Grade 3: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Increased, Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 1, Grade 4: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Increased, Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 2, Grade 0: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Increased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 2, Grade 1: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Increased, Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 2, Grade 2: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Increased, Grade 2, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 2, Grade 3: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Increased, Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 2, Grade 4: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Increased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 3, Grade 0: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Increased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 3, Grade 1: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Increased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 3, Grade 2: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Increased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 3, Grade 4: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Increased, Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 4, Grade 0: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Increased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 4, Grade 1: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Increased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 4, Grade 2: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Increased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Grade 4, Grade 3: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Lymphocyte Count Increased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased, Missing, Grade 0: number analyzed (Participants) | 0 | 252 | 0 | 0 | 0 | 6 | 0 | 0
  Lymphocyte Count Increased, Missing, Grade 0 |  | 2 |  |  |  | 1 |  |
  Lymphocyte Count Increased, Missing, Grade 1: number analyzed (Participants) | 0 | 252 | 0 | 0 | 0 | 6 | 0 | 0
  Lymphocyte Count Increased, Missing, Grade 1 |  | 0 |  |  |  | 0 |  |
  Lymphocyte Count Increased, Missing, Grade 2: number analyzed (Participants) | 0 | 252 | 0 | 0 | 0 | 6 | 0 | 0
  Lymphocyte Count Increased, Missing, Grade 2 |  | 0 |  |  |  | 0 |  |
  Lymphocyte Count Increased, Missing, Grade 3: number analyzed (Participants) | 0 | 252 | 0 | 0 | 0 | 6 | 0 | 0
  Lymphocyte Count Increased, Missing, Grade 3 |  | 0 |  |  |  | 0 |  |
  Lymphocyte Count Increased, Missing, Grade 4: number analyzed (Participants) | 0 | 252 | 0 | 0 | 0 | 6 | 0 | 0
  Lymphocyte Count Increased, Missing, Grade 4 |  | 0 |  |  |  | 0 |  |
  Neutrophil Count Decreased, Grade 0, Grade 1: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Neutrophil Count Decreased, Grade 0, Grade 1 | 1 | 3 | 3 | 0 | 1 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 0, Grade 2: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Neutrophil Count Decreased, Grade 0, Grade 2 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 0, Grade 3: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Neutrophil Count Decreased, Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 0, Grade 4: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Neutrophil Count Decreased, Grade 0, Grade 4 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 1, Grade 0: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Neutrophil Count Decreased, Grade 1, Grade 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 1, Grade 2: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Neutrophil Count Decreased, Grade 1, Grade 2 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 1, Grade 3: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Neutrophil Count Decreased, Grade 1, Grade 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 1, Grade 4: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Neutrophil Count Decreased, Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 2, Grade 0: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Neutrophil Count Decreased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 2, Grade 1: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Neutrophil Count Decreased, Grade 2, Grade 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 2, Grade 3: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Neutrophil Count Decreased, Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 2, Grade 4: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Neutrophil Count Decreased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 3, Grade 0: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Neutrophil Count Decreased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 3, Grade 1: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Neutrophil Count Decreased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 3, Grade 2: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Neutrophil Count Decreased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 3, Grade 4: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Neutrophil Count Decreased, Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 4, Grade 0: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Neutrophil Count Decreased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 4, Grade 1: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Neutrophil Count Decreased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 4, Grade 2: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Neutrophil Count Decreased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Grade 4, Grade 3: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Neutrophil Count Decreased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased, Missing, Grade 0: number analyzed (Participants) | 0 | 252 | 0 | 0 | 0 | 6 | 0 | 0
  Neutrophil Count Decreased, Missing, Grade 0 |  | 2 |  |  |  | 1 |  |
  Neutrophil Count Decreased, Missing, Grade 1: number analyzed (Participants) | 0 | 252 | 0 | 0 | 0 | 6 | 0 | 0
  Neutrophil Count Decreased, Missing, Grade 1 |  | 0 |  |  |  | 0 |  |
  Neutrophil Count Decreased, Missing, Grade 2: number analyzed (Participants) | 0 | 252 | 0 | 0 | 0 | 6 | 0 | 0
  Neutrophil Count Decreased, Missing, Grade 2 |  | 0 |  |  |  | 0 |  |
  Neutrophil Count Decreased, Missing, Grade 3: number analyzed (Participants) | 0 | 252 | 0 | 0 | 0 | 6 | 0 | 0
  Neutrophil Count Decreased, Missing, Grade 3 |  | 0 |  |  |  | 0 |  |
  Neutrophil Count Decreased, Missing, Grade 4: number analyzed (Participants) | 0 | 252 | 0 | 0 | 0 | 6 | 0 | 0
  Neutrophil Count Decreased, Missing, Grade 4 |  | 0 |  |  |  | 0 |  |
  Platelet Count Decreased, Grade 0, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Platelet Count Decreased, Grade 0, Grade 1 | 0 | 21 | 3 | 0 | 0 | 1 | 0 | 0
  Platelet Count Decreased, Grade 0, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Platelet Count Decreased, Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 0, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Platelet Count Decreased, Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 0, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Platelet Count Decreased, Grade 0, Grade 4 | 0 | 8 | 2 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 1, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Platelet Count Decreased, Grade 1, Grade 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 1, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Platelet Count Decreased, Grade 1, Grade 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 1, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Platelet Count Decreased, Grade 1, Grade 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 1, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Platelet Count Decreased, Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 2, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Platelet Count Decreased, Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 2, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Platelet Count Decreased, Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 2, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Platelet Count Decreased, Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 2, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Platelet Count Decreased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 3, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Platelet Count Decreased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 3, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Platelet Count Decreased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 3, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Platelet Count Decreased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 3, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Platelet Count Decreased, Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 4, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Platelet Count Decreased, Grade 4, Grade 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 4, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Platelet Count Decreased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 4, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Platelet Count Decreased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased, Grade 4, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Platelet Count Decreased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 0, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  White Blood Cell Decreased, Grade 0, Grade 1 | 1 | 19 | 4 | 1 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 0, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  White Blood Cell Decreased, Grade 0, Grade 2 | 0 | 4 | 0 | 1 | 1 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 0, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  White Blood Cell Decreased, Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 0, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  White Blood Cell Decreased, Grade 0, Grade 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 1, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  White Blood Cell Decreased, Grade 1, Grade 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 1, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  White Blood Cell Decreased, Grade 1, Grade 2 | 0 | 5 | 1 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 1, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  White Blood Cell Decreased, Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 1, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  White Blood Cell Decreased, Grade 1, Grade 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 2, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  White Blood Cell Decreased, Grade 2, Grade 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 2, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  White Blood Cell Decreased, Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 2, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  White Blood Cell Decreased, Grade 2, Grade 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 2, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  White Blood Cell Decreased, Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 3, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  White Blood Cell Decreased, Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 3, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  White Blood Cell Decreased, Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 3, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  White Blood Cell Decreased, Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 3, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  White Blood Cell Decreased, Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 4, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  White Blood Cell Decreased, Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 4, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  White Blood Cell Decreased, Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 4, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  White Blood Cell Decreased, Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased, Grade 4, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  White Blood Cell Decreased, Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 0, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Leukocytosis , Grade 0, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 0, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Leukocytosis , Grade 0, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 0, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Leukocytosis , Grade 0, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 0, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Leukocytosis , Grade 0, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 1, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Leukocytosis , Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 1, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Leukocytosis , Grade 1, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 1, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Leukocytosis , Grade 1, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 1, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Leukocytosis , Grade 1, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 2, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Leukocytosis , Grade 2, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 2, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Leukocytosis , Grade 2, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 2, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Leukocytosis , Grade 2, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 2, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Leukocytosis , Grade 2, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 3, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Leukocytosis , Grade 3, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 3, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Leukocytosis , Grade 3, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 3, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Leukocytosis , Grade 3, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 3, Grade 4: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Leukocytosis , Grade 3, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 4, Grade 0: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Leukocytosis , Grade 4, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 4, Grade 1: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Leukocytosis , Grade 4, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 4, Grade 2: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Leukocytosis , Grade 4, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis , Grade 4, Grade 3: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Leukocytosis , Grade 4, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

28. Secondary Outcome: Part 2B: Number of Participants With Worst Case Hematology Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Normal ranges were 0.01 to 0.3*10^9 cells/L (basophils), 0 to 500 cells/L(eosinophils), 41 to 50 percentage of RBC in blood (hematocrit), 1,000 - 4,800 lymphocytes per microliter (ÂµL) of blood (lymphocytes), 80-100 fl (erythrocytes, mean corpuscular volume), 2 to 8 percentage of WBC (monocytes), 40 to 60 cells/mcL (neutrophils) and Women: 4.2 to 5.4 million RBC/ mcL of blood and Men: 4.7 to 6.1 million RBC/ mcL (erythrocytes count). Participants were counted in worst case category that their value changes to low, normal or no change [NC] or high), unless there is NC in their category. Participants whose laboratory value category was unchanged (e.g. High to High) or whose value became normal, were recorded in "To Normal or No Change" category. Participants were counted twice if participant had values that changed To Low and To High, so percentages may not add to 100%.
Time Frame: Up to approximately 367 weeks
Population: All Treated Population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B: Fela 0.100 mg/kg + Pembro 200 mg | Part 2B: Fela 0.300 mg/kg + Pembro 200 mg | Part 2B: Fela 1.000 mg/kg + Pembro 200 mg | Part 2B: Fela 3.000 mg/kg + Pembro 200 mg | Part 2B: Fela 24 mg + Pembro 200 mg | Part 2B: Fela 48 mg + Pembro 400 mg | Part 2B: Fela 160 mg + Pembro 400 mg | Part 2B: Fela 80 mg + Pembro 200 mg
Number analyzed (Participants) | 14 | 255 | 44 | 23 | 4 | 6 | 5 | 1
Participants
  Basophils, To Low: number analyzed (Participants) | 14 | 241 | 40 | 23 | 4 | 6 | 5 | 1
  Basophils, To Low | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils, To Normal or No Change: number analyzed (Participants) | 14 | 241 | 40 | 23 | 4 | 6 | 5 | 1
  Basophils, To Normal or No Change | 14 | 224 | 39 | 22 | 4 | 6 | 5 | 1
  Basophils, To High: number analyzed (Participants) | 14 | 241 | 40 | 23 | 4 | 6 | 5 | 1
  Basophils, To High | 0 | 10 | 1 | 1 | 0 | 0 | 0 | 0
  Eosinophils, To Low: number analyzed (Participants) | 14 | 249 | 42 | 23 | 4 | 6 | 5 | 1
  Eosinophils, To Low | 0 | 22 | 2 | 1 | 0 | 0 | 1 | 0
  Eosinophils, To Normal or No Change: number analyzed (Participants) | 14 | 249 | 42 | 23 | 4 | 6 | 5 | 1
  Eosinophils, To Normal or No Change | 14 | 192 | 29 | 20 | 4 | 6 | 4 | 1
  Eosinophils, To High: number analyzed (Participants) | 14 | 249 | 42 | 23 | 4 | 6 | 5 | 1
  Eosinophils, To High | 0 | 39 | 12 | 2 | 0 | 0 | 0 | 0
  Hematocrit, To Low: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Hematocrit, To Low | 4 | 73 | 18 | 7 | 4 | 3 | 0 | 0
  Hematocrit, To Normal or No Change: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Hematocrit, To Normal or No Change | 10 | 169 | 22 | 16 | 0 | 3 | 5 | 1
  Hematocrit, To High: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Hematocrit, To High | 0 | 12 | 3 | 0 | 0 | 0 | 0 | 0
  Lymphocytes, To Low: number analyzed (Participants) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
  Lymphocytes, To Low |  | 2 | 1 |  |  |  |  |
  Lymphocytes, To Normal or No Change: number analyzed (Participants) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
  Lymphocytes, To Normal or No Change |  | 0 | 0 |  |  |  |  |
  Lymphocytes, To High: number analyzed (Participants) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
  Lymphocytes, To High |  | 0 | 0 |  |  |  |  |
  Erythrocytes, Mean Corpuscular Volume, To Low: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Erythrocytes, Mean Corpuscular Volume, To Low |  | 0 |  |  |  |  |  |
  Erythrocytes, Mean Corpuscular Volume, To Normal or No Change: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Erythrocytes, Mean Corpuscular Volume, To Normal or No Change |  | 0 |  |  |  |  |  |
  Erythrocytes, Mean Corpuscular Volume, To High: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Erythrocytes, Mean Corpuscular Volume, To High |  | 1 |  |  |  |  |  |
  Monocytes, To Low: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Monocytes, To Low | 0 | 8 | 2 | 0 | 0 | 0 | 0 | 0
  Monocytes, To Normal or No Change: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Monocytes, To Normal or No Change | 11 | 181 | 27 | 15 | 2 | 5 | 5 | 1
  Monocytes, To High: number analyzed (Participants) | 14 | 252 | 42 | 23 | 4 | 6 | 5 | 1
  Monocytes, To High | 3 | 63 | 13 | 8 | 2 | 1 | 0 | 0
  Neutrophils, To Low: number analyzed (Participants) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
  Neutrophils, To Low |  | 0 | 0 |  |  |  |  |
  Neutrophils, To Normal or No Change: number analyzed (Participants) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
  Neutrophils, To Normal or No Change |  | 0 | 0 |  |  |  |  |
  Neutrophils, To High: number analyzed (Participants) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
  Neutrophils, To High |  | 2 | 1 |  |  |  |  |
  Erythrocytes, To Low: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Erythrocytes, To Low | 4 | 66 | 13 | 6 | 0 | 3 | 0 | 0
  Erythrocytes, To Normal or No Change: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Erythrocytes, To Normal or No Change | 10 | 180 | 29 | 16 | 3 | 3 | 5 | 1
  Erythrocytes, To High: number analyzed (Participants) | 14 | 253 | 42 | 23 | 4 | 6 | 5 | 1
  Erythrocytes, To High | 0 | 12 | 0 | 1 | 1 | 0 | 0 | 0

29. Secondary Outcome: Part 2B: Number of Participants With Worst Case Urinalysis Results Post-Baseline Relative to Baseline
Description: as for outcome 7
Time Frame: Up to approximately 367 weeks
Population: All treated population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B: Fela 0.100 mg/kg + Pembro 200 mg | Part 2B: Fela 0.300 mg/kg + Pembro 200 mg | Part 2B: Fela 1.000 mg/kg + Pembro 200 mg | Part 2B: Fela 3.000 mg/kg + Pembro 200 mg | Part 2B: Fela 24 mg + Pembro 200 mg | Part 2B: Fela 48 mg + Pembro 400 mg | Part 2B: Fela 160 mg + Pembro 400 mg | Part 2B: Fela 80 mg + Pembro 200 mg
Number analyzed (Participants) | 14 | 253 | 44 | 23 | 4 | 5 | 5 | 1
Participants
  Glucose, No Change/Decreased: number analyzed (Participants) | 14 | 252 | 44 | 23 | 4 | 5 | 5 | 1
  Glucose, No Change/Decreased | 14 | 228 | 42 | 21 | 4 | 5 | 5 | 1
  Glucose, Any increase: number analyzed (Participants) | 14 | 252 | 44 | 23 | 4 | 5 | 5 | 1
  Glucose, Any increase | 0 | 24 | 2 | 2 | 0 | 0 | 0 | 0
  Ketones, No Change/Decreased | 13 | 183 | 31 | 16 | 3 | 4 | 4 | 1
  Ketones, Any increase | 1 | 70 | 13 | 7 | 1 | 1 | 1 | 0
  Occult Blood, No Change/Decreased: number analyzed (Participants) | 11 | 236 | 40 | 22 | 4 | 5 | 5 | 1
  Occult Blood, No Change/Decreased | 8 | 129 | 28 | 15 | 3 | 2 | 4 | 1
  Occult Blood, Any increase: number analyzed (Participants) | 11 | 236 | 40 | 22 | 4 | 5 | 5 | 1
  Occult Blood, Any increase | 3 | 107 | 12 | 7 | 1 | 3 | 1 | 0

30. Secondary Outcome: Part 2B: Number of Participants With Dose Modifications of Feladilimab
Description: as for outcome 16
Time Frame: Up to approximately 367 weeks
Population: All treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B: Fela 0.100 mg/kg + Pembro 200 mg | Part 2B: Fela 0.300 mg/kg + Pembro 200 mg | Part 2B: Fela 1.000 mg/kg + Pembro 200 mg | Part 2B: Fela 3.000 mg/kg + Pembro 200 mg | Part 2B: Fela 24 mg + Pembro 200 mg | Part 2B: Fela 48 mg + Pembro 400 mg | Part 2B: Fela 160 mg + Pembro 400 mg | Part 2B: Fela 80 mg + Pembro 200 mg
Number analyzed (Participants) | 14 | 255 | 44 | 23 | 4 | 6 | 5 | 1
Participants
  Dose delays | 2 | 31 | 5 | 1 | 0 | 1 | 0 | 0
  Dose escalations | 0 | 10 | 1 | 1 | 0 | 0 | 0 | 0
  Infusion interruptions | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0

31. Secondary Outcome: Part 1A: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants with immune-related confirmed complete response (irCR) or ir confirmed partial response (irPR) per Immune-related Response Evaluation Criteria in Solid Tumors Criteria (irRECIST). irCR is defined as disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 millimeters (mm). irPR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters.
Time Frame: Up to approximately 367 weeks
Population: All Treated population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1A: Feladilimab (Fela) 0.001 Milligram/Kilogram (mg/kg) | Part 1A: Fela 0.003 mg/kg | Part 1A: Fela 0.010 mg/kg | Part 1A: Fela 0.030 mg/kg | Part 1A: Fela 0.100 mg/kg | Part 1A: Fela 0.300 mg/kg | Part 1A: Fela 1.000 mg/kg | Part 1A: Fela 3.000 mg/kg | Part 1A: Fela 10.000 mg/kg
Number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 15 | 27 | 7
Percentage of Participants | 0 [0.0 to 97.5] | 0 [0.0 to 97.5] | 0 [0.0 to 84.2] | 0 [0.0 to 41.0] | 8 [1.0 to 27.0] | 0 [0.0 to 13.7] | 0 [0.0 to 21.8] | 0 [0.0 to 12.8] | 0 [0.0 to 41.0]

32. Secondary Outcome: Part 1A: Disease Control Rate (DCR)
Description: DCR was defined as percentage of participants with best overall response of irCR or irPR at any time + ir stable disease (irSD) meeting the minimum time criteria from the start of treatment until ir disease progression (irPD) or death due to any cause or the start of new anticancer therapy/crossover. irCR is defined as disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm. irPR defined as at least 30% decrease in the sum of diameters of target lesions, taking as a reference, the baseline sum of the diameters. irSD defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease. IrPD defined as the date of radiological disease progression based on imaging data per irRECIST. A one-week visit window was considered in the duration of irSD, i.e. a minimum of 8 weeks (irSD>=9 weeks) and 17 weeks (irSD>=18 weeks) were considered.
Time Frame: Up to approximately 367 weeks
Population: All Treated population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1A: Feladilimab (Fela) 0.001 Milligram/Kilogram (mg/kg) | Part 1A: Fela 0.003 mg/kg | Part 1A: Fela 0.010 mg/kg | Part 1A: Fela 0.030 mg/kg | Part 1A: Fela 0.100 mg/kg | Part 1A: Fela 0.300 mg/kg | Part 1A: Fela 1.000 mg/kg | Part 1A: Fela 3.000 mg/kg | Part 1A: Fela 10.000 mg/kg
Number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 15 | 27 | 7
Percentage of Participants
  >=9 Weeks | 0 [0.0 to 97.5] | 0 [0.0 to 97.5] | 0 [0.0 to 84.2] | 43 [9.9 to 81.6] | 29 [12.6 to 51.1] | 28 [12.1 to 49.4] | 33 [11.8 to 61.6] | 22 [8.6 to 42.3] | 29 [3.7 to 71.0]
  >=18 Weeks | 0 [0.0 to 97.5] | 0 [0.0 to 97.5] | 0 [0.0 to 84.2] | 14 [0.4 to 57.9] | 17 [4.7 to 37.4] | 24 [9.4 to 45.1] | 13 [1.7 to 40.5] | 7 [0.9 to 24.3] | 0 [0.0 to 41.0]

33. Secondary Outcome: Part 1A: Overall Survival (OS)
Description: OS was defined as the interval between the date of first assigned study therapy/randomization and date of death due to any cause.
Time Frame: Up to approximately 367 weeks
Population: All Treated population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1A: Feladilimab (Fela) 0.001 Milligram/Kilogram (mg/kg) | Part 1A: Fela 0.003 mg/kg | Part 1A: Fela 0.010 mg/kg | Part 1A: Fela 0.030 mg/kg | Part 1A: Fela 0.100 mg/kg | Part 1A: Fela 0.300 mg/kg | Part 1A: Fela 1.000 mg/kg | Part 1A: Fela 3.000 mg/kg | Part 1A: Fela 10.000 mg/kg
Number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 15 | 27 | 7
Months | 4.3 [NA to NA] — 95% CI could not be estimated as only a single participant was analyzed. | 12.6 [NA to NA] — 95% CI could not be estimated as only a single participant was analyzed. | 14.0 [2.0 to 25.9] | 4.9 [3.5 to 8.0] | 6.7 [2.7 to 10.6] | 9.1 [4.0 to 12.9] | 9.1 [3.9 to 17.5] | 6.7 [5.4 to 9.2] | 7.3 [3.8 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events.

34. Secondary Outcome: Part 1A: Progression-free Survival (PFS)
Description: PFS was defined as the interval between the date of first dose of study treatment (or date of randomization for randomized cohorts) and the date of disease progression according to radiological response from investigator assessment, or death due to any cause, whichever occurs earlier. Disease progression was defined as the date of radiological disease progression based on imaging data per RECIST v1.1
Time Frame: Up to approximately 367 weeks
Population: All Treated
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1A: Feladilimab (Fela) 0.001 Milligram/Kilogram (mg/kg) | Part 1A: Fela 0.003 mg/kg | Part 1A: Fela 0.010 mg/kg | Part 1A: Fela 0.030 mg/kg | Part 1A: Fela 0.100 mg/kg | Part 1A: Fela 0.300 mg/kg | Part 1A: Fela 1.000 mg/kg | Part 1A: Fela 3.000 mg/kg | Part 1A: Fela 10.000 mg/kg
Number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 15 | 27 | 7
Months | 1.2 [NA to NA] — 95% CI could not be estimated as only a single participant was analyzed. | 1.9 [NA to NA] — 95% CI could not be estimated as only a single participant was analyzed. | 2.1 [2.0 to 2.1] | 2.1 [1.3 to 3.9] | 2.0 [1.5 to 2.1] | 1.9 [1.6 to 3.7] | 2.1 [1.2 to 4.2] | 1.9 [1.8 to 2.1] | 1.9 [1.6 to 4.0]

35. Secondary Outcome: Part 1A: Time to Overall Response (TTR)
Description: TTR was defined as the time from date of first dose of study treatment/randomization to the date of first documented confirmed (=4 weeks) CR or PR. CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 mm. PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters.
Time Frame: Up to approximately 367 weeks
Population: All Treated Population with a confirmed CR or PR. Only responders were included for the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1A: Feladilimab (Fela) 0.001 Milligram/Kilogram (mg/kg) | Part 1A: Fela 0.003 mg/kg | Part 1A: Fela 0.010 mg/kg | Part 1A: Fela 0.030 mg/kg | Part 1A: Fela 0.100 mg/kg | Part 1A: Fela 0.300 mg/kg | Part 1A: Fela 1.000 mg/kg | Part 1A: Fela 3.000 mg/kg | Part 1A: Fela 10.000 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Months |  |  |  |  | 2.3 [NA to NA] — 95% CI could not be estimated as only a single participant was analyzed. |  |  |  |

36. Secondary Outcome: Part 1A: Duration of Response (DOR)
Description: DOR was defined as the interval of time in months from the date of the first documented evidence of a response (confirmed CR or PR) to the date of first documented evidence of disease progression according to radiological response from investigator assessment per RECIST v1.1, or date of last adequate assessment of response or the date of death due to any cause (whichever occurs earlier). CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 mm. PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters. Disease progression was defined as the date of radiological disease progression based on imaging data per RECIST v1.1.
Time Frame: Up to approximately 367 weeks
Population: All Treated Population with a confirmed CR or PR. Only responders were included for the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1A: Feladilimab (Fela) 0.001 Milligram/Kilogram (mg/kg) | Part 1A: Fela 0.003 mg/kg | Part 1A: Fela 0.010 mg/kg | Part 1A: Fela 0.030 mg/kg | Part 1A: Fela 0.100 mg/kg | Part 1A: Fela 0.300 mg/kg | Part 1A: Fela 1.000 mg/kg | Part 1A: Fela 3.000 mg/kg | Part 1A: Fela 10.000 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Months |  |  |  |  | 10.3 [NA to NA] — 95% CI could not be estimated as only a single participant was analyzed. |  |  |  |

37. Secondary Outcome: Part 2A: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants with irCR or irPR per irRECIST. irCR is defined as disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeters (mm). irPR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters.
Time Frame: Up to approximately 367 weeks
Population: All Treated population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2A: Fela 0.010 mg/kg + Pembrolizumab (Pembro) 200 mg | Part 2A: Fela 0.030 mg/kg + Pembro 200 mg | Part 2A: Fela 0.100 mg/kg + Pembro 200 mg | Part 2A: Fela 0.300 mg/kg + Pembro 200 mg | Part 2A: Fela 1.000 mg/kg + Pembro 200 mg | Part 2A: Fela 3.000 mg/kg + Pembro 200 mg | Part 2A: Fela 8 mg + GSK3174998 8 mg | Part 2A: Fela 8 mg + GSK3174998 24 mg | Part 2A: Fela 24 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 80 mg | Part 2A: Fela 24 mg + Chemotherapy | Part 2A: Fela 80 mg + Chemotherapy | Part 2A: Fela 24 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 80 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 24 mg + Dostarlimab 500 mg + Cobolimab 300 mg | Part 2A: Fela 24 mg + Bintrafusp Alfa 2400 mg
Number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 16 | 4 | 3 | 6 | 36 | 13 | 22 | 1 | 4
Percentage of Participants | 20 [0.5 to 71.6] | 0 [0.0 to 52.2] | 20 [0.5 to 71.6] | 25 [3.2 to 65.1] | 27 [6.0 to 61.0] | 18 [2.3 to 51.8] | 0 [0.0 to 97.5] | 0 [0.0 to 60.2] | 0 [0.0 to 20.6] | 0 [0.0 to 60.2] | 33 [0.8 to 90.6] | 50 [11.8 to 88.2] | 14 [4.7 to 29.5] | 46 [19.2 to 74.9] | 41 [20.7 to 63.6] | 0 [0.0 to 97.5] | 50 [6.8 to 93.2]

38. Secondary Outcome: Part 2A: Disease Control Rate (DCR)
Description: DCR was defined as percentage of participants with best overall response of irCR or irPR at any time + irSD meeting the minimum time criteria from the start of treatment until irPD or death due to any cause or the start of new anticancer therapy/crossover. irCR defined as disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm. irPR defined as at least 30% decrease in the sum of diameters of target lesions, taking as a reference, the baseline sum of the diameters. irSD defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease. IrPD defined as the date of radiological disease progression based on imaging data per irRECIST. A one-week visit window was considered in the duration of irSD, i.e. a minimum of 8 weeks (irSD>=9 weeks) and 17 weeks (irSD>=18 weeks) were considered.
Time Frame: Up to approximately 367 weeks
Population: All Treated population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2A: Fela 0.010 mg/kg + Pembrolizumab (Pembro) 200 mg | Part 2A: Fela 0.030 mg/kg + Pembro 200 mg | Part 2A: Fela 0.100 mg/kg + Pembro 200 mg | Part 2A: Fela 0.300 mg/kg + Pembro 200 mg | Part 2A: Fela 1.000 mg/kg + Pembro 200 mg | Part 2A: Fela 3.000 mg/kg + Pembro 200 mg | Part 2A: Fela 8 mg + GSK3174998 8 mg | Part 2A: Fela 8 mg + GSK3174998 24 mg | Part 2A: Fela 24 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 80 mg | Part 2A: Fela 24 mg + Chemotherapy | Part 2A: Fela 80 mg + Chemotherapy | Part 2A: Fela 24 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 80 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 24 mg + Dostarlimab 500 mg + Cobolimab 300 mg | Part 2A: Fela 24 mg + Bintrafusp Alfa 2400 mg
Number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 16 | 4 | 3 | 6 | 36 | 13 | 22 | 1 | 4
Percentage of Participants
  >=9 Weeks | 20 [0.5 to 71.6] | 40 [5.3 to 85.3] | 40 [5.3 to 85.3] | 38 [8.5 to 75.5] | 27 [6.0 to 61.0] | 55 [23.4 to 83.3] | 0 [0.0 to 97.5] | 0 [0.0 to 60.2] | 19 [4.0 to 45.6] | 25 [0.6 to 80.6] | 33 [0.8 to 90.6] | 67 [22.3 to 95.7] | 58 [40.8 to 74.5] | 77 [46.2 to 95.0] | 86 [65.1 to 97.1] | 0 [0.0 to 97.5] | 50 [6.8 to 93.2]
  >=18 Weeks | 20 [0.5 to 71.6] | 0 [0.0 to 52.2] | 20 [0.5 to 71.6] | 25 [3.2 to 65.1] | 27 [6.0 to 61.0] | 36 [10.9 to 69.2] | 0 [0.0 to 97.5] | 0 [0.0 to 60.2] | 13 [1.6 to 38.3] | 0 [0.0 to 60.2] | 33 [0.8 to 90.6] | 67 [22.3 to 95.7] | 44 [27.9 to 61.9] | 62 [31.6 to 86.1] | 73 [49.8 to 89.3] | 0 [0.0 to 97.5] | 50 [6.8 to 93.2]

39. Secondary Outcome: Part 2A: Overall Survival (OS)
Description: as for outcome 33
Time Frame: Up to approximately 367 weeks
Population: All Treated
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2A: Fela 0.010 mg/kg + Pembrolizumab (Pembro) 200 mg | Part 2A: Fela 0.030 mg/kg + Pembro 200 mg | Part 2A: Fela 0.100 mg/kg + Pembro 200 mg | Part 2A: Fela 0.300 mg/kg + Pembro 200 mg | Part 2A: Fela 1.000 mg/kg + Pembro 200 mg | Part 2A: Fela 3.000 mg/kg + Pembro 200 mg | Part 2A: Fela 8 mg + GSK3174998 8 mg | Part 2A: Fela 8 mg + GSK3174998 24 mg | Part 2A: Fela 24 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 80 mg | Part 2A: Fela 24 mg + Chemotherapy | Part 2A: Fela 80 mg + Chemotherapy | Part 2A: Fela 24 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 80 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 24 mg + Dostarlimab 500 mg + Cobolimab 300 mg | Part 2A: Fela 24 mg + Bintrafusp Alfa 2400 mg
Number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 16 | 4 | 3 | 6 | 36 | 13 | 22 | 1 | 4
Months | NA [1.1 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 5.3 [1.9 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 9.3 [2.2 to 23.5] | 18.4 [6.9 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 12.7 [3.8 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 14.6 [4.4 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 4.1 [NA to NA] — 95% CI could not be estimated as only a single participant was analyzed. | 3.0 [0.8 to 13.9] | 8.2 [3.1 to 10.4] | 6.1 [1.2 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 8.6 [2.2 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 7.5 [5.7 to 13.8] | 8.2 [4.9 to 12.6] | 18.5 [9.4 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 16.1 [10.5 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | NA [NA to NA] — Median and 95% CI could not be estimated as only a single participant was analyzed. | NA [13.2 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events.

40. Secondary Outcome: Part 2A: Progression-free Survival (PFS)
Description: as for outcome 34
Time Frame: Up to approximately 367 weeks
Population: All Treated
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2A: Fela 0.010 mg/kg + Pembrolizumab (Pembro) 200 mg | Part 2A: Fela 0.030 mg/kg + Pembro 200 mg | Part 2A: Fela 0.100 mg/kg + Pembro 200 mg | Part 2A: Fela 0.300 mg/kg + Pembro 200 mg | Part 2A: Fela 1.000 mg/kg + Pembro 200 mg | Part 2A: Fela 3.000 mg/kg + Pembro 200 mg | Part 2A: Fela 8 mg + GSK3174998 8 mg | Part 2A: Fela 8 mg + GSK3174998 24 mg | Part 2A: Fela 24 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 80 mg | Part 2A: Fela 24 mg + Chemotherapy | Part 2A: Fela 80 mg + Chemotherapy | Part 2A: Fela 24 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 80 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 24 mg + Dostarlimab 500 mg + Cobolimab 300 mg | Part 2A: Fela 24 mg + Bintrafusp Alfa 2400 mg
Number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11 | 1 | 4 | 16 | 4 | 3 | 6 | 36 | 13 | 22 | 1 | 4
Months | 2.0 [1.1 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 1.9 [0.3 to 3.9] | 1.9 [1.8 to 6.0] | 2.1 [1.5 to 7.6] | 2.1 [1.4 to 7.2] | 2.0 [1.5 to 17.3] | 1.9 [NA to NA] — 95% CI could not be estimated as only a single participant was analyzed. | 1.7 [0.8 to 3.0] | 2.0 [1.4 to 2.1] | 1.6 [1.1 to 4.2] | 2.1 [1.7 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 5.7 [1.2 to 6.1] | 4.5 [2.6 to 6.0] | 6.7 [1.9 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 7.3 [4.1 to 10.7] | 1.9 [NA to NA] — 95% CI could not be estimated as only a single participant was analyzed. | NA [2.1 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events.

41. Secondary Outcome: Part 2A: Time to Overall Response (TTR)
Description: as for outcome 35
Time Frame: Up to approximately 367 weeks
Population: All Treated Population with a confirmed CR or PR. Only responders were included for the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2A: Fela 0.010 mg/kg + Pembrolizumab (Pembro) 200 mg | Part 2A: Fela 0.030 mg/kg + Pembro 200 mg | Part 2A: Fela 0.100 mg/kg + Pembro 200 mg | Part 2A: Fela 0.300 mg/kg + Pembro 200 mg | Part 2A: Fela 1.000 mg/kg + Pembro 200 mg | Part 2A: Fela 3.000 mg/kg + Pembro 200 mg | Part 2A: Fela 8 mg + GSK3174998 8 mg | Part 2A: Fela 8 mg + GSK3174998 24 mg | Part 2A: Fela 24 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 80 mg | Part 2A: Fela 24 mg + Chemotherapy | Part 2A: Fela 80 mg + Chemotherapy | Part 2A: Fela 24 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 80 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 24 mg + Dostarlimab 500 mg + Cobolimab 300 mg | Part 2A: Fela 24 mg + Bintrafusp Alfa 2400 mg
Number analyzed (Participants) | 1 | 0 | 1 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 6 | 7 | 0 | 2
Months | 2.1 [NA to NA] — 95% CI could not be estimated as only a single participant was analyzed. |  | 2.0 [NA to NA] — 95% CI could not be estimated as only a single participant was analyzed. | 2.8 [1.4 to 4.1] | 3.0 [1.9 to 4.0] | 11.0 [4.0 to 18.0] |  |  |  |  | 2.1 [NA to NA] — 95% CI could not be estimated as only a single participant was analyzed. | 1.6 [1.3 to 1.9] | 2.1 [2.0 to 4.0] | 1.6 [1.4 to 2.8] | 2.1 [1.4 to 4.2] |  | 2.1 [2.0 to 2.1]

42. Secondary Outcome: Part 2A: Duration of Response (DOR)
Description: DOR was defined as the interval of time in months from the date of the first documented evidence of a response (confirmed CR or PR) to the date of first documented evidence of disease progression according to radiological response from investigator assessment per RECIST v1.1, or date of last adequate assessment of response or the date of death due to any cause (whichever occurs earlier). CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 mm. PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters. Disease progression is defined as the date of radiological disease progression based on imaging data per RECIST v1.1.
Time Frame: Up to approximately 367 weeks
Population: All Treated Population with a confirmed CR or PR. Only responders are included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2A: Fela 0.010 mg/kg + Pembrolizumab (Pembro) 200 mg | Part 2A: Fela 0.030 mg/kg + Pembro 200 mg | Part 2A: Fela 0.100 mg/kg + Pembro 200 mg | Part 2A: Fela 0.300 mg/kg + Pembro 200 mg | Part 2A: Fela 1.000 mg/kg + Pembro 200 mg | Part 2A: Fela 3.000 mg/kg + Pembro 200 mg | Part 2A: Fela 8 mg + GSK3174998 8 mg | Part 2A: Fela 8 mg + GSK3174998 24 mg | Part 2A: Fela 24 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 80 mg | Part 2A: Fela 24 mg + Chemotherapy | Part 2A: Fela 80 mg + Chemotherapy | Part 2A: Fela 24 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 80 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 24 mg + Dostarlimab 500 mg + Cobolimab 300 mg | Part 2A: Fela 24 mg + Bintrafusp Alfa 2400 mg
Number analyzed (Participants) | 1 | 0 | 1 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 6 | 7 | 0 | 2
Months | NA [NA to NA] — Median and 95% CI could not be estimated as only a single participant was analyzed. |  | 4.1 [NA to NA] — 95% CI could not be estimated as only a single participant was analyzed. | 14.3 [6.3 to 22.2] | NA [3.2 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 13.8 [NA to NA] — 95% CI could not be estimated due to insufficient number of participants with events. |  |  |  |  | NA [NA to NA] — Median and 95% CI could not be estimated as only a single participant was analyzed. | 4.5 [4.2 to 4.8] | 22.5 [4.0 to 22.5] | NA [4.9 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 6.0 [4.6 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. |  | NA [NA to NA] — Median and 95% CI could not be estimated due to insufficient number of participants with events.

43. Secondary Outcome: Part 1B: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a confirmed irCR or confirmed irPR per irRECIST. irCR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. irPR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters.
Time Frame: Up to approximately 367 weeks
Population: All Treated population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1B: Fela 0.300 mg/kg | Part 1B: Fela 1.000 mg/kg | Part 1B: Fela 24 mg
Number analyzed (Participants) | 39 | 115 | 59
Percentage of Participants | 5 [0.6 to 17.3] | 4 [1.4 to 9.9] | 8 [2.8 to 18.7]

44. Secondary Outcome: Part 1B: Disease Control Rate (DCR)
Description: DCR was defined as percentage of participants with best overall response of irCR or irPR at any time + irSD meeting the minimum time criteria from the start of treatment until irPD or death due to any cause or the start of new anticancer therapy/crossover. irCR is defined as disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm. irPR defined as at least 30% decrease in the sum of diameters of target lesions, taking as a reference, the baseline sum of the diameters. irSD defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease. IrPD defined as the date of radiological disease progression based on imaging data per irRECIST. A one-week visit window was considered in the duration of irSD, i.e. a minimum of 8 weeks (irSD>=9 weeks) and 17 weeks (irSD>=18 weeks) were considered.
Time Frame: Up to approximately 367 weeks
Population: All Treated population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1B: Fela 0.300 mg/kg | Part 1B: Fela 1.000 mg/kg | Part 1B: Fela 24 mg
Number analyzed (Participants) | 39 | 115 | 59
Percentage of Participants
  >=9 Weeks | 38 [23.4 to 55.4] | 39 [30.2 to 48.7] | 39 [26.5 to 52.6]
  >=18 Weeks | 23 [11.1 to 39.3] | 23 [15.3 to 31.3] | 19 [9.7 to 30.9]

45. Secondary Outcome: Part 1B: Overall Survival (OS)
Description: as for outcome 33
Time Frame: Up to approximately 367 weeks
Population: All Treated
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1B: Fela 0.300 mg/kg | Part 1B: Fela 1.000 mg/kg | Part 1B: Fela 24 mg
Number analyzed (Participants) | 39 | 115 | 59
Months | 10.5 [6.7 to 17.3] | 9.4 [7.9 to 12.9] | 7.8 [6.5 to 8.7]

46. Secondary Outcome: Part 1B: Progression-free Survival (PFS)
Description: as for outcome 34
Time Frame: Up to approximately 367 weeks
Population: All Treated
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1B: Fela 0.300 mg/kg | Part 1B: Fela 1.000 mg/kg | Part 1B: Fela 24 mg
Number analyzed (Participants) | 39 | 115 | 59
Months | 2.1 [2.0 to 3.9] | 2.1 [2.0 to 2.6] | 2.1 [2.0 to 2.3]

47. Secondary Outcome: Part 1B: Time to Overall Response (TTR)
Description: as for outcome 35
Time Frame: Up to approximately 367 weeks
Population: All Treated Population with a confirmed CR or PR. Only responders are included in the analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1B: Fela 0.300 mg/kg | Part 1B: Fela 1.000 mg/kg | Part 1B: Fela 24 mg
Number analyzed (Participants) | 2 | 2 | 3
Months | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 3.9] | 3.8 [2.0 to 4.3]

48. Secondary Outcome: Part 1B: Duration of Response (DOR)
Description: as for outcome 42
Time Frame: Up to approximately 367 weeks
Population: All Treated Population with a confirmed CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1B: Fela 0.300 mg/kg | Part 1B: Fela 1.000 mg/kg | Part 1B: Fela 24 mg
Number analyzed (Participants) | 2 | 2 | 3
Months | 7.3 [4.2 to 10.4] | 11.8 [6.1 to 17.5] | 7.2 [6.1 to 8.2]

49. Secondary Outcome: Part 2B: Overall Response Rate (ORR)
Description: as for outcome 43
Time Frame: Up to approximately 367 weeks
Population: All Treated population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2B: Fela 0.100 mg/kg + Pembro 200 mg | Part 2B: Fela 0.300 mg/kg + Pembro 200 mg | Part 2B: Fela 1.000 mg/kg + Pembro 200 mg | Part 2B: Fela 3.000 mg/kg + Pembro 200 mg | Part 2B: Fela 24 mg + Pembro 200 mg | Part 2B: Fela 48 mg + Pembro 400 mg | Part 2B: Fela 160 mg + Pembro 400 mg | Part 2B: Fela 80 mg + Pembro 200 mg
Number analyzed (Participants) | 14 | 255 | 44 | 23 | 4 | 6 | 5 | 1
Percentage of Participants | 7 [0.2 to 33.9] | 20 [14.9 to 25.0] | 18 [8.2 to 32.7] | 30 [13.2 to 52.9] | 0 [0.0 to 60.2] | 17 [0.4 to 64.1] | 0 [0.0 to 52.2] | 0 [0.0 to 97.5]

50. Secondary Outcome: Part 2B: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants with a best overall response of irCR or irPR at any time plus irSD meeting the minimum time criteria from the start of treatment until irPD or death due to any cause or the start of new anticancer therapy/crossover. irCR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. irPR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters. irSD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease. irPD is defined as the date of radiological disease progression based on imaging data per irRECIST. A one-week visit window was considered in the duration of irSD, i.e. a minimum of 8 weeks (irSD>=9 weeks) and 17 weeks (irSD>=18 weeks) were considered.
Time Frame: Up to approximately 367 weeks
Population: All Treated population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2B: Fela 0.100 mg/kg + Pembro 200 mg | Part 2B: Fela 0.300 mg/kg + Pembro 200 mg | Part 2B: Fela 1.000 mg/kg + Pembro 200 mg | Part 2B: Fela 3.000 mg/kg + Pembro 200 mg | Part 2B: Fela 24 mg + Pembro 200 mg | Part 2B: Fela 48 mg + Pembro 400 mg | Part 2B: Fela 160 mg + Pembro 400 mg | Part 2B: Fela 80 mg + Pembro 200 mg
Number analyzed (Participants) | 14 | 255 | 44 | 23 | 4 | 6 | 5 | 1
Percentage of Participants
  >=9 Weeks | 29 [8.4 to 58.1] | 58 [52.1 to 64.5] | 43 [28.3 to 59.0] | 57 [34.5 to 76.8] | 50 [6.8 to 93.2] | 33 [4.3 to 77.7] | 0 [0.0 to 52.2] | 0 [0.0 to 97.5]
  >=18 Weeks | 21 [4.7 to 50.8] | 39 [32.8 to 45.1] | 27 [15.0 to 42.8] | 35 [16.4 to 57.3] | 25 [0.6 to 80.6] | 33 [4.3 to 77.7] | 0 [0.0 to 52.2] | 0 [0.0 to 97.5]

51. Secondary Outcome: Part 2B: Overall Survival (OS)
Description: as for outcome 33
Time Frame: Up to approximately 367 weeks
Population: All Treated
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2B: Fela 0.100 mg/kg + Pembro 200 mg | Part 2B: Fela 0.300 mg/kg + Pembro 200 mg | Part 2B: Fela 1.000 mg/kg + Pembro 200 mg | Part 2B: Fela 3.000 mg/kg + Pembro 200 mg | Part 2B: Fela 24 mg + Pembro 200 mg | Part 2B: Fela 48 mg + Pembro 400 mg | Part 2B: Fela 160 mg + Pembro 400 mg | Part 2B: Fela 80 mg + Pembro 200 mg
Number analyzed (Participants) | 14 | 255 | 44 | 23 | 4 | 6 | 5 | 1
Months | 8.9 [3.4 to 15.6] | 12.5 [10.1 to 15.2] | 12.1 [8.9 to 19.9] | 10.8 [5.3 to 28.1] | NA [2.3 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | NA [2.7 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 4.7 [0.5 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 1.1 [NA to NA] — 95% CI could not be estimated as only a single participant was analyzed.

52. Secondary Outcome: Part 2B: Progression-free Survival (PFS)
Description: as for outcome 34
Time Frame: Up to approximately 367 weeks
Population: All Treated
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2B: Fela 0.100 mg/kg + Pembro 200 mg | Part 2B: Fela 0.300 mg/kg + Pembro 200 mg | Part 2B: Fela 1.000 mg/kg + Pembro 200 mg | Part 2B: Fela 3.000 mg/kg + Pembro 200 mg | Part 2B: Fela 24 mg + Pembro 200 mg | Part 2B: Fela 48 mg + Pembro 400 mg | Part 2B: Fela 160 mg + Pembro 400 mg | Part 2B: Fela 80 mg + Pembro 200 mg
Number analyzed (Participants) | 14 | 255 | 44 | 23 | 4 | 6 | 5 | 1
Months | 2.6 [1.1 to 4.2] | 3.9 [2.8 to 4.0] | 2.3 [2.0 to 4.0] | 4.4 [2.1 to 6.4] | 2.1 [1.1 to 8.4] | 3.1 [1.4 to 13.7] | 1.5 [0.5 to 2.3] | 0.8 [NA to NA] — 95% CI could not be estimated as only a single participant was analyzed.

53. Secondary Outcome: Part 2B: Time to Overall Response (TTR)
Description: as for outcome 35
Time Frame: Up to approximately 367 weeks
Population: All Treated Population with a confirmed CR or PR. Only responders were included for the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2B: Fela 0.100 mg/kg + Pembro 200 mg | Part 2B: Fela 0.300 mg/kg + Pembro 200 mg | Part 2B: Fela 1.000 mg/kg + Pembro 200 mg | Part 2B: Fela 3.000 mg/kg + Pembro 200 mg | Part 2B: Fela 24 mg + Pembro 200 mg | Part 2B: Fela 48 mg + Pembro 400 mg | Part 2B: Fela 160 mg + Pembro 400 mg | Part 2B: Fela 80 mg + Pembro 200 mg
Number analyzed (Participants) | 1 | 44 | 8 | 6 | 0 | 1 | 0 | 0
Months | 2.1 [NA to NA] — 95% CI could not be estimated as only a single participant was analyzed. | 2.1 [2.0 to 3.9] | 2.0 [1.3 to 2.6] | 2.1 [1.9 to 4.1] |  | 2.2 [NA to NA] — 95% CI could not be estimated as only a single participant was analyzed. |  |

54. Secondary Outcome: Part 2B: Duration of Response (DOR)
Description: DOR was defined as the interval of time in months from the date of the first documented evidence of a response (confirmed CR or PR) to the date of first documented evidence of disease progression according to radiological response from investigator assessment per RECIST v1.1, or date of last adequate assessment of response or the date of death due to any cause (whichever occurs earlier). CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters. Disease progression is defined as the date of radiological disease progression based on imaging data per RECIST v1.1
Time Frame: Up to approximately 367 weeks
Population: All Treated Population with a confirmed CR or PR. Only responders were included for the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2B: Fela 0.100 mg/kg + Pembro 200 mg | Part 2B: Fela 0.300 mg/kg + Pembro 200 mg | Part 2B: Fela 1.000 mg/kg + Pembro 200 mg | Part 2B: Fela 3.000 mg/kg + Pembro 200 mg | Part 2B: Fela 24 mg + Pembro 200 mg | Part 2B: Fela 48 mg + Pembro 400 mg | Part 2B: Fela 160 mg + Pembro 400 mg | Part 2B: Fela 80 mg + Pembro 200 mg
Number analyzed (Participants) | 1 | 44 | 8 | 6 | 0 | 1 | 0 | 0
Months | 6.1 [NA to NA] — 95% CI could not be estimated as only a single participant was analyzed. | 13.8 [8.3 to 19.5] | 18.7 [4.3 to 38.0] | 24.6 [2.6 to 24.6] |  | 11.5 [NA to NA] — 95% CI could not be estimated as only a single participant was analyzed. |  |

55. Secondary Outcome: Part 1A: Maximum Observed Plasma Concentration (Cmax) and Minimum Observed Plasma Concentration (Ctau) of Feladilimab
Description: Blood samples were collected for Pharmacokinetic (PK) analysis. PK analysis was calculated based on standard non-compartmental method.
Time Frame: Pre-dose; end of infusion (EOI); 0.5, 1, 2, 4, 6, 8, 24, 48-72, 96-120 hours POST EOI; week 1; week 2; Pre-dose and 0.5 hours POST EOI in week 3; week 4; week 5; Pre-dose and 0.5 hours POST EOI in week 6, 9, 12 15; Pre-dose in week 21 and 33
Population: Pharmacokinetic Population included as all participants from the all treated population for whom a PK sample was obtained and analyzed. Only those participants with data available at specified categories have been analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram/millilitre (ug/mL)
Arm/Group | Part 1A: Fela 0.003 mg/kg | Part 1A: Feladilimab (Fela) 0.001 Milligram/Kilogram (mg/kg) | Part 1A: Fela 0.010 mg/kg | Part 1A: Fela 0.030 mg/kg | Part 1A: Fela 0.100 mg/kg | Part 1A: Fela 0.300 mg/kg | Part 1A: Fela 1.000 mg/kg | Part 1A: Fela 3.000 mg/kg | Part 1A: Fela 10.000 mg/kg
Number analyzed (Participants) | 1 | 1 | 2 | 3 | 5 | 3 | 4 | 3 | 3
Microgram/millilitre (ug/mL)
  Cmax, Cycle 1 | 0.0887 (NA) — Geometric coefficient of variation could not be calculated for single participant. | NA (NA) — No concentration data were collected. Therefore, no PK analysis was performed. | 0.2038 (12.6253) | 1.7433 (90.5940) | 2.3041 (14.0076) | 6.4643 (23.7989) | 18.3809 (24.4093) | 74.7985 (16.0934) | 193.7782 (17.1955)
  Ctau, Cycle 1: number analyzed (Participants) | 1 | 1 | 0 | 0 | 5 | 3 | 3 | 3 | 3
  Ctau, Cycle 1 | NA (NA) — No concentration data were collected. Therefore, no PK analysis was performed. | NA (NA) — No concentration data were collected. Therefore, no PK analysis was performed. |  |  | 0.2868 (62.2180) | 1.0533 (9.2565) | 4.3093 (21.6033) | 11.3112 (85.3459) | 38.0810 (22.3643)
  Ctau, Cycle 6: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1
  Ctau, Cycle 6 | NA (NA) — No concentration data were collected. Therefore, no PK analysis was performed. | NA (NA) — No concentration data were collected. Therefore, no PK analysis was performed. |  | 0.2426 (NA) — Geometric coefficient of variation could not be calculated for single participant. | 0.3510 (NA) — Geometric coefficient of variation could not be calculated for single participant. |  | 11.9562 (NA) — Geometric coefficient of variation could not be calculated for single participant. |  | 35.9660 (NA) — Geometric coefficient of variation could not be calculated for single participant.

56. Secondary Outcome: Part 1A: Area Under the Concentration-time Curve From Time 0 to 504 Hours After Dosing [AUC (0-504h)] of Feladilimab
Description: Blood samples were collected for PK analysis. PK analysis was calculated based on standard non-compartmental method.
Time Frame: Pre-dose; end of infusion (EOI); 0.5, 1, 2, 4, 6, 8, 24, 48-72, 96-120 hours post-EOI; week 1; week 2; Pre-dose and 0.5 hours post-EOI in week 3; week 4; week 5; Pre-dose and 0.5 hours post-EOI in week 6, 9, 12 15; Pre-dose in week 21 and 33
Population: Pharmacokinetic Population. As pre-specified in the protocol, only specified treatment arms were planned for this outcome measure and hence there are 0 participants analyzed for rest of the arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*microgram/millilitre (h*ug/mL)
Arm/Group | Part 1A: Feladilimab (Fela) 0.001 Milligram/Kilogram (mg/kg) | Part 1A: Fela 0.003 mg/kg | Part 1A: Fela 0.010 mg/kg | Part 1A: Fela 0.030 mg/kg | Part 1A: Fela 0.100 mg/kg | Part 1A: Fela 0.300 mg/kg | Part 1A: Fela 1.000 mg/kg | Part 1A: Fela 3.000 mg/kg | Part 1A: Fela 10.000 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 1 | 5 | 2 | 1 | 1 | 0
Hour*microgram/millilitre (h*ug/mL) |  |  |  | 134.6206 (NA) — Geometric coefficient of variation could not be calculated for single participant. | 373.6877 (23.2053) | 1156.5768 (6.8031) | 4839.0026 (NA) — Geometric coefficient of variation could not be calculated for single participant. | 11368.0960 (NA) — Geometric coefficient of variation could not be calculated for single participant. |

57. Secondary Outcome: Part 2A: Ctau of Pembrolizumab
Description: Blood samples were collected for PK analysis. PK analysis was calculated based on standard non-compartmental method.
Time Frame: Pre-dose and 24 hours post-EOI on day 1; week 1; week 2; Pre-dose in week 3; week 4; week 5; Pre-dose in week 9, 15, 18, 21, 33, 45, 57, 69, 81 and 93
Population: Pharmacokinetic Population. Data is presented for participants who received feladilimab in combination with Pembrolizumab. Only those participants with data available at specified categories have been analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part 2A: Fela 0.010 mg/kg + Pembrolizumab (Pembro) 200 mg | Part 2A: Fela 0.030 mg/kg + Pembro 200 mg | Part 2A: Fela 0.100 mg/kg + Pembro 200 mg | Part 2A: Fela 0.300 mg/kg + Pembro 200 mg | Part 2A: Fela 1.000 mg/kg + Pembro 200 mg | Part 2A: Fela 3.000 mg/kg + Pembro 200 mg
Number analyzed (Participants) | 3 | 2 | 5 | 4 | 5 | 7
ug/mL
  Cycle 1 | 10.8032 (55.7461) | 19.2951 (41.0160) | 16.7039 (47.9340) | 13.9035 (31.9060) | 12.9277 (42.3634) | 15.1724 (40.5000)
  Cycle 6: number analyzed (Participants) | 1 | 1 | 0 | 2 | 1 | 3
  Cycle 6 | 35.1000 (NA) — Geometric coefficient of variation could not be calculated for single participant. | 62.3000 (NA) — Geometric coefficient of variation could not be calculated for single participant. |  | 35.3321 (21.9877) | 35.6000 (NA) — Geometric coefficient of variation could not be calculated for single participant. | 35.6444 (63.8554)

58. Secondary Outcome: Part 2A: AUC (0-504h) of Pembrolizumab
Description: Blood samples were collected for PK analysis. PK analysis was calculated based on standard non-compartmental method.
Time Frame: as for outcome 57
Population: Pharmacokinetic Population. Data is presented for participants who received feladilimab in combination with Pembrolizumab. As pre-specified in the protocol, only specified treatment arms were planned and hence there are 0 participants analyzed for rest of the arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Part 2A: Fela 0.010 mg/kg + Pembrolizumab (Pembro) 200 mg | Part 2A: Fela 0.030 mg/kg + Pembro 200 mg | Part 2A: Fela 0.100 mg/kg + Pembro 200 mg | Part 2A: Fela 0.300 mg/kg + Pembro 200 mg | Part 2A: Fela 1.000 mg/kg + Pembro 200 mg | Part 2A: Fela 3.000 mg/kg + Pembro 200 mg
Number analyzed (Participants) | 1 | 0 | 0 | 1 | 1 | 2
h*ug/mL | 11363.9193 (NA) — Geometric coefficient of variation could not be calculated for single participant. |  |  | 11556.7001 (NA) — Geometric coefficient of variation could not be calculated for single participant. | 19158.7768 (NA) — Geometric coefficient of variation could not be calculated for single participant. | 17928.7606 (32.2374)

59. Secondary Outcome: Part 2A: Cmax and Ctau of GSK3174998
Description: Blood samples were collected for PK analysis. PK analysis was calculated based on standard non-compartmental method.
Time Frame: as for outcome 57
Population: Pharmacokinetic Population. Data is presented for participants who received feladilimab in combination with GSK3174998. As pre-specified in the protocol, only specified treatment arms were planned and hence there are 0 participants analyzed for rest of the arms. Only those participants with data available at specified categories have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part 2A: Fela 8 mg + GSK3174998 8 mg | Part 2A: Fela 8 mg + GSK3174998 24 mg | Part 2A: Fela 24 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 80 mg
Number analyzed (Participants) | 0 | 3 | 16 | 4 | 3
ug/mL
  Cmax, Cycle 1 |  | 5.1078 (27.7040) | 6.6367 (47.5930) | 5.5967 (10.5455) | 22.7767 (13.7397)
  Ctau, Cycle 1: number analyzed (Participants) | 0 | 1 | 10 | 2 | 3
  Ctau, Cycle 1 |  | 0.6700 (NA) — Geometric coefficient of variation could not be calculated for single participant. | 0.6484 (52.4342) | 0.5893 (72.0699) | 4.5862 (50.0449)
  Ctau, Cycle 6: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0
  Ctau, Cycle 6 |  |  | 0.5663 (94.4364) |  |

60. Secondary Outcome: Part 2A: AUC (0-504 h) of GSK3174998
Description: Blood samples were collected for PK analysis. PK analysis was calculated based on standard non-compartmental method.
Time Frame: as for outcome 57
Population: Pharmacokinetic Population. Data is presented for participants who received feladilimab in combination with GSK3174998. As pre-specified in the protocol, only specified treatment arms were planned and hence there are 0 participants analyzed for rest of the arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Part 2A: Fela 8 mg + GSK3174998 8 mg | Part 2A: Fela 8 mg + GSK3174998 24 mg | Part 2A: Fela 24 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 80 mg
Number analyzed (Participants) | 0 | 1 | 7 | 3 | 2
h*ug/mL |  | 1038.4544 (NA) — Geometric coefficient of variation could not be calculated for single participant. | 953.0313 (9.2381) | 703.8874 (2.7723) | 4606.4365 (21.6164)

61. Secondary Outcome: Part 1B: Cmax and Ctau of Feladilimab
Description: Blood samples were collected for PK analysis. PK analysis was calculated based on standard non-compartmental method.
Time Frame: Pre-dose; end of infusion (EOI); 0.5, 1, 2, 4, 6, 8, 24, 48-72, 96-120 hours post-EOI; week 1; week 2; Pre-dose and 0.5 hours post-EOI in week 3; week 4; week 5; Pre-dose and 0.5 hours post-EOI in week 6, 9, 12 15; Pre-dose in week 21, 33 and 45
Population: Pharmacokinetic Population. Only those participants with data available at specified categories have been analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part 1B: Fela 0.300 mg/kg | Part 1B: Fela 1.000 mg/kg | Part 1B: Fela 24 mg
Number analyzed (Participants) | 18 | 29 | 34
ug/mL
  BIOMARKER, Cmax, Cycle 1: number analyzed (Participants) | 0 | 0 | 34
  BIOMARKER, Cmax, Cycle 1 |  |  | 6.9732 (25.8747)
  BIOMARKER, Ctau, Cycle 1: number analyzed (Participants) | 0 | 0 | 18
  BIOMARKER, Ctau, Cycle 1 |  |  | 1.1411 (45.6223)
  BIOMARKER, Ctau, Cycle 6: number analyzed (Participants) | 0 | 0 | 2
  BIOMARKER, Ctau, Cycle 6 |  |  | 2.0597 (61.8911)
  BLADDER/UROTHELIAL, Cmax, Cycle 1: number analyzed (Participants) | 3 | 11 | 0
  BLADDER/UROTHELIAL, Cmax, Cycle 1 | 3.2855 (98.7868) | 25.8491 (15.5203) |
  BLADDER/UROTHELIAL, Ctau, Cycle 1: number analyzed (Participants) | 3 | 10 | 0
  BLADDER/UROTHELIAL, Ctau, Cycle 1 | 0.5029 (151.5778) | 5.3950 (39.3125) |
  BLADDER/UROTHELIAL, Ctau, Cycle 6: number analyzed (Participants) | 0 | 4 | 0
  BLADDER/UROTHELIAL, Ctau, Cycle 6 |  | 13.6665 (21.8363) |
  CERVICAL, Cmax, Cycle 1: number analyzed (Participants) | 0 | 10 | 0
  CERVICAL, Cmax, Cycle 1 |  | 27.2607 (28.7319) |
  CERVICAL, Ctau, Cycle 1: number analyzed (Participants) | 0 | 9 | 0
  CERVICAL, Ctau, Cycle 1 |  | 3.8347 (51.9848) |
  CERVICAL, Ctau, Cycle 6: number analyzed (Participants) | 0 | 2 | 0
  CERVICAL, Ctau, Cycle 6 |  | 12.7002 (14.0710) |
  JAPAN PK/PD, Cmax, Cycle 1: number analyzed (Participants) | 4 | 3 | 0
  JAPAN PK/PD, Cmax, Cycle 1 | 5.8973 (10.9555) | 22.4768 (11.3862) |
  JAPAN PK/PD, Ctau, Cycle 1: number analyzed (Participants) | 3 | 3 | 0
  JAPAN PK/PD, Ctau, Cycle 1 | 1.2533 (9.3514) | 5.1381 (12.9597) |
  JAPAN PK/PD, Ctau, Cycle 6: number analyzed (Participants) | 0 | 1 | 0
  JAPAN PK/PD, Ctau, Cycle 6 |  | 10.9800 (NA) — Geometric coefficient of variation could not be calculated for single participant. |
  MELANOMA, Cmax, Cycle 1: number analyzed (Participants) | 18 | 18 | 0
  MELANOMA, Cmax, Cycle 1 | 6.2711 (24.5290) | 23.9959 (23.9522) |
  MELANOMA, Ctau, Cycle 1: number analyzed (Participants) | 16 | 15 | 0
  MELANOMA, Ctau, Cycle 1 | 1.2025 (33.0632) | 4.3924 (55.2035) |
  MELANOMA, Ctau, Cycle 6: number analyzed (Participants) | 7 | 5 | 0
  MELANOMA, Ctau, Cycle 6 | 2.6320 (46.3462) | 11.2405 (32.8873) |
  MSI-H/DMMR, Cmax, Cycle 1: number analyzed (Participants) | 10 | 12 | 0
  MSI-H/DMMR, Cmax, Cycle 1 | 5.4181 (38.5999) | 25.6766 (27.3384) |
  MSI-H/DMMR, Ctau, Cycle 1: number analyzed (Participants) | 10 | 10 | 0
  MSI-H/DMMR, Ctau, Cycle 1 | 0.9976 (41.4153) | 5.1437 (46.0134) |
  MSI-H/DMMR, Ctau, Cycle 6: number analyzed (Participants) | 4 | 4 | 0
  MSI-H/DMMR, Ctau, Cycle 6 | 2.5409 (61.5161) | 9.7769 (143.2225) |
  NSCLC, Cmax, Cycle 1: number analyzed (Participants) | 5 | 29 | 0
  NSCLC, Cmax, Cycle 1 | 8.4009 (38.8531) | 24.2697 (29.1958) |
  NSCLC, Ctau, Cycle 1: number analyzed (Participants) | 4 | 27 | 0
  NSCLC, Ctau, Cycle 1 | 1.4713 (39.3325) | 5.4292 (55.3073) |
  NSCLC, Ctau, Cycle 6: number analyzed (Participants) | 1 | 9 | 0
  NSCLC, Ctau, Cycle 6 | 4.2630 (NA) — Geometric coefficient of variation could not be calculated for single participant. | 8.6574 (62.7001) |
  VIRAL-POSITIVE, Cmax, Cycle 1: number analyzed (Participants) | 0 | 17 | 0
  VIRAL-POSITIVE, Cmax, Cycle 1 |  | 24.2995 (25.3201) |
  VIRAL-POSITIVE, Ctau, Cycle 1: number analyzed (Participants) | 0 | 16 | 0
  VIRAL-POSITIVE, Ctau, Cycle 1 |  | 5.0751 (45.1953) |
  VIRAL-POSITIVE, Ctau, Cycle 6: number analyzed (Participants) | 0 | 3 | 0
  VIRAL-POSITIVE, Ctau, Cycle 6 |  | 11.0416 (36.7974) |

62. Secondary Outcome: Part 1B: AUC (0-504 h) of Feladilimab
Description: Blood samples were collected for PK analysis. PK analysis was calculated based on standard non-compartmental method.
Time Frame: as for outcome 61
Population: Pharmacokinetic Population. Only those participants with data available at specified categories have been analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Part 1B: Fela 0.300 mg/kg | Part 1B: Fela 1.000 mg/kg | Part 1B: Fela 24 mg
Number analyzed (Participants) | 12 | 30 | 11
h*ug/mL
  BIOMARKER: number analyzed (Participants) | 0 | 0 | 11
  BIOMARKER |  |  | 1076.8681 (27.3988)
  BLADDER/UROTHELIAL: number analyzed (Participants) | 1 | 5 | 0
  BLADDER/UROTHELIAL | 632.0762 (NA) — Geometric coefficient of variation could not be calculated for single participant. | 5026.8004 (24.5736) |
  CERVICAL: number analyzed (Participants) | 0 | 4 | 0
  CERVICAL |  | 5222.1970 (5.6103) |
  JAPAN PK/PD: number analyzed (Participants) | 4 | 3 | 0
  JAPAN PK/PD | 1237.7314 (9.6008) | 4525.7373 (5.5353) |
  MELANOMA: number analyzed (Participants) | 12 | 9 | 0
  MELANOMA | 1206.7402 (18.6679) | 4048.7261 (29.9449) |
  MSI-H/DMMR: number analyzed (Participants) | 4 | 4 | 0
  MSI-H/DMMR | 1048.2771 (24.6105) | 5952.2979 (59.1357) |
  NSCLC: number analyzed (Participants) | 0 | 30 | 0
  NSCLC |  | 4731.8292 (31.1548) |
  VIRAL-POSITIVE: number analyzed (Participants) | 0 | 10 | 0
  VIRAL-POSITIVE |  | 4337.5163 (26.4590) |

63. Secondary Outcome: Part 2B: Cmax and Ctau of Feladilimab
Description: Blood samples were collected for PK analysis. PK analysis was calculated based on standard non-compartmental method.
Time Frame: Pre-dose; EOI; 0.5, 1, 2, 4, 6, 8, 24, 48-72, 96-120 hours post-EOI; week 1; week 2; Pre-dose and 0.5 hours post-EOI in week 3; week 4; week 5; Pre-dose and 0.5, 4 hours post-EOI in week 6, 9, 12 and15; Pre-dose in week 18, 21, 33, 45, 57, 69, 81 and 93
Population: Pharmacokinetic Population. Data is presented for participants who received feladilimab in combination with Pembro. Only those participants with data available at specified categories have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part 2B: Fela 0.100 mg/kg + Pembro 200 mg | Part 2B: Fela 0.300 mg/kg + Pembro 200 mg | Part 2B: Fela 1.000 mg/kg + Pembro 200 mg | Part 2B: Fela 3.000 mg/kg + Pembro 200 mg | Part 2B: Fela 24 mg + Pembro 200 mg | Part 2B: Fela 48 mg + Pembro 400 mg | Part 2B: Fela 160 mg + Pembro 400 mg | Part 2B: Fela 80 mg + Pembro 200 mg
Number analyzed (Participants) | 13 | 91 | 24 | 22 | 3 | 2 | 2 | 1
ug/mL
  BLADDER/UROTHELIAL, Cmax, Cycle 1: number analyzed (Participants) | 0 | 44 | 0 | 0 | 0 | 0 | 0 | 0
  BLADDER/UROTHELIAL, Cmax, Cycle 1 |  | 7.0435 (16.0950) |  |  |  |  |  |
  BLADDER/UROTHELIAL, Ctau, Cycle 1: number analyzed (Participants) | 0 | 37 | 0 | 0 | 0 | 0 | 0 | 0
  BLADDER/UROTHELIAL, Ctau, Cycle 1 |  | 1.1346 (49.2057) |  |  |  |  |  |
  BLADDER/UROTHELIAL, Ctau, Cycle 6: number analyzed (Participants) | 0 | 12 | 0 | 0 | 0 | 0 | 0 | 0
  BLADDER/UROTHELIAL, Ctau, Cycle 6 |  | 2.5980 (39.5677) |  |  |  |  |  |
  CERVICAL, Cmax, Cycle 1: number analyzed (Participants) | 0 | 32 | 1 | 0 | 0 | 0 | 0 | 0
  CERVICAL, Cmax, Cycle 1 |  | 7.8457 (25.6236) | 31.0460 (NA) — Geometric coefficient of variation could not be calculated for single participant |  |  |  |  |
  CERVICAL, Ctau, Cycle 1: number analyzed (Participants) | 0 | 26 | 1 | 0 | 0 | 0 | 0 | 0
  CERVICAL, Ctau, Cycle 1 |  | 1.1026 (86.6644) | 8.3270 (NA) — Geometric coefficient of variation could not be calculated for single participant |  |  |  |  |
  CERVICAL, Ctau, Cycle 6: number analyzed (Participants) | 0 | 12 | 1 | 0 | 0 | 0 | 0 | 0
  CERVICAL, Ctau, Cycle 6 |  | 3.5457 (51.5684) | 19.2960 (NA) — Geometric coefficient of variation could not be calculated for single participant |  |  |  |  |
  HNSCC Q6W, Cmax, Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
  HNSCC Q6W, Cmax, Cycle 1 |  |  |  |  |  | 12.7362 (35.6947) | 70.9208 (22.9901) |
  HNSCC Q6W, Ctau, Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  HNSCC Q6W, Ctau, Cycle 1 |  |  |  |  |  |  | 6.6970 (NA) — Geometric coefficient of variation could not be calculated for single participant |
  HNSCC RANDOMIZED, Cmax, Cycle 1: number analyzed (Participants) | 13 | 1 | 24 | 22 | 0 | 0 | 0 | 0
  HNSCC RANDOMIZED, Cmax, Cycle 1 | 2.2993 (35.4890) | 6.8500 (NA) — Geometric coefficient of variation could not be calculated for single participant | 21.7283 (27.2945) | 71.1264 (25.9928) |  |  |  |
  HNSCC RANDOMIZED, Ctau, Cycle 1: number analyzed (Participants) | 9 | 1 | 18 | 17 | 0 | 0 | 0 | 0
  HNSCC RANDOMIZED, Ctau, Cycle 1 | 0.3314 (75.4863) | 1.2350 (NA) — Geometric coefficient of variation could not be calculated for single participant | 4.3179 (32.9785) | 14.0320 (34.6240) |  |  |  |
  HNSCC RANDOMIZED, Ctau, Cycle 6: number analyzed (Participants) | 2 | 0 | 3 | 3 | 0 | 0 | 0 | 0
  HNSCC RANDOMIZED, Ctau, Cycle 6 | 0.4949 (141.2509) |  | 15.0674 (100.4531) | 78.2867 (251.8571) |  |  |  |
  HNSCC_CPS<1, Cmax, Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1
  HNSCC_CPS<1, Cmax, Cycle 1 |  |  |  |  | 11.7572 (72.5188) |  |  | 39.4240 (NA) — Geometric coefficient of variation could not be calculated for single participant
  HNSCC_CPS<1, Ctau, Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  HNSCC_CPS<1, Ctau, Cycle 1 |  |  |  |  | 1.4240 (NA) — Geometric coefficient of variation could not be calculated for single participant |  |  |
  JAPAN PK/PD, Cmax, Cycle 1: number analyzed (Participants) | 0 | 2 | 3 | 3 | 0 | 0 | 0 | 0
  JAPAN PK/PD, Cmax, Cycle 1 |  | 7.8198 (7.7572) | 21.5695 (8.9060) | 69.9207 (31.4654) |  |  |  |
  JAPAN PK/PD, Ctau, Cycle 1: number analyzed (Participants) | 0 | 3 | 3 | 3 | 0 | 0 | 0 | 0
  JAPAN PK/PD, Ctau, Cycle 1 |  | 0.8800 (77.4102) | 4.3511 (28.1270) | 15.7566 (16.4440) |  |  |  |
  JAPAN PK/PD, Ctau, Cycle 6: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  JAPAN PK/PD, Ctau, Cycle 6 |  |  |  | 37.7140 (NA) — Geometric coefficient of variation could not be calculated for single participant |  |  |  |
  MELANOMA, Cmax, Cycle 1: number analyzed (Participants) | 0 | 8 | 14 | 0 | 0 | 0 | 0 | 0
  MELANOMA, Cmax, Cycle 1 |  | 8.3936 (43.1529) | 25.7542 (12.1953) |  |  |  |  |
  MELANOMA, Ctau, Cycle 1: number analyzed (Participants) | 0 | 4 | 13 | 0 | 0 | 0 | 0 | 0
  MELANOMA, Ctau, Cycle 1 |  | 1.4839 (42.9808) | 4.2946 (47.1494) |  |  |  |  |
  MELANOMA, Ctau, Cycle 6: number analyzed (Participants) | 0 | 4 | 5 | 0 | 0 | 0 | 0 | 0
  MELANOMA, Ctau, Cycle 6 |  | 3.2491 (66.9061) | 8.3404 (58.4213) |  |  |  |  |
  MSI-H/DMMR, Cmax, Cycle 1: number analyzed (Participants) | 0 | 17 | 0 | 0 | 0 | 0 | 0 | 0
  MSI-H/DMMR, Cmax, Cycle 1 |  | 7.4487 (20.8910) |  |  |  |  |  |
  MSI-H/DMMR, Ctau, Cycle 1: number analyzed (Participants) | 0 | 13 | 0 | 0 | 0 | 0 | 0 | 0
  MSI-H/DMMR, Ctau, Cycle 1 |  | 1.2458 (75.5891) |  |  |  |  |  |
  MSI-H/DMMR, Ctau, Cycle 6: number analyzed (Participants) | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0
  MSI-H/DMMR, Ctau, Cycle 6 |  | 3.3140 (32.6114) |  |  |  |  |  |
  NSCLC, Cmax, Cycle 1: number analyzed (Participants) | 0 | 91 | 2 | 0 | 0 | 0 | 0 | 0
  NSCLC, Cmax, Cycle 1 |  | 8.1306 (47.5103) | 16.0295 (88.7297) |  |  |  |  |
  NSCLC, Ctau, Cycle 1: number analyzed (Participants) | 0 | 73 | 2 | 0 | 0 | 0 | 0 | 0
  NSCLC, Ctau, Cycle 1 |  | 1.0848 (63.6879) | 2.7263 (66.3138) |  |  |  |  |
  NSCLC, Ctau, Cycle 6: number analyzed (Participants) | 0 | 26 | 0 | 0 | 0 | 0 | 0 | 0
  NSCLC, Ctau, Cycle 6 |  | 3.0399 (53.4515) |  |  |  |  |  |
  VIRAL-POSITIVE, Cmax, Cycle 1: number analyzed (Participants) | 0 | 15 | 0 | 0 | 0 | 0 | 0 | 0
  VIRAL-POSITIVE, Cmax, Cycle 1 |  | 7.5533 (20.0814) |  |  |  |  |  |
  VIRAL-POSITIVE, Ctau, Cycle 1: number analyzed (Participants) | 0 | 12 | 0 | 0 | 0 | 0 | 0 | 0
  VIRAL-POSITIVE, Ctau, Cycle 1 |  | 1.0357 (66.5632) |  |  |  |  |  |
  VIRAL-POSITIVE, Ctau, Cycle 6: number analyzed (Participants) | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
  VIRAL-POSITIVE, Ctau, Cycle 6 |  | 1.9175 (77.2467) |  |  |  |  |  |

64. Secondary Outcome: Part 2B: AUC (0-504 h) of Feladilimab
Description: Blood samples were collected for PK analysis. PK analysis was calculated based on standard non-compartmental method.
Time Frame: as for outcome 63
Population: Pharmacokinetic Population. Data is presented for participants who received feladilimab in combination with 200 mg Pembro. Only those participants with data available at specified categories have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Part 2B: Fela 0.100 mg/kg + Pembro 200 mg | Part 2B: Fela 0.300 mg/kg + Pembro 200 mg | Part 2B: Fela 1.000 mg/kg + Pembro 200 mg | Part 2B: Fela 3.000 mg/kg + Pembro 200 mg | Part 2B: Fela 24 mg + Pembro 200 mg | Part 2B: Fela 80 mg + Pembro 200 mg
Number analyzed (Participants) | 7 | 55 | 15 | 11 | 0 | 0
h*ug/mL
  BLADDER/UROTHELIAL: number analyzed (Participants) | 0 | 25 | 0 | 0 | 0 | 0
  BLADDER/UROTHELIAL |  | 1205.2673 (24.3543) |  |  |  |
  CERVICAL: number analyzed (Participants) | 0 | 14 | 0 | 0 | 0 | 0
  CERVICAL |  | 1254.7759 (39.2813) |  |  |  |
  HNSCC RANDOMIZED: number analyzed (Participants) | 7 | 1 | 15 | 11 | 0 | 0
  HNSCC RANDOMIZED | 294.2888 (46.7592) | 1500.4305 (NA) — Geometric coefficient of variation could not be calculated for single participant. | 4225.4602 (33.1105) | 13829.6005 (18.4367) |  |
  JAPAN PK/PD: number analyzed (Participants) | 0 | 2 | 2 | 1 | 0 | 0
  JAPAN PK/PD |  | 1367.0149 (359.19195) | 4258.3090 (280.08094) | 13890.8203 (NA) — Geometric coefficient of variation could not be calculated for single participant. |  |
  MELANOMA: number analyzed (Participants) | 0 | 8 | 14 | 0 | 0 | 0
  MELANOMA |  | 1082.3162 (48.1386) | 4098.4237 (45.2413) |  |  |
  MSI-H/DMMR: number analyzed (Participants) | 0 | 8 | 0 | 0 | 0 | 0
  MSI-H/DMMR |  | 1264.0452 (280.10101) |  |  |  |
  NSCLC: number analyzed (Participants) | 0 | 55 | 2 | 0 | 0 | 0
  NSCLC |  | 1318.6658 (664.64033) | 3071.5346 (1879.01269) |  |  |
  VIRAL-POSITIVE: number analyzed (Participants) | 0 | 7 | 0 | 0 | 0 | 0
  VIRAL-POSITIVE |  | 1415.2121 (355.25950) |  |  |  |

65. Secondary Outcome: Part 2B: AUC (0-1008 h) of Feladilimab
Description: Blood samples were collected for PK analysis. PK analysis was calculated based on standard non-compartmental method.
Time Frame: as for outcome 63
Population: Pharmacokinetic Population. Data is presented for participants who received feladilimab in combination with 400 mg Pembro. Only those participants with data available at specified categories have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Part 2B: Fela 48 mg + Pembro 400 mg | Part 2B: Fela 160 mg + Pembro 400 mg
Number analyzed (Participants) | 1 | 1
h*ug/mL | 3829.5867 (NA) — Geometric coefficient of variation could not be calculated for single participant. | 22182.5834 (NA) — Geometric coefficient of variation could not be calculated for single participant.

66. Secondary Outcome: Part 2B: Cmax and Ctau of Pembrolizumab
Description: Blood samples were collected for PK analysis. PK analysis was calculated based on standard non-compartmental method.
Time Frame: as for outcome 63
Population: Pharmacokinetic Population. As pre-specified in the protocol, PK data were not collected and analyzed for Pembrolizumab. Therefore, this PK parameter was not reported in this study.
Arm/Group | Part 2B: Fela 0.100 mg/kg + Pembro 200 mg | Part 2B: Fela 0.300 mg/kg + Pembro 200 mg | Part 2B: Fela 1.000 mg/kg + Pembro 200 mg | Part 2B: Fela 3.000 mg/kg + Pembro 200 mg | Part 2B: Fela 24 mg + Pembro 200 mg | Part 2B: Fela 48 mg + Pembro 400 mg | Part 2B: Fela 160 mg + Pembro 400 mg | Part 2B: Fela 80 mg + Pembro 200 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

67. Secondary Outcome: Part 2B: AUC (0-504h) of Pembrolizumab
Description: Blood samples were collected for PK analysis. PK analysis was calculated based on standard non-compartmental method.
Time Frame: as for outcome 63
Population: as for outcome 66
Arm/Group | Part 2B: Fela 0.100 mg/kg + Pembro 200 mg | Part 2B: Fela 0.300 mg/kg + Pembro 200 mg | Part 2B: Fela 1.000 mg/kg + Pembro 200 mg | Part 2B: Fela 3.000 mg/kg + Pembro 200 mg | Part 2B: Fela 24 mg + Pembro 200 mg | Part 2B: Fela 48 mg + Pembro 400 mg | Part 2B: Fela 160 mg + Pembro 400 mg | Part 2B: Fela 80 mg + Pembro 200 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

68. Secondary Outcome: Part 1A: Number of Participants With Positive Results in Anti-drug Antibody (ADA) Test by Feladilimab Dose Level
Description: Serum samples collected and tested for the presence of ADA with a screening assay.
Time Frame: Up to approximately 367 weeks
Population: All Treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: Feladilimab (Fela) 0.001 Milligram/Kilogram (mg/kg) | Part 1A: Fela 0.003 mg/kg | Part 1A: Fela 0.010 mg/kg | Part 1A: Fela 0.030 mg/kg | Part 1A: Fela 0.100 mg/kg | Part 1A: Fela 0.300 mg/kg | Part 1A: Fela 1.000 mg/kg | Part 1A: Fela 3.000 mg/kg | Part 1A: Fela 10.000 mg/kg
Number analyzed (Participants) | 1 | 1 | 2 | 7 | 24 | 25 | 15 | 27 | 7
Participants | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0

69. Secondary Outcome: Part 2A: Number of Participants With Positive Results in ADA Test by Feladilimab in Combination With GSK3174998 Dose Level
Description: Serum samples collected and tested for the presence of ADA with a screening assay.
Time Frame: Up to approximately 367 weeks
Population: All Treated population. Only participants who received GSK317499 with Feladilimab were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: Fela 8 mg + GSK3174998 8 mg | Part 2A: Fela 8 mg + GSK3174998 24 mg | Part 2A: Fela 24 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 80 mg
Number analyzed (Participants) | 1 | 4 | 16 | 4 | 3
Participants | 0 | 0 | 1 | 0 | 0

70. Secondary Outcome: Part 2A: Number of Participants With Positive Results in ADA Test by Feladilimab Dose Level in Combination With Pembrolizumab
Description: Serum samples collected and tested for the presence of ADA with a screening assay.
Time Frame: Up to approximately 367 weeks
Population: All Treated population. Only participants who received 200 mg pembrolizumab with Feladilimab were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: Fela 0.010 mg/kg + Pembrolizumab (Pembro) 200 mg | Part 2A: Fela 0.030 mg/kg + Pembro 200 mg | Part 2A: Fela 0.100 mg/kg + Pembro 200 mg | Part 2A: Fela 0.300 mg/kg + Pembro 200 mg | Part 2A: Fela 1.000 mg/kg + Pembro 200 mg | Part 2A: Fela 3.000 mg/kg + Pembro 200 mg
Number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11
Participants | 1 | 0 | 0 | 0 | 0 | 0

71. Secondary Outcome: Part 2A: Number of Participants With Positive Results in ADA in Pembrolizumab
Description: Serum samples collected and tested for the presence of ADA with a screening assay.
Time Frame: Up to approximately 367 weeks
Population: as for outcome 70
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: Fela 0.010 mg/kg + Pembrolizumab (Pembro) 200 mg | Part 2A: Fela 0.030 mg/kg + Pembro 200 mg | Part 2A: Fela 0.100 mg/kg + Pembro 200 mg | Part 2A: Fela 0.300 mg/kg + Pembro 200 mg | Part 2A: Fela 1.000 mg/kg + Pembro 200 mg | Part 2A: Fela 3.000 mg/kg + Pembro 200 mg
Number analyzed (Participants) | 5 | 5 | 5 | 8 | 11 | 11
Participants | 0 | 0 | 0 | 0 | 0 | 0

72. Secondary Outcome: Part 2A: Number of Participants With Positive Results in ADA in GSK3174998
Description: Serum samples collected and tested for the presence of ADA with a screening assay.
Time Frame: Up to approximately 367 weeks
Population: All Treated population. Only participants who received GSK3174998 with Feladilimab were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: Fela 8 mg + GSK3174998 8 mg | Part 2A: Fela 8 mg + GSK3174998 24 mg | Part 2A: Fela 24 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 80 mg
Number analyzed (Participants) | 1 | 4 | 16 | 4 | 3
Participants | 0 | 0 | 1 | 0 | 0

73. Secondary Outcome: Part 2A: Number of Participants With Positive Results in ADA Test by Feladilimab Combination With Chemotherapies Dose Level
Description: Serum samples collected and tested for the presence of ADA with a screening assay.
Time Frame: Up to approximately 367 weeks
Population: All Treated population. Only participants who received Chemotherapy with Feladilimab were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: Fela 24 mg + Chemotherapy | Part 2A: Fela 80 mg + Chemotherapy | Part 2A: Fela 24 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 80 mg + 200 mg Pembro + Chemotherapy
Number analyzed (Participants) | 6 | 36 | 13 | 22
Participants | 0 | 0 | 0 | 0

74. Secondary Outcome: Part 1B: Number of Participants With Positive Results in ADA Test by Feladilimab Dose Level
Description: Serum samples collected and tested for the presence of ADA with a screening assay.
Time Frame: Up to approximately 367 weeks
Population: All Treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1B: Fela 0.300 mg/kg | Part 1B: Fela 1.000 mg/kg | Part 1B: Fela 24 mg
Number analyzed (Participants) | 39 | 115 | 59
Participants | 0 | 0 | 1

75. Secondary Outcome: Part 2B: Number of Participants With Positive Results in ADA Test by Feladilimab Dose Level
Description: Serum samples collected and tested for the presence of ADA with a screening assay.
Time Frame: Up to approximately 367 weeks
Population: All Treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B: Fela 0.100 mg/kg + Pembro 200 mg | Part 2B: Fela 0.300 mg/kg + Pembro 200 mg | Part 2B: Fela 1.000 mg/kg + Pembro 200 mg | Part 2B: Fela 3.000 mg/kg + Pembro 200 mg | Part 2B: Fela 24 mg + Pembro 200 mg | Part 2B: Fela 48 mg + Pembro 400 mg | Part 2B: Fela 160 mg + Pembro 400 mg | Part 2B: Fela 80 mg + Pembro 200 mg
Number analyzed (Participants) | 14 | 255 | 44 | 23 | 4 | 6 | 5 | 1
Participants | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0

76. Secondary Outcome: Part 2B: Number of Participants With Positive Results in ADA in Pembrolizumab
Description: Serum samples collected and tested for the presence of ADA with a screening assay.
Time Frame: Up to approximately 367 weeks
Population: All Treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2B: Fela 0.100 mg/kg + Pembro 200 mg | Part 2B: Fela 0.300 mg/kg + Pembro 200 mg | Part 2B: Fela 1.000 mg/kg + Pembro 200 mg | Part 2B: Fela 3.000 mg/kg + Pembro 200 mg | Part 2B: Fela 24 mg + Pembro 200 mg | Part 2B: Fela 48 mg + Pembro 400 mg | Part 2B: Fela 160 mg + Pembro 400 mg | Part 2B: Fela 80 mg + Pembro 200 mg
Number analyzed (Participants) | 14 | 255 | 44 | 23 | 4 | 6 | 5 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

77. Secondary Outcome: Part 1A: Receptor Occupancy of Feladilimab
Description: Blood samples were collected to assess the cluster of differentiation 4 (CD4+) and cluster of differentiation 8 (CD8+) receptor occupancy by Feladilimab as a pharmacodynamic analysis. It was assessed using validated flow cytometry assay.
Time Frame: Up to approximately 367 weeks
Population: All treated population. As pre-specified in the protocol, only specified treatment arms were planned and hence there are 0 participants analyzed for rest of the arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent receptor occupancy
Arm/Group | Part 1A: Feladilimab (Fela) 0.001 Milligram/Kilogram (mg/kg) | Part 1A: Fela 0.003 mg/kg | Part 1A: Fela 0.010 mg/kg | Part 1A: Fela 0.030 mg/kg | Part 1A: Fela 0.100 mg/kg | Part 1A: Fela 0.300 mg/kg | Part 1A: Fela 1.000 mg/kg | Part 1A: Fela 3.000 mg/kg | Part 1A: Fela 10.000 mg/kg
Number analyzed (Participants) | 0 | 0 | 2 | 7 | 24 | 25 | 15 | 27 | 7
percent receptor occupancy
  %CD4+ |  |  | 74.643 (NA) — Geometric coefficient of variation could not be estimated due to insufficient number of participants with events. | 25.406 (21.423) | 90.229 (9.932) | 96.559 (2.934) | 94.007 (7.904) | 99.553 (1.559) | 96.030 (6.652)
  %CD8+ |  |  | 70.043 (NA) — Geometric coefficient of variation could not be estimated due to insufficient number of participants with events. | 16.646 (283.345) | 76.985 (16.349) | 80.933 (23.480) | 88.546 (10.383) | 95.934 (7.156) | 82.965 (29.404)

78. Secondary Outcome: Part 2A: Receptor Occupancy of Feladilimab
Description: as for outcome 77
Time Frame: Up to approximately 367 weeks
Population: All treated population. Analysis was planned for only Feladilimab and therefore arms are clubbed based on Feladilimab dosage for this endpoint. As pre-specified in the protocol, only specified treatment arms were planned and hence there are 0 participants analyzed for rest of the arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent receptor occupancy
Groups:
- Part 2A: Fela 8 mg + GSK3174998 8/24 mg: Participants with advanced solid tumors received 8 mg feladilimab IV infusion in combination with 8 mg or 24 mg of GSK3174998 IV infusion Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2A: Fela 80 mg + GSK3174998 24/80 mg: Participants with advanced solid tumors received 80 mg feladilimab IV infusion in combination with 24 mg or 80 mg of GSK3174998 IV infusion Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2A: Fela 24 mg + Chemotherapy (+/-Pembrolizumab): Participants with advanced solid tumors received 24 mg feladilimab IV infusion in combination with chemotherapy +/- 200 mg pembrolizumab Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2A: Fela 80 mg + Chemotherapy (+/- Pembrolizumab): Participants with advanced solid tumors received 80 mg feladilimab IV infusion in combination with chemotherapy +/- 200 mg pembrolizumab Q3W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
Arm/Group | Part 2A: Fela 0.010 mg/kg + Pembrolizumab (Pembro) 200 mg | Part 2A: Fela 0.030 mg/kg + Pembro 200 mg | Part 2A: Fela 0.100 mg/kg + Pembro 200 mg | Part 2A: Fela 0.300 mg/kg + Pembro 200 mg | Part 2A: Fela 1.000 mg/kg + Pembro 200 mg | Part 2A: Fela 3.000 mg/kg + Pembro 200 mg | Part 2A: Fela 8 mg + GSK3174998 8/24 mg | Part 2A: Fela 24 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 24/80 mg | Part 2A: Fela 24 mg + Chemotherapy (+/-Pembrolizumab) | Part 2A: Fela 80 mg + Chemotherapy (+/- Pembrolizumab) | Part 2A: Fela 24 mg + Dostarlimab 500 mg + Cobolimab 300 mg | Part 2A: Fela 24 mg + Bintrafusp Alfa 2400 mg
Number analyzed (Participants) | 5 | 0 | 5 | 8 | 11 | 11 | 5 | 16 | 7 | 19 | 58 | 0 | 0
percent receptor occupancy
  %CD4+ | 87.351 (4.630) |  | 97.962 (2.282) | 98.244 (1.888) | 99.364 (1.333) | 99.704 (0.995) | 93.157 (1.017) | 97.324 (3.753) | 99.887 (0.176) | 96.417 (7.179) | 94.324 (36.547) |  |
  %CD8+ | 82.973 (13.323) |  | 99.782 (4.173) | 93.448 (10.622) | 97.995 (3.700) | 100.887 (2.264) | 79.261 (4.878) | 93.221 (8.141) | 96.540 (4.157) | 94.960 (7.366) | 101.528 (18.835) |  |

79. Secondary Outcome: Part 1B: Receptor Occupancy of Feladilimab
Description: as for outcome 77
Time Frame: Up to approximately 367 weeks
Population: All treated population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent receptor occupancy
Arm/Group | Part 1B: Fela 0.300 mg/kg | Part 1B: Fela 1.000 mg/kg | Part 1B: Fela 24 mg
Number analyzed (Participants) | 39 | 115 | 59
percent receptor occupancy
  %CD4+ | 96.520 (4.258) | 99.179 (3.926) | 98.128 (2.192)
  %CD8+ | 90.111 (11.700) | 96.160 (9.429) | 81.219 (21.037)

80. Secondary Outcome: Part 2B: Receptor Occupancy of Feladilimab
Description: as for outcome 77
Time Frame: Up to approximately 367 weeks
Population: as for outcome 77
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent receptor occupancy
Arm/Group | Part 2B: Fela 0.100 mg/kg + Pembro 200 mg | Part 2B: Fela 0.300 mg/kg + Pembro 200 mg | Part 2B: Fela 1.000 mg/kg + Pembro 200 mg | Part 2B: Fela 3.000 mg/kg + Pembro 200 mg | Part 2B: Fela 24 mg + Pembro 200 mg | Part 2B: Fela 48 mg + Pembro 400 mg | Part 2B: Fela 160 mg + Pembro 400 mg | Part 2B: Fela 80 mg + Pembro 200 mg
Number analyzed (Participants) | 14 | 255 | 44 | 23 | 4 | 6 | 5 | 0
percent receptor occupancy
  %CD4+ | 95.795 (4.267) | 95.750 (8.757) | 99.004 (1.658) | 99.988 (0.827) | 87.194 (NA) — geometric coefficient of variation could not be estimated due to insufficient number of participants with events. | 101.663 (2.364) | 100.790 (1.198) |
  %CD8+ | 89.773 (8.360) | 93.581 (9.049) | 96.900 (4.013) | 102.610 (9.138) | 57.856 (NA) — geometric coefficient of variation could not be estimated due to insufficient number of participants with events. | 106.059 (14.555) | 103.802 (6.179) |

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious adverse events (non-SAEs) and serious adverse events (SAEs) were collected up to approximately 367 weeks.
Description: All participants who received at least one dose of study treatment.
Groups:
- Part 2B: Fela 0.100 mg/kg + Pembro 200 mg: Participants with advanced solid tumors received 0.100 mg/kg feladilimab IV infusion in combination with 200 mg of pembro IV infusion every 6 Week (Q6W) of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2B: Fela 0.300 mg/kg + Pembro 200 mg: Participants with advanced solid tumors received 0.300 mg/kg feladilimab IV infusion in combination with 200 mg of pembro IV infusion Q6W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2B: Fela 1.000 mg/kg + Pembro 200 mg: Participants with advanced solid tumors received 1.000 mg/kg feladilimab IV infusion in combination with 200 mg of pembro IV infusion Q6W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2B: Fela 3.000 mg/kg + Pembro 200 mg: Participants with advanced solid tumors received 3.000 mg/kg feladilimab IV infusion in combination with 200 mg of pembro IV infusion Q6W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2B: Fela 24 mg + Pembro 200 mg: Participants with advanced solid tumors received 24 mg feladilimab IV infusion in combination with 200 mg of pembro IV infusion Q6W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2B: Fela 48 mg + Pembro 400 mg: Participants with advanced solid tumors received 48 mg feladilimab IV infusion in combination with 400 mg of pembro IV infusion Q6W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2B: Fela 160 mg + Pembro 400 mg: Participants with advanced solid tumors received 160 mg feladilimab IV infusion in combination with 400 mg of pembro IV infusion Q6W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
- Part 2B: Fela 80 mg + Pembro 200 mg: Participants with advanced solid tumors received 80 mg feladilimab IV infusion in combination with 400 mg of pembro IV infusion Q6W of each 21-day Cycle up to until disease progression, unacceptable toxicity, or withdrawal of consent, or for up to maximum of 35 cycles.
Arm/Group | Part 1A: Feladilimab (Fela) 0.001 Milligram/Kilogram (mg/kg) | Part 1A: Fela 0.003 mg/kg | Part 1A: Fela 0.010 mg/kg | Part 1A: Fela 0.030 mg/kg | Part 1A: Fela 0.100 mg/kg | Part 1A: Fela 0.300 mg/kg | Part 1A: Fela 1.000 mg/kg | Part 1A: Fela 3.000 mg/kg | Part 1A: Fela 10.000 mg/kg | Part 1B: Fela 0.300 mg/kg | Part 1B: Fela 1.000 mg/kg | Part 1B: Fela 24 mg | Part 2A: Fela 0.010 mg/kg + Pembrolizumab (Pembro) 200 mg | Part 2A: Fela 0.030 mg/kg + Pembro 200 mg | Part 2A: Fela 0.100 mg/kg + Pembro 200 mg | Part 2A: Fela 0.300 mg/kg + Pembro 200 mg | Part 2A: Fela 1.000 mg/kg + Pembro 200 mg | Part 2A: Fela 3.000 mg/kg + Pembro 200 mg | Part 2A: Fela 8 mg + GSK3174998 8 mg | Part 2A: Fela 8 mg + GSK3174998 24 mg | Part 2A: Fela 24 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 24 mg | Part 2A: Fela 80 mg + GSK3174998 80 mg | Part 2A: Fela 24 mg + Chemotherapy | Part 2A: Fela 80 mg + Chemotherapy | Part 2A: Fela 24 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 80 mg + 200 mg Pembro + Chemotherapy | Part 2A: Fela 24 mg + Dostarlimab 500 mg + Cobolimab 300 mg | Part 2A: Fela 24 mg + Bintrafusp Alfa 2400 mg | Part 2B: Fela 0.100 mg/kg + Pembro 200 mg | Part 2B: Fela 0.300 mg/kg + Pembro 200 mg | Part 2B: Fela 1.000 mg/kg + Pembro 200 mg | Part 2B: Fela 3.000 mg/kg + Pembro 200 mg | Part 2B: Fela 24 mg + Pembro 200 mg | Part 2B: Fela 48 mg + Pembro 400 mg | Part 2B: Fela 160 mg + Pembro 400 mg | Part 2B: Fela 80 mg + Pembro 200 mg | Crossover: Fela 0.100 mg/kg + Pembro 200 mg | Crossover: Fela 0.300 mg/kg + Pembro 200 mg | Crossover: Fela 1.000 mg/kg + Pembro 200 mg | Crossover: Fela 3.000 mg/kg + Pembro 200 mg | Crossover: Fela 24 mg + Pembro 200 mg | Crossover: Pembro 200 mg
All-Cause Mortality (participants affected / at risk) | 1/1 | 1/1 | 2/2 | 7/7 | 18/24 | 17/25 | 11/15 | 21/27 | 3/7 | 25/39 | 69/115 | 48/59 | 2/5 | 4/5 | 5/5 | 6/8 | 6/11 | 7/11 | 1/1 | 3/4 | 13/16 | 3/4 | 2/3 | 4/6 | 31/36 | 7/13 | 13/22 | 0/1 | 1/4 | 12/14 | 202/255 | 31/44 | 17/23 | 2/4 | 3/6 | 3/5 | 1/1 | 1/1 | 14/19 | 32/42 | 2/2 | 1/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 1/2 | 2/7 | 6/24 | 8/25 | 4/15 | 12/27 | 1/7 | 9/39 | 44/115 | 19/59 | 3/5 | 2/5 | 3/5 | 2/8 | 3/11 | 4/11 | 0/1 | 2/4 | 5/16 | 2/4 | 1/3 | 4/6 | 13/36 | 3/13 | 17/22 | 0/1 | 1/4 | 3/14 | 126/255 | 17/44 | 7/23 | 1/4 | 2/6 | 2/5 | 1/1 | 0/1 | 4/19 | 12/42 | 1/2 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 2/2 | 7/7 | 19/24 | 23/25 | 12/15 | 17/27 | 6/7 | 32/39 | 101/115 | 51/59 | 5/5 | 5/5 | 5/5 | 5/8 | 8/11 | 10/11 | 0/1 | 4/4 | 14/16 | 3/4 | 3/3 | 6/6 | 36/36 | 13/13 | 22/22 | 1/1 | 4/4 | 13/14 | 236/255 | 40/44 | 21/23 | 4/4 | 5/6 | 4/5 | 1/1 | 1/1 | 15/19 | 26/42 | 1/2 | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1A: Feladilimab (Fela) 0.001 Milligram/Kilogram (mg/kg) (N=1) | Part 1A: Fela 0.003 mg/kg (N=1) | Part 1A: Fela 0.010 mg/kg (N=2) | Part 1A: Fela 0.030 mg/kg (N=7) | Part 1A: Fela 0.100 mg/kg (N=24) | Part 1A: Fela 0.300 mg/kg (N=25) | Part 1A: Fela 1.000 mg/kg (N=15) | Part 1A: Fela 3.000 mg/kg (N=27) | Part 1A: Fela 10.000 mg/kg (N=7) | Part 1B: Fela 0.300 mg/kg (N=39) | Part 1B: Fela 1.000 mg/kg (N=115) | Part 1B: Fela 24 mg (N=59) | Part 2A: Fela 0.010 mg/kg + Pembrolizumab (Pembro) 200 mg (N=5) | Part 2A: Fela 0.030 mg/kg + Pembro 200 mg (N=5) | Part 2A: Fela 0.100 mg/kg + Pembro 200 mg (N=5) | Part 2A: Fela 0.300 mg/kg + Pembro 200 mg (N=8) | Part 2A: Fela 1.000 mg/kg + Pembro 200 mg (N=11) | Part 2A: Fela 3.000 mg/kg + Pembro 200 mg (N=11) | Part 2A: Fela 8 mg + GSK3174998 8 mg (N=1) | Part 2A: Fela 8 mg + GSK3174998 24 mg (N=4) | Part 2A: Fela 24 mg + GSK3174998 24 mg (N=16) | Part 2A: Fela 80 mg + GSK3174998 24 mg (N=4) | Part 2A: Fela 80 mg + GSK3174998 80 mg (N=3) | Part 2A: Fela 24 mg + Chemotherapy (N=6) | Part 2A: Fela 80 mg + Chemotherapy (N=36) | Part 2A: Fela 24 mg + 200 mg Pembro + Chemotherapy (N=13) | Part 2A: Fela 80 mg + 200 mg Pembro + Chemotherapy (N=22) | Part 2A: Fela 24 mg + Dostarlimab 500 mg + Cobolimab 300 mg (N=1) | Part 2A: Fela 24 mg + Bintrafusp Alfa 2400 mg (N=4) | Part 2B: Fela 0.100 mg/kg + Pembro 200 mg (N=14) | Part 2B: Fela 0.300 mg/kg + Pembro 200 mg (N=255) | Part 2B: Fela 1.000 mg/kg + Pembro 200 mg (N=44) | Part 2B: Fela 3.000 mg/kg + Pembro 200 mg (N=23) | Part 2B: Fela 24 mg + Pembro 200 mg (N=4) | Part 2B: Fela 48 mg + Pembro 400 mg (N=6) | Part 2B: Fela 160 mg + Pembro 400 mg (N=5) | Part 2B: Fela 80 mg + Pembro 200 mg (N=1) | Crossover: Fela 0.100 mg/kg + Pembro 200 mg (N=1) | Crossover: Fela 0.300 mg/kg + Pembro 200 mg (N=19) | Crossover: Fela 1.000 mg/kg + Pembro 200 mg (N=42) | Crossover: Fela 3.000 mg/kg + Pembro 200 mg (N=2) | Crossover: Fela 24 mg + Pembro 200 mg (N=1) | Crossover: Pembro 200 mg (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac aneurysm (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myopericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia of malignancy (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blindness (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orocutaneous fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug intolerance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Performance status decreased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected fistula (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infective aneurysm (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infective myositis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 13 (14) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour perforation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Priapism (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 9 (11) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheal compression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1A: Feladilimab (Fela) 0.001 Milligram/Kilogram (mg/kg) (N=1) | Part 1A: Fela 0.003 mg/kg (N=1) | Part 1A: Fela 0.010 mg/kg (N=2) | Part 1A: Fela 0.030 mg/kg (N=7) | Part 1A: Fela 0.100 mg/kg (N=24) | Part 1A: Fela 0.300 mg/kg (N=25) | Part 1A: Fela 1.000 mg/kg (N=15) | Part 1A: Fela 3.000 mg/kg (N=27) | Part 1A: Fela 10.000 mg/kg (N=7) | Part 1B: Fela 0.300 mg/kg (N=39) | Part 1B: Fela 1.000 mg/kg (N=115) | Part 1B: Fela 24 mg (N=59) | Part 2A: Fela 0.010 mg/kg + Pembrolizumab (Pembro) 200 mg (N=5) | Part 2A: Fela 0.030 mg/kg + Pembro 200 mg (N=5) | Part 2A: Fela 0.100 mg/kg + Pembro 200 mg (N=5) | Part 2A: Fela 0.300 mg/kg + Pembro 200 mg (N=8) | Part 2A: Fela 1.000 mg/kg + Pembro 200 mg (N=11) | Part 2A: Fela 3.000 mg/kg + Pembro 200 mg (N=11) | Part 2A: Fela 8 mg + GSK3174998 8 mg (N=1) | Part 2A: Fela 8 mg + GSK3174998 24 mg (N=4) | Part 2A: Fela 24 mg + GSK3174998 24 mg (N=16) | Part 2A: Fela 80 mg + GSK3174998 24 mg (N=4) | Part 2A: Fela 80 mg + GSK3174998 80 mg (N=3) | Part 2A: Fela 24 mg + Chemotherapy (N=6) | Part 2A: Fela 80 mg + Chemotherapy (N=36) | Part 2A: Fela 24 mg + 200 mg Pembro + Chemotherapy (N=13) | Part 2A: Fela 80 mg + 200 mg Pembro + Chemotherapy (N=22) | Part 2A: Fela 24 mg + Dostarlimab 500 mg + Cobolimab 300 mg (N=1) | Part 2A: Fela 24 mg + Bintrafusp Alfa 2400 mg (N=4) | Part 2B: Fela 0.100 mg/kg + Pembro 200 mg (N=14) | Part 2B: Fela 0.300 mg/kg + Pembro 200 mg (N=255) | Part 2B: Fela 1.000 mg/kg + Pembro 200 mg (N=44) | Part 2B: Fela 3.000 mg/kg + Pembro 200 mg (N=23) | Part 2B: Fela 24 mg + Pembro 200 mg (N=4) | Part 2B: Fela 48 mg + Pembro 400 mg (N=6) | Part 2B: Fela 160 mg + Pembro 400 mg (N=5) | Part 2B: Fela 80 mg + Pembro 200 mg (N=1) | Crossover: Fela 0.100 mg/kg + Pembro 200 mg (N=1) | Crossover: Fela 0.300 mg/kg + Pembro 200 mg (N=19) | Crossover: Fela 1.000 mg/kg + Pembro 200 mg (N=42) | Crossover: Fela 3.000 mg/kg + Pembro 200 mg (N=2) | Crossover: Fela 24 mg + Pembro 200 mg (N=1) | Crossover: Pembro 200 mg (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (7) | 5 (5) | 4 (5) | 2 (2) | 2 (2) | 7 (7) | 29 (32) | 6 (7) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 16 (22) | 4 (4) | 9 (9) | 0 (0) | 0 (0) | 3 (3) | 53 (61) | 8 (8) | 6 (6) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (5) | 1 (1) | 2 (4) | 0 (0) | 1 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 14 (28) | 3 (4) | 5 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 6 (12) | 4 (5) | 3 (7) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac aneurysm (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 13 (13) | 4 (4) | 4 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 2 (3) | 2 (2) | 2 (2) | 1 (1) | 9 (11) | 9 (10) | 7 (7) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 31 (39) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 6 (6) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (9) | 2 (2) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 5 (5) | 0 (0) | 2 (2) | 13 (14) | 11 (12) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 4 (4) | 4 (5) | 0 (0) | 1 (1) | 1 (1) | 36 (42) | 8 (9) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 3 (6) | 3 (3) | 0 (0) | 6 (6) | 21 (27) | 9 (10) | 0 (0) | 1 (1) | 1 (1) | 1 (7) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 2 (4) | 1 (2) | 1 (1) | 1 (1) | 12 (13) | 1 (1) | 7 (10) | 0 (0) | 1 (1) | 0 (0) | 46 (64) | 7 (9) | 8 (8) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 14 (15) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 3 (4) | 6 (10) | 0 (0) | 8 (13) | 24 (29) | 9 (11) | 3 (4) | 2 (2) | 3 (3) | 1 (5) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 5 (6) | 20 (25) | 5 (5) | 11 (14) | 0 (0) | 1 (1) | 2 (2) | 46 (62) | 7 (9) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 7 (8) | 0 (0) | 0 (0) | 0 (0)
Noninfective gingivitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (6) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 5 (7) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (2) | 2 (2) | 3 (5) | 0 (0) | 5 (5) | 18 (19) | 2 (2) | 1 (1) | 3 (3) | 3 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 2 (3) | 1 (1) | 6 (6) | 2 (3) | 6 (7) | 0 (0) | 1 (1) | 1 (1) | 28 (39) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 2 (2) | 1 (1) | 4 (6) | 2 (2) | 11 (15) | 27 (28) | 15 (15) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (5) | 1 (1) | 1 (1) | 3 (4) | 10 (14) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 48 (53) | 10 (16) | 4 (6) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 5 (5) | 0 (0) | 1 (1) | 0 (0)
Catheter site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 5 (5) | 4 (4) | 3 (3) | 6 (7) | 0 (0) | 5 (6) | 20 (27) | 9 (11) | 1 (2) | 1 (1) | 5 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 8 (10) | 4 (4) | 10 (10) | 0 (0) | 2 (2) | 1 (3) | 46 (51) | 8 (9) | 4 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 6 (9) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 7 (7) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 13 (16) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 6 (6) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 3 (4) | 1 (2) | 2 (2) | 4 (7) | 14 (18) | 6 (6) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 5 (5) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 33 (37) | 12 (12) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cytolysis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected bite (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheostomy infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 14 (18) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 21 (30) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiation associated pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site discomfort (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site oedema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 6 (8) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 24 (34) | 3 (5) | 5 (10) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (3) | 2 (2) | 0 (0) | 2 (3) | 7 (10) | 7 (8) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 23 (28) | 3 (6) | 5 (8) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 9 (9) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 32 (40) | 4 (5) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 7 (17) | 4 (10) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 5 (9) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 14 (14) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cell death (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 1 (1) | 2 (2) | 6 (7) | 1 (2) | 5 (6) | 13 (16) | 7 (7) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 6 (7) | 4 (4) | 4 (5) | 0 (0) | 0 (0) | 1 (1) | 39 (42) | 4 (4) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 15 (16) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (9) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (10) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 7 (8) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 7 (7) | 14 (18) | 3 (3) | 2 (3) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 5 (6) | 0 (0) | 1 (1) | 1 (1) | 36 (40) | 7 (8) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 3 (3) | 2 (3) | 3 (7) | 15 (17) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (4) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 32 (35) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (6) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 16 (16) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 7 (9) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (7) | 7 (9) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 12 (15) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 10 (11) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 12 (12) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Akathisia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electric shock sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fine motor skill dysfunction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 8 (12) | 5 (5) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (7) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 13 (13) | 6 (8) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 6 (6) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 12 (13) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Personality change (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 11 (13) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 4 (5) | 2 (2) | 2 (2) | 13 (13) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 8 (10) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 44 (51) | 6 (6) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 19 (19) | 7 (7) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 1 (2) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 42 (47) | 6 (6) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased viscosity of upper respiratory secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 10 (11) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulite (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dandruff (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 13 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (9) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 6 (6) | 7 (8) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 23 (26) | 8 (9) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 1 (2) | 2 (2) | 13 (14) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 7 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin warm (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-08-20): https://cdn.clinicaltrials.gov/large-docs/55/NCT02723955/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/55/NCT02723955/SAP_001.pdf